# **Appendix 16.1.9 Documentation of Statistical Methods**

Integrated Analysis Plan Version 1.0, 22 November 2019

Statistical Analysis Output

WinNonlin Core Output

WinNonlin Plots

Final 1.0

## Integrated Analysis Plan

Clinical Trial Protocol Identification No. MS200095 0038

Title

An open-label, single-dose, randomized, 2-period, 2-sequence cross-over, single-center Phase I trial in healthy subjects to assess the bioequivalence of tepotinib tablet formulation 3 administered as 5 tablets of 100 mg versus 2 tablets of 250 mg

dose strength

Trial Phase

Ι

Investigational Medicinal

Tepotinib (MSC2156119J)

Product(s)

Clinical Trial Protocol

Version

05 Sep 2019 / Version 1.0

Integrated Analysis Plan Author

**Coordinating Author** 

| Function Author / Biostatistician | PI | Merck | PI | |
|---|---|---|---|---|
| DI Nondana DI | Function | | Author / Biostati | stician |
| ri Nuvisan ri | PI | Nuvisan | PI | |

Integrated Analysis Plan Date and Version 22 Nov 2019 / Final Version 1.0

Integrated Analysis Plan Reviewers



#### Confidential

This document is the property of Merck KGaA, Darmstadt, Germany, or one of its affiliated companies.

It is intended for restricted use only and may not - in full or part - be passed on, reproduced, published or used without express permission of Merck KGaA, Darmstadt, Germany or its affiliate.

Copyright © 2019 by Merck KGaA, Darmstadt, Germany or its affiliate. All rights reserved.

## Signature Page

Integrated Analysis Plan: MS200095 0038

An open-label, single-dose, randomized, 2-period, 2-sequence cross-over, single-center Phase I trial in healthy subjects to assess the bioequivalence of tepotinib tablet formulation 3 administered as 5 tablets of 100 mg versus 2 tablets of 250 mg dose strength

Approval of the IAP by all Merck Data Analysis Responsibles is documented within Cara. With the approval within Cara, the Merck responsible for each of the analysis also takes responsibility that all reviewers' comments are addressed adequately.

| Merck responsible | | Date | Signature |
|-------------------|--------|------------|-----------------|
| PI | ,Merck | Via Cara a | pproval process |
| PI | , | Via Cara a | pproval process |
| PI | Merck | | |

# 1 Table of Contents

| Integrated Analy | sis Plan | 1 |
|---|---|---|
| Signature Page | 2 | |
| 1 | Table of Contents | 3 |
| 2 | List of Abbreviations and Definition of Terms | 5 |
| 3 | Modification History | 6 |
| 4 | Purpose of the Integrated Analysis Plan | 6 |
| 5 | Objectives and Endpoints | 7 |
| 6 | Overview of Planned Analyses | 7 |
| 6.1 | Interim Analysis | 7 |
| 6.2 | Final Analysis | 8 |
| 7 | Changes to the Planned Analyses in the Clinical Trial Protocol | 8 |
| 8 | Protocol Deviations and Analysis Sets | 8 |
| 8.1 | Definition of Protocol Deviations and Analysis Sets | 8 |
| 8.2 | Definition of Analysis Sets | 9 |
| 9 | General Specifications for Data Analyses | 9 |
| 10 | Trial Subjects | 11 |
| 10.1 | Disposition of Subjects and Discontinuations | 11 |
| 10.2 | Protocol Deviations | 12 |
| 10.2.1 | Important Protocol Deviations | 12 |
| 10.2.2 | Reasons Leading to the Exclusion from an Analysis Set | 12 |
| 11 | Demographics and Other Baseline Characteristics | 12 |
| 11.1 | Demographics | 12 |
| 11.2 | Medical History | 13 |
| 11.3 | Other Baseline Characteristics | 13 |
| 12 | Previous or Concomitant Medications/Procedures | 13 |
| 13 | Treatment Compliance and Exposure | 14 |
| 14 | Efficacy Analyses | 14 |
| 15 | Safety Analyses | 14 |
| 15.1 | Adverse Events | 14 |
| 15.1.1 | All Adverse Events | 15 |

| • | Final 1. |
|---|---|
| Adverse Events Leading to Treatment Discontinuation | 16 |
| Deaths, Other Serious Adverse Events, and Other Significant<br>Adverse Events | 16 |
| Deaths | 16 |
| Serious Adverse Events | 16 |
| Other Significant Adverse Event | 17 |
| Adverse Events of Special Interest | 17 |
| Clinical Laboratory Evaluation | 17 |
| Vital Signs | 18 |
| ECG Evaluation | 18 |
| Analyses of Other Endpoints | 19 |
| Pharmacokinetics | 19 |
| ations for Plasma Concentration Data | 19 |
| ations for PK Parameter Data | 19 |
| Primary Endpoints | 20 |
| Secondary Endpoints | 21 |
| Exploratory Endpoints | 21 |
| Plasma Concentration Data | 21 |
| Estimation of Individual Pharmacokinetic Parameters | 22 |
| Pharmacogenetics | 24 |
| References | 25 |
| Appendices | 25 |
| | Adverse Events Deaths Serious Adverse Events Other Significant Adverse Event Adverse Events of Special Interest Clinical Laboratory Evaluation Vital Signs ECG Evaluation Analyses of Other Endpoints Pharmacokinetics ations for Plasma Concentration Data |

MS200095 0038 Final 1.0

## 2 List of Abbreviations and Definition of Terms

AE Adverse Event

AESI Adverse Event of Special Interest

ANOVA Analysis of VARIANCE

BMI Body Mass Index

eCRF Electronic Case Report Form

CSR Clinical Study Report
CV% Coefficient of Variation

ECG Electrocardiogram

GeoCV% Geometric Coefficient of Variation

GeoMean Geometric Mean

IAP Integrated Analysis Plan

ICH International Conference on Harmonization

IMP Investigational Medicinal Product
LCI Lower Confidence Interval Bound

LLOQ Lower Limit of Quantification

Max Maximum

MCAR Missing Completely at Random

MedDRA Medical Dictionary for Regulatory Activities

Min Minimum

NCI-CTCAE National Cancer Institute – Common Terminology Criteria for Adverse

**Events** 

PD Pharmacodynamics
PGx Pharmacogenetics
PK Pharmacokinetics
PT Preferred Term
Q1 First Quartile
Q3 Third Quartile

QTcF Corrected QT interval per Fridericia's formula

MS200095\_0038 Final 1.0

SAE Serious Adverse Event SDTM Study Data Tabulation Model SEM Standard Error of the Mean SOC System Organ Class TEAE Treatment Emergent Adverse Event Tablet Formulation 3 TF3 UCI Upper Confidence Interval Bound ULOQ Upper Limit of Quantification

## 3 Modification History

| Unique<br>Identifier for<br>Version | Date of<br>IAP Version | Author | Changes from the Previous Version |
|---|---|---|---|
| Final 1.0 | 22-NOV-2019 | PI<br>,<br>Nuvisan | Original Document |

## 4 Purpose of the Integrated Analysis Plan

The purpose of this integrated analysis plan (IAP) is to document technical and detailed specifications for the final analysis of data collected for protocol MS200095\_0038. Results of the analyses described in this IAP will be included in the Clinical Study Report (CSR). Additionally, the planned analyses identified in this IAP will be included in regulatory submissions or future manuscripts. Any post-hoc or unplanned analyses performed to provide results for inclusion in the CSR but not identified in this prospective IAP will be clearly identified in the CSR.

The IAP is based upon section 8 (Statistics) of the trial protocol and protocol amendments and is prepared in compliance with ICH E9.

MS200095\_0038 Final 1.0

# **5** Objectives and Endpoints

| | | Objective | Endpoint | IAP<br>section |
|---|---|---|---|---|
| Primary<br>Objectives | • | To demonstrate bioequivalence between 5 tablets of the 100 mg dose strength of tepotinib tablet formulation 3 (TF3, test treatment) and 2 tablets of the 250 mg dose strength of TF3 (reference treatment) after single dose administration in healthy subjects under fasting conditions | <ul> <li>Primary Endpoints:</li> <li>Area under the plasma concentration-time curve (AUC) from time zero (=dosing time) to the last sampling time at which the concentration is at or above the lower limit of quantification (AUC₀-t).</li> <li>AUC from time zero extrapolated to infinity (AUC₀-∞).</li> <li>Maximum plasma concentration (Cmax) of tepotinib observed from time zero to 168 h postdose of each period.</li> </ul> | 16.1.1 |
| Secondary<br>Objectives | • | To further investigate the Pharmacokinetic (PK) of tepotinib. | Secondary endpoints: Time to reach C <sub>max</sub> (t <sub>max</sub> ), terminal half-life (t <sub>1/2</sub> ), apparent total body clearance considering the fraction of dose absorbed (CL/f) and apparent volume of distribution during terminal phase (V <sub>z</sub> /f) of tepotinib observed from time zero to 168 h postdose of each period. | 16.1.2 |
| | • | To further assess the safety and tolerability of tepotinib TF3 under fasting conditions. | <ul> <li>Occurrence of treatment-emergent<br/>adverse events (TEAEs; incidence,<br/>frequency, intensity and causality),<br/>occurrence of changes in safety<br/>laboratory assessments, 12-lead<br/>electrocardiograms (ECGs) and vital<br/>signs.</li> </ul> | 15 |
| Exploratory<br>Objectives | • | To investigate the PK of tepotinib metabolites. | PK profiles of tepotinib metabolites: AUC <sub>0-t</sub> , AUC <sub>0-∞</sub> , C <sub>max</sub> , t <sub>max</sub> , t <sub>1/2</sub> of tepotinib metabolites observed from time zero to 168 h postdose of each period. | 16.1.3 |
| | • | To explore the effect of pharmacogenetics (PGx) and variations of associated genes on the PK profile of tepotinib (if applicable). | <ul> <li>Genetic variants and mutations in<br/>genes that potentially influence PK of<br/>tepotinib.</li> </ul> | 16.2 |

# **6** Overview of Planned Analyses

# 6.1 Interim Analysis

No interim analysis is planned for this trial.

## 6.2 Final Analysis

The final, planned analyses identified in the Clinical Trial Protocol and in this IAP will be performed after the last subject has completed the last visit, i.e. end of trial visit/early termination visit with all trial data in-house, all data queries resolved, and the database locked.

Nodatabase can be locked until this IAP has been approved.

# 7 Changes to the Planned Analyses in the Clinical Trial Protocol

The statistical methods as described in the protocol were adopted.

# **8** Protocol Deviations and Analysis Sets

## 8.1 Definition of Protocol Deviations and Analysis Sets

Important protocol deviations are protocol deviations that might significantly affect the completeness, accuracy, and/or reliability of the trial data or that might significantly affect a subject's rights, safety, or well-being.

No formal data review meeting will be held. However, the following deviations will be identified and confirmed before the database is locked: Important protocol deviations include

- Deviations from the inclusion and exclusion criteria
- Concomitant medication violations (see Section 6.5.1 of the protocol)
- Use of prohibited medicines (see Section 6.5.2 of the protocol)
- Subjects that receive incorrect treatment or dose
- Sample processing errors that may lead to inaccurate bioanalytical results
- Vomiting or diarrhea following oral dosing (these instances will be discussed on a caseby-case basis)
- Deviation from Good Clinical Practice
- Non-compliance to trial procedures or deviations from trial procedures likely to affect the primary endpoints (e.g. subject develops withdrawal criteria whilst on the trial but is not withdrawn)
- Deviation from trial medication compliance in terms of medical conditions and/or adverse events (AEs) that may have interfered with drug disposition or with respect to factors likely to affect the primary endpoints

All important protocol deviations will be documented in Clinical Data Interchange Standard Consortium (CDISC) Study Data Tabulation Model (SDTM) datasets whether identified through sites monitoring or medical review.

## 8.2 Definition of Analysis Sets

| Analysis Set | Description |
|---|---|
| Screening | All subjects who signed informed consent. |
| Safety | The Safety Analysis Set will include all subjects who have received at least 1 dose of planned Investigational Medicinal Product (IMP) and have had 1 subsequent safety assessment. |
| PK | The PK Analysis Set will include all subjects without any relevant protocol deviations with respect to PK and absence of factors likely to affect the comparability of PK results, with adequate trial medication compliance, and who have valid primary endpoints for both treatments. |

Relevant decisions will be made before database lock.

# **9** General Specifications for Data Analyses

Statistical analyses will be performed using the computer program package SAS<sup>®</sup> System for Windows<sup>TM</sup> (Version 9.4 or later; SAS Institute, Cary, North Carolina, USA).

The results of this trial will be reported using summary tables, figures, and data listings, as appropriate. All data will be summarized overall and/or by treatment and/or by scheduled time point, as appropriate.

For demographic, baseline and safety assessments, continuous measurements will be summarized by means of descriptive statistics (i.e. number and percentage of observations, number and percentage of missing observations, mean, standard deviation [SD], median, the first and third quartile [Q1 and Q3], minimum [Min], and maximum [Max]) and categorical data will be summarized by means of frequency tables (i.e. count and percentages), if not stated otherwise. Mean, Median, Q1, Q3, Min, Max will have the same precision as the SDTM data (decimal places). SD will be presented with one decimal place more than the mean. For subject disposition and demographic tables the denominator will be the number of subjects in the analysis set. Counts of missing observations will be included as a separate category.

Concentrations of tepotinib and its metabolites in plasma will be presented in tables and descriptively summarized by treatment and nominal time point using n, arithmetic mean, SD, standard error of the mean (SEM), median, minimum, maximum and CV%. Values below the lower limit of quantification (LLOQ) will be taken as zero for descriptive statistics of PK concentrations. Descriptive statistics of PK parameters will additionally show the geometric mean (GeoMean), the geometric coefficient of variation (GeoCV%), and the 95% CI for the GeoMean.

Graphical displays will be given, where appropriate. PK variables will be calculated and listed for all subjects who provide sufficient concentration-time data. Invalid data and their exclusion from statistical analysis will be discussed with the sponsor and flagged accordingly in the listings.

If not otherwise specified, 'baseline' refers to the last scheduled measurement before administration of the first drug in each period.

However, if a subject is missing the baseline collection, the previous non-missing evaluation could become the baseline value (e.g. from screening/admission). If no baseline or previous to baseline evaluations exist, then the baseline value will be treated as missing.

The following calculations and derivations, as applicable, will be used:

- Change from baseline: post-baseline visit value baseline value
- Duration of AE (in days hh:mm) = end date and time start date and time of the AE, if missing time for either the beginning or end then = end date start date + 1; in case of multiple records for the same AE, the duration will be calculated over all these records
- Days hh:mm from dosing = start date and time of the event date and time dose administration (for TEAEs); if missing time for either the dosing or event then = event start date date of dose administration + 1
- Rel. Day in period of AE = start date of the event date of First Admin in period + 1 (for AEs on or after the day of dosing)
- Rel. Day in trial of AE = start date of the event date of First Admin (for AEs before the day of dosing of the trial only)

Repeated and unscheduled laboratory assessments will be included and flagged as repeats in the subject data listings, but not used for summary tables statistics (unless the scheduled measurement was considered unreliable, e.g. due to technical reasons, and needed to be replaced by an unscheduled repeat measurement).

In this Phase I PK trial missing observations will be assumed to be missing completely at random (MCAR). No action will be taken to handle missing data. A subject who withdraws prior to the

last planned observation in a trial period will be included in the analyses up to the time of discontinuation.

The following treatment labels will be used:

- 5 x 100 mg TF3
- 2 x 250 mg TF3

Details of the statistical analysis will be provided in the subsequent sections.

## 10 Trial Subjects

The subsections in this section include specifications for reporting subject disposition and treatment/trial discontinuations. Additionally, procedures for reporting protocol deviations are provided.

# 10.1 Disposition of Subjects and Discontinuations

The following will be presented in a summary table:

- Total number of subjects screened (i.e. subjects who gave informed consent)
- Number of screened subjects who discontinued from the trial prior to treatment overall and grouped by the main reason for discontinuation:
  - o Subject did not meet all eligibility criteria
  - Withdrew consent
  - Adverse event
  - Lost to follow-up
  - Death
  - Other
- Number of treated subjects by treatment and overall
- Number and percentage of treated subjects who completed trial by treatment and overall
- Number and percentage of treated subjects who discontinued the trial, with the primary reason of discontinuation by treatment and overall:
  - Adverse event
  - o Lost to follow-up

- Protocol non-compliance
- Death
- Withdrew consent
- Other

A listing of discontinued subjects will be provided.

### 10.2 Protocol Deviations

## **10.2.1 Important Protocol Deviations**

Listings of important protocol deviations will be provided including the date and relative day in relation to dosing in the relevant period.

## 10.2.2 Reasons Leading to the Exclusion from an Analysis Set

All criteria/reasons leading to the exclusion of a subject from an analysis set (including clinically important protocol deviations) will be listed based on the safety set.

Reasons for excluding individual PK concentrations will also be listed separately and flagged in the main listing based on the safety analysis set.

# 11 Demographics and Other Baseline Characteristics

# 11.1 Demographics

Summaries will be given for both the safety and the PK set, if different.

Demographic characteristics will be listed by subject and summarized using the following information from the Screening/Baseline Visit electronic Case Report From (eCRF) pages.

Demographic characteristics:

- Sex: male, female
- Race: Black or African American, American Indian or Alaska Native, Asian, Native Hawaiian or Pacific Islander, White, Other
- Ethnic origin: Hispanic or Latino, Not Hispanic or Latino, Japanese, Not Japanese
- Age (years): summary statistics
- Height (cm) at Baseline: summary statistics

- Weight (kg) at Baseline: summary statistics
- BMI (kg/m²) at Baseline: summary statistics

Age will be taken from the eCRF and cannot be derived from the data because only the year of birth is collected in the eCRF.

BMI will be re-derived (i.e. not taken directly from the database) according to the following formula:

• BMI  $(kg/m^2)$  = weight (kg) / (height (m) \* height (m))

## 11.2 Medical History

The medical history will be listed by subject including the preferred term (PT) and Medical Dictionary for Regulatory Activities (MedDRA) system organ class (SOC) body term using MedDRA latest version.

## 11.3 Other Baseline Characteristics

Other baseline characteristics will be listed by subject and summarized using the following information from the Screening/Baseline Visit eCRF pages.

Other baseline characteristics:

- Smoking status
- Alcohol consumption

#### 12 Previous or Concomitant Medications/Procedures

**Previous medications** are medications, other than trial medications and pre-medications for trial drug, which started and stopped before first administration of trial drug.

Concomitant treatments are medications, other than trial medications, which are taken by subjects any time on-trial (on or after the first day of trial drug treatment for each subject).

In case the date values will not allow to unequivocally allocate a medication to previous or concomitant medication the medication will be considered as concomitant medication.

Any previous and concomitant medication will be encoded with WHO-DD, latest version. Prior and concomitant medications will be listed by subject (all subjects).

MS200095 0038 Final 1.0

The following information will be displayed in a listing: generic or trade name (as reported in CRF), WHO drug name (including ATC-2nd level and PT), dose/unit, route, frequency, reason for use, start/end date and time.

Concomitant procedures will be presented in a data listing.

## 13 Treatment Compliance and Exposure

A listing of date and time of each drug administration and each blood sampling including time deviations will be provided sorted by subject.

## 14 Efficacy Analyses

Not applicable.

# 15 Safety Analyses

The subsections in this section include specifications for summarizing safety endpoints that are common across clinical trials such as adverse events, laboratory tests and vital signs.

Safety data analysis will be conducted on the Safety Analysis Set.

## **15.1** Adverse Events

The number and percentage of subjects experiencing at least one TEAE will be summarized by treatment as well as the number of events. A TEAE is an AE with onset after start of treatment. Tables by relationship to trial drug and by severity will be generated. AEs will be coded using MedDRA terminology, latest version.

If an event was reported more than once, the worst severity will be tabulated.

Incomplete TEAE-related dates will be flagged in listings and handled as follows:

- In case the onset date is missing completely or missing partially but the onset month and year or the onset year are equal to the start of trial treatment, then the onset date will be replaced by the minimum of start of trial treatment and TEAE resolution date.
- In all other cases the missing onset day or missing onset month will be replaced by 1.
- Incomplete stop dates will be replaced by the last day of the month (if day is missing only), if not resulting in a date later than the date of subject's death. In the latter case, the date of death will be used to impute the incomplete stop date.
- In all other cases the incomplete stop date will not be imputed.

#### 15.1.1 All Adverse Events

All AEs recorded during the course of the trial (i.e. assessed from signature of informed consent until the end of the Follow-up/End of Trial visit) will be coded according to MedDRA latest version and assigned to a SOC and PT.

TEAEs will be summarized by severity, using MedDRA latest version, with PT as event category and MedDRA primary SOC body term as body system category. The severity of AEs will be graded using the "National Cancer Institute - Common Terminology Criteria for Adverse Events" (NCI-CTCAE) guideline, version 5.0 (publication date: 27 Nov 2017), as detailed in the trial protocol.

TEAEs related to trial treatment are those events with relationship missing, unknown or related.

The following will be summarized in an overview table with the number and percentage of subjects (and the number of events) by treatment and overall:

- Any TEAEs
- Any trial treatment related TEAEs
- Any serious TEAEs
- Any trial treatment related serious TEAEs
- Any TEAE (grade >=3)
- Any trial treatment related TEAEs (grade >=3)
- Any TEAEs leading to death
- Any trial treatment related TEAEs leading to death

TEAEs will be summarized by treatment and overall in tables with:

- The number and percentage of subjects by treatment with at least one TEAE and the number of events overall and by SOC and PT. Group/SOC terms will be sorted alphabetically and PTs within each group/SOC term will be sorted by descending frequency.
- The number and percentage of subjects by treatment with at least one non-serious TEAE and the number of non-serious TEAE applying frequency threshold of 5%. Group/SOC terms will be sorted alphabetically and PTs within each group/SOC term will be sorted by descending frequency.

In addition the following tables will be provided. Group/SOC terms will be sorted alphabetically and PTs within each group/SOC term will be sorted by descending frequency (based on all treatment groups combined):

- A table by severity of TEAEs with the number and percentage of subjects by treatment with at least one TEAE and the number of events by SOC and PT.
- A table by relationship to trial treatment with the number and percentage of subjects by treatment with at least one TEAE and the number of events by SOC and PT.

Pre-treatment AEs (AEs with onset after informed consent but before start of treatment) and TEAEs will be listed separately.

# 15.1.2 Adverse Events Leading to Treatment Discontinuation

TEAEs leading to permanent discontinuation of trial treatment will be summarized by treatment and overall including number of subjects, percentage and number of events.

A listing of TEAEs leading to permanent discontinuation of a trial treatment will additionally be provided.

# 15.2 Deaths, Other Serious Adverse Events, and Other Significant Adverse Events

### **15.2.1 Deaths**

All deaths as well as reason for death will be based on information from the "Report of Subject Death" CRFs.

Listing of deaths, if any, will be provided displaying date and cause of death (including TEAE leading to death and relatedness to trial treatment, when applicable), and date and time of treatment administration.

#### 15.2.2 Serious Adverse Events

A summary table of serious adverse events (SAEs), if any, by treatment and overall will be provided displaying the number and percentage of subjects by treatment with at least one SAE and the number of SAE overall and by system organ class and preferred term. Group/SOC terms and PTs within each group/SOC term will be sorted alphabetically.

Listing of SAEs, if any, will be provided in addition.

## 15.2.3 Other Significant Adverse Event

## **15.2.3.1** Adverse Events of Special Interest

Healthy subjects might experience asymptomatic elevations in serum lipase and amylase. Any elevation in serum lipase and amylase of Grade  $\geq 3$  will lead to the recording of an adverse event of special interest (AESI). The severity of these AEs should be defined based on clinical judgment of the Investigator and defined according to NCI-CTCAE Severity Scale.

AESIs will be presented in a separate data listing.

## 15.3 Clinical Laboratory Evaluation

All laboratory data will be reported with SI units. Laboratory parameters will be listed by subject and time-point and summarized indicating the treatment at the respective time-point using descriptive statistics for absolute values and change from baseline over time and by post-dose CTCAE grade shift relative to baseline. Shift tables will be based on NCI-CTCAE grades, where possible, and on normal ranges otherwise.

Shift tables will be presented for:

- End of Trial/Follow-up versus Screening
- Discharge Day 4 versus Pre-dose/Baseline (Tepotinib administration) within periods.

Laboratory values that are outside the normal range will also be flagged in the data listings, along with corresponding normal ranges and NCI-CTCAE grade. Any out-of-range values will additionally be listed separately including NCI-CTCAE grade.

See section 7.4.3 of the clinical study protocol for a table of the safety laboratory evaluations.

Safety laboratory values are separated into:

- Hematology
- Biochemistry
- Urinalysis
- Other tests

Tables will be produced for the groups Hematology and Biochemistry.

## 15.4 Vital Signs

Vital signs will be listed by subject and time-point and summarized for absolute values and changes-from-baseline (period-baseline) by visit and treatment using descriptive statistics. Descriptive statistics tables will start at baseline.

#### 15.5 ECG Evaluation

Electrocardiogram (ECG) data will be listed by subject and time-point and summarized by absolute values and changes-from-baseline (period-baseline) by treatment group using descriptive statistics. Baseline is the pre-dose assessment in each period. See section 9 for a description of how missing baseline values are handled. Descriptive statistics tables will start at baseline. Clinically significant ECG findings for individual subjects will be listed and summarized.

The time intervals (PR, QRS, RR, QT and corrected QT intervals [based on Fridericia's formula, QTcF]) will be summarized descriptively by treatment. In case of triplicate ECGs, the mean of these measurements will be considered in summary tables.

The Fridericia's Correction (QTcF) is derived as follows:

Fridericia's Correction (QTcF) 
$$QTc_f = \frac{QT}{\sqrt[3]{RR}}$$

where: RR = RR-interval measured in seconds.

QTcF values will be categorized according to their absolute values into the categories:

- $\bullet$  < 430 ms,
- $> 430 \text{ and} \le 450 \text{ ms}$ ,
- $> 450 \text{ and} \le 480 \text{ ms}$ ,
- > 480 and  $\leq$  500 ms, and
- > 500 ms.

and categorized according to their absolute change from period baseline into the categories:

- $\leq$  30 ms,
- > 30 and  $\le 60$  ms, and
- $\bullet$  > 60 ms.

MS200095 0038 Final 1.0

The number and percentage of subjects by these categories at any post-dose assessment will be tabulated by treatment group. All ECG measurements and changes from period baseline will be listed, with abnormalities (as reported of the Investigator on the ECG eCRF page) indicated.

Investigator reported interpretation results will also be tabulated by treatment using the number and percentage of subjects for each interpretation category (Normal, Abnormal Not Clinically Significant [NCS], Abnormal Clinically Significant [CS]). In case of triplicate ECGs, the worst interpretation will be considered in these frequency tables.

# 16 Analyses of Other Endpoints

#### 16.1 Pharmacokinetics

## **General Specifications for Plasma Concentration Data**

Concentrations of tepotinib and its metabolites in plasma will be presented in tables and descriptively summarized by treatment and nominal time point using number of observations (n), Mean, SD, SEM, median, Min, Max, and CV%. Descriptive statistics of PK concentration data will be calculated using values with the same precision as the source data, and rounded for reporting purposes only. The following conventions will be applied when reporting descriptive statistics of PK concentration data:

Mean, Min, Median, Max: 3 significant digits

SD, SEM: 4 significant digits

CV%: 1 decimal place

Values below the LLOQ of the assay will be taken as zero for summary statistics of PK concentration data. For final evaluations values greater than the upper limit of quantification (ULOQ) are not accepted and should be replaced by valid numeric values from dilution measurement. Missing concentrations (e.g. no sample, insufficient sample volume for analysis, no result or result not valid) will be reported and used generally as "no result" ("N.R."). Pre-dose samples that occur before the first drug administration will be assigned a time of 0 hours, as if the sample had been taken simultaneously with the study drug administration.

All available concentration data will be listed. Data of participants not in the PK analysis set or invalid data will be flagged accordingly. Any flags will be included in ADaM, respectively.

# **General Specifications for PK Parameter Data**

PK parameter data will be descriptively summarized: n, Mean, SEM, SD, CV%, Min, median, Max, geometric mean (GeoMean), the geometric coefficient of variation (GeoCV%) and the 95% confidence interval for the GeoMean (LCI 95% GM, UCI 95% GM).

MS200095\_0038 Final 1.0

PK parameter  $C_{max}$  will be reported with the same precision as the source data. All other PK parameters will be reported to 3 significant figures. In export datasets, as well as in the SDTM PP domain, PK parameters will be provided with full precision, and will not be rounded. Descriptive statistics of PK parameter data will be calculated using full precision values, and rounded for reporting purposes only.

The following conventions will be applied when reporting descriptive statistics of PK parameter data:

Mean, Min, Median, Max, GeoMean, 95% CI: 3 significant digits

SD, SEM: 4 significant digits

CV%, GeoCV%: 1 decimal place

Ratio of GeoMean and 95% CI 4 decimal places

To ensure a reliable estimate of the extent of exposure, AUC<sub>extra</sub> should be less than or equal to 20%. If AUC<sub>extra</sub> is greater than 20%, all parameters derived using  $\lambda_z$  (i.e.  $\lambda_z$ ,  $t_{1/2}$ , AUC<sub>0-\infty</sub>, AUC<sub>extra</sub>, V<sub>z</sub>/f, CL/F) will be listed, but set to missing for the calculation of descriptive statistics.

All statistical analyses and descriptive summaries of PK data will be performed on the PK Analysis Set. All available concentration/PK data will be listed. Data of subjects not in the PK Analysis Set or invalid data will be flagged accordingly. Any flags will be included in ADaM, respectively.

# **16.1.1 Primary Endpoints**

The primary endpoints will be descriptively summarized. Scatter plots will be produced for the individual PK parameters by treatment group indicating the geometric means within each treatment group.

#### **Statistical Hypotheses (Bioequivalence)**

The following null hypothesis for the ratio of the geometric means will be used to assess bioequivalence:

H<sub>0</sub>:  $\mu_T/\mu_R \le 0.8000$  or  $1.2500 \le \mu_T/\mu_R$  for at least one parameter (AUC<sub>0-t</sub> or

 $AUC_{0-\infty}$  or  $C_{max}$ )

H<sub>1</sub>:  $0.8000 < \mu_T/\mu_R < 1.2500$  for all parameters (AUC<sub>0-t</sub> and AUC<sub>0-\infty</sub> and C<sub>max</sub>)

where  $\mu_T$  and  $\mu_R$  are the geometric means for the test and reference treatment respectively.

The test treatment is 5 tablets of the 100 mg dose strength of TF3 and reference is 2 tablets of the 250 mg dose strength of TF3, both under fasting condition.

An analysis of variance (ANOVA) model with TREATMENT, PERIOD, SEQUENCE as fixed effects and SUBJECT(SEQUENCE) as random effect will be fitted to log-transformed primary endpoints  $AUC_{0-t}$ ,  $AUC_{0-\infty}$  and  $C_{max}$  based on the PK analysis set.

Treatment differences 5 x 100 mg TF3 - 2 x 250 mg TF3 under fasting condition on the log scale will be estimated for  $C_{max}$ ,  $AUC_{0-t}$ , and  $AUC_{0-\infty}$  together with their 90% CIs. Point estimates and CIs will be back-transformed to the original scale.

The null hypothesis will be rejected if the 90% CI for the ratio of the geometric mean lies within the interval 0.8000 to 1.2500 for all parameters.

## 16.1.2 Secondary Endpoints

The secondary PK endpoints will be descriptively summarized by treatment and listed.

## 16.1.3 Exploratory Endpoints

The PK endpoints  $AUC_{0-t}$ ,  $AUC_{0-\infty}$ ,  $C_{max}$ ,  $t_{max}$ ,  $t_{1/2}$  of tepotinib metabolites observed from time zero to 168 h post-dose of each period for the tepotinib metabolites MSC2571109A and MSC2571107A will be descriptively summarized by treatment and listed.

Similar analyses as for the primary endpoints will be performed for the parameters based on the metabolites of tepotinib, using 90% CIs for the comparison 5 x 100 mg TF3 - 2 x 250 mg TF3, both under fasting condition.

The ANOVA model will have the same effects as the primary analysis applied to log-transformed PK parameters  $C_{max}$ ,  $AUC_{0-t}$ , and  $AUC_{0-\infty}$ .

A mixed model with TREATMENT, PERIOD, SEQUENCE as fixed effects and SUBJECT(SEQUENCE) as random effect will be applied.

## 16.1.4 Plasma Concentration Data

The following figures will be produced for the tepotinib and metabolites (MSC2571109A and MSC2571107A) plasma concentrations:

- Arithmetic mean plasma concentration-time profiles overlaying all treatments on linear and semi-logarithmic scale
- Arithmetic mean plasma concentration-time profiles overlaying all treatments on linear scale including SD error bars
- Individual plasma concentration-time profiles overlaying subjects, for each treatment separately on linear and semi-logarithmic scale

• Individual plasma concentration-time profiles overlaying all treatments, separately for each subject on linear and semi-logarithmic scale

The following listings will be produced for the tepotinib and metabolites plasma concentrations:

• Plasma concentrations will be listed by nominal time by treatment. Excluded plasma concentrations will be flagged.

## 16.1.5 Estimation of Individual Pharmacokinetic Parameters

The following non-compartmental PK parameters (see will be calculated from the individual plasma total tepotinib and metabolites concentration-time data using commercial software such as Phoenix®/WinNonlin® (Version 6.4 or higher) at Nuvisan GmbH.

Table 1 Definition of PK Parameters for Tepotinib and its Metabolites After Single Dose Administration

| Symbol | Definition |
|---|---|
| AUC <sub>0-t</sub> | Area under the plasma concentration-time curve (AUC) from time zero (= dosing time) to the last sampling time (t <sub>last</sub> ) at which the concentration is at or above the lower limit of quantification (LLOQ), calculated using the mixed log linear trapezoidal rule (ie linear up/log down) |
| AUC <sub>0-t</sub> /D | AUC <sub>0-t</sub> divided by dose |
| AUC <sub>0-24</sub> | AUC from 0 to 24 hours, calculated using mixed log linear trapezoidal rule (linear up, log down) |
| $AUC_{0-24}/D$ | AUC <sub>0-24</sub> divided by dose |
| $\mathrm{AUC}_{0\text{-}\infty}$ | AUC from time zero (= dosing time) extrapolated to infinity, calculated as $AUC_{0\text{-t}} + AUC_{extra}$ . $AUC_{extra}$ represents the extrapolated part of $AUC_{0\text{-}\infty}$ calculated by $C_{lastpred}/\lambda_z$ , where $C_{lastpred}$ is the predicted plasma concentration at the last sampling time point, calculated from the log-linear regression line for $\lambda_z$ determination at which the measured plasma concentration is at or above LLOQ |
| $AUC_{0-\infty}/D$ | AUC₀-∞ divided by dose |
| $C_{\text{max}}$ | Maximum plasma concentration observed |
| C <sub>max</sub> /D | C <sub>max</sub> divided by dose |

MS200095 0038 Final 1.0

| Symbol | Definition |
|---|---|
| t <sub>last</sub> | The last sampling time at which the plasma concentration is at or above the lower limit of quantification |
| $t_{max}$ | Time to reach the maximum observed plasma concentration |
| $t_{1/2}$ | Terminal half-life, calculated as $ln(2)/\lambda_z$ |
| $\lambda_{z}$ | Terminal rate constant determined from the terminal slope of<br>the log-transformed plasma concentration curve using linear<br>regression on terminal data points of the curve |
| CL/F | Apparent total body clearance of drug from plasma following extravascular administration, calculated as dose/AUC $_{0-\infty}$ |
| $V_z/f$ | Apparent volume of distribution during the terminal phase following extravascular administration |
| AUC <sub>extra</sub> | The AUC from time t <sub>last</sub> extrapolated to infinity |
| AUC <sub>extra</sub> % | $AUC_{extra} / AUC_{0-\infty} x 100.$ |

Individual PK parameters will be calculated using actual sampling times. If the actual sampling time is missing, then the nominal sampling times will be used instead. The pre-dose sample will be considered as if it had been taken simultaneously with the administration of study drug. PK variables will be evaluated and listed for all subjects who provide sufficient concentration-time data.

Plasma concentrations below LLOQ willbe taken as zero for calculating the AUC. Plasma concentrations below LLOQ after the last quantifiable data point will not be considered for the determination of  $\lambda_z$ .

The following PK parameters will be calculated for diagnostic purposes and listed, but will not be summarized:

- The time interval (h) of the log-linear regression ( $\lambda_{z \text{ low}}$ ,  $\lambda_{z \text{ upp}}$ ) to determine  $\lambda_{z}$ .
- Number of data points included in the log-linear regression analysis to determine  $\lambda_z$ .
- Goodness of fit statistic (Rsq) for calculation of  $\lambda_z$ .

The regression analysis should contain data from at least 3 different time points in the terminal phase consistent with the assessment of a straight line on the log-transformed scale. Phoenix WinNonlin best fit methodology will be used as standard. The last quantifiable concentration

should always be included in the regression analysis, while the concentration at  $t_{max}$  and any <LLOQ concentrations that occur after the last quantifiable data point should not be used.

The coefficient of correlation ( $R^2$ ) should be  $\geq 0.8$  and the observation period over which the regression line is estimated should be at least twofold the resulting  $t_{1/2}$  itself. If these criteria are not met, then the corresponding values should be flagged in the listing displaying Individual Plasma Pharmacokinetic Diagnostic Parameters for Each Treatment. Any flags should be included in the study specific SDTM/ADaM. Then the rate constants and all derived parameters (e.g.  $AUC_{0-\infty}$ , % $AUC_{extra}$ , CL/f,  $t_{1/2}$ , and  $V_Z/f$ ) will be included in the parameter listings and will be discussed appropriately in alignment with the protocol lead and quantitative pharmacology representative.

The following interpolation or extrapolation rules apply when calculating AUC<sub>0-24</sub>:

- If the time point 24 hours falls within the time range in which samples were taken, but does not coincide with an observed data point, then a linear interpolation is performed to estimate the corresponding concentration value.
- If the time point 24 hours occurs after the last measurable concentration and the terminal regression ( $\lambda_z$ ) is estimable, then  $\lambda_z$  is used to estimate the concentration at time 24 hours. If  $\lambda_z$  cannot be estimated the partial area will not be calculated.

The IMP dose administered is given for the monohydrate hydrochloride salt (i.e. 500 mg IMP). A conversion factor for the freebase IMP was calculated and will be applied when 'dose' is used in deriving PK parameter formulas needing a dose value (CL/f).

Conversion factor = Molecular weight (MW) of base IMP divided by MW of salt form IMP = 492.574 g/mol / 547.05 g/mol = 0.9004

Amount of dose \* conversion factor = actual dose of IMP: 500 mg \* 0.9004 = 450 mg

The Phoenix WinNonlin NCA Core Output will be provided in a separate listing.

# 16.2 Pharmacogenetics

Pharmacogenetic sampling is mandatory for trial participation. An additional separate ICF will be used. One blood sample should be collected in duplicate on Day -1 of the first treatment period prior to administration. The pharmacogenetic samples will be analyzed conditionally in case of unexpected PK profiles. The results of the PGx analysis, as applicable, will be described in a separate report.

Tepotinib (MSC2156119J) Bioequivalence of 5 tablets of 100 mg vs 2 tablets of 250 mg TF3 of tepotinib

MS200095\_0038 Final 1.0

17 References

N.A.

18 Appendices

None.

| 16. | .1.9.2: Statistical Analysis Output | 2 |
|---|---|---|
| | Listing 16.1.9.2.1: Statistical Output of Primary Analysis | 3 |
| | Listing 16.1.9.2.2: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571109A | 21 |
| | Listing 16.1.9.2.3: Statistical Output of Exploratory Analysis - Tepotinib | 30 |

16.1.9.2: Statistical Analysis Output

16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.1: Statistical Output of Primary Analysis

Parameter: AUCO-inf (h\*ng/mL) for Tepotinib

The Mixed Procedure

Model Information

Data Set WORK.PKPARS Dependent Variable LOGAVAL

Covariance Structure Variance Components

Estimation Method REML Residual Variance Method Profile Model-Based Fixed Effects SE Method Degrees of Freedom Method Containment

Class Level Information

Class Levels Values TRTA1 RТ 2 1 2 APERTOD

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.12; SDTM package: 15JAN2020

Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-prim-anova.sas, 28JAN2020 12:59 

16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.1: Statistical Output of Primary Analysis

Parameter: AUCO-inf (h\*ng/mL) for Tepotinib

The Mixed Procedure

Class Level Information

Class Levels Values
USUBJID 18

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.12; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-prim-anova.sas, 28JAN2020 12:59


\_\_\_\_\_\_

16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.1: Statistical Output of Primary Analysis

Parameter: AUCO-inf (h\*ng/mL) for Tepotinib

The Mixed Procedure

Class Level Information

Class Levels Values

SEQUENCE 2 RT TR

Dimensions

Covariance Parameters 2
Columns in X 7
Columns in Z 18
Subjects 1
Max Obs Per Subject 35

Number of Observations

Number of Observations Read 35 Number of Observations Used 35 Number of Observations Not Used 0

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.12; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-prim-anova.sas, 28JAN2020 12:59


16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.1: Statistical Output of Primary Analysis

Parameter: AUCO-inf (h\*ng/mL) for Tepotinib

The Mixed Procedure

Iteration History

| Iteration | Evaluations | -2 Res Log Like | Criterion |
|-----------|-------------|-----------------|------------|
| 0 | 1 | 27.82729226 | |
| 1 | 2 | 14.18487139 | 0.00009191 |
| 2 | 1 | 14.18286276 | 0.00000010 |
| 3 | 1 | 14.18286061 | 0.00000000 |

Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Estimate

USUBJID(SEQUENCE) 0.08236
Residual 0.02311

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.12; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-prim-anova.sas, 28JAN2020 12:59


#### 16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.1: Statistical Output of Primary Analysis

Parameter: AUCO-inf (h\*ng/mL) for Tepotinib

The Mixed Procedure

Fit Statistics

| -2 Res Log Likelihood | 14.2 |
|--------------------------|------|
| AIC (smaller is better) | 18.2 |
| AICC (smaller is better) | 18.6 |
| BIC (smaller is better) | 20.0 |

Type 3 Tests of Fixed Effects

| | Num | Den | | |
|----------|-----|-----|---------|--------|
| Effect | DF | DF | F Value | Pr > F |
| TRTA1 | 1 | 15 | 3.34 | 0.0875 |
| APERIOD | 1 | 15 | 5.68 | 0.0308 |
| SEQUENCE | 1 | 16 | 1.42 | 0.2502 |

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.12; SDTM package: 15JAN2020

Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-prim-anova.sas, 28JAN2020 12:59 

16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.1: Statistical Output of Primary Analysis

Parameter: AUCO-inf (h\*ng/mL) for Tepotinib

The Mixed Procedure

Least Squares Means

| Effect | TRTA1 | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper | |
|---|---|---|---|---|---|---|---|---|---|---|
| TRTA1<br>TRTA1 | R<br>T | 9.7527<br>9.6576 | 0.07654<br>0.07747 | 15<br>15 | 127.41<br>124.66 | <.0001<br><.0001 | 0.1 | 9.6186<br>9.5218 | 9.8869<br>9.7934 | |
| Differences of Least Squares Means | | | | | | | | | | |
| Effect | TRTA1 | _TRTA1 | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| TRTA1 | Т | R | -0.09516 | 0.05206 | 15 | -1.83 | 0.0875 | 0.1 | -0.1864 | -0.00390 |

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.12; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-prim-anova.sas, 28JAN2020 12:59


\_\_\_\_\_

16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.1: Statistical Output of Primary Analysis

Parameter: AUCO-t (h\*ng/mL) for Tepotinib

The Mixed Procedure

Model Information

Data Set WORK.PKPARS
Dependent Variable LOGAVAL

Covariance Structure Variance Components

Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Containment

Class Level Information

Class Levels Values
TRTA1 2 R T
APERIOD 2 1 2

\_\_\_\_\_

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.12; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-prim-anova.sas, 28JAN2020 12:59


16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Levels Values

Listing 16.1.9.2.1: Statistical Output of Primary Analysis

Parameter: AUCO-t (h\*ng/mL) for Tepotinib

The Mixed Procedure

Class

Class Level Information

USUBJID 18 PI

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.12; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-prim-anova.sas, 28JAN2020 12:59


\_\_\_\_\_

16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.1: Statistical Output of Primary Analysis

Parameter: AUCO-t (h\*ng/mL) for Tepotinib

The Mixed Procedure

Class Level Information

Class Levels Values

SEQUENCE 2 RT TR

Dimensions

Covariance Parameters 2
Columns in X 7
Columns in Z 18
Subjects 1
Max Obs Per Subject 35

Number of Observations

Number of Observations Read 35 Number of Observations Used 35 Number of Observations Not Used 0

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.12; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-prim-anova.sas, 28JAN2020 12:59


16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.1: Statistical Output of Primary Analysis

Parameter: AUCO-t (h\*ng/mL) for Tepotinib

The Mixed Procedure

Iteration History

| Iteration | Evaluations | -2 Res Log Like | Criterion |
|-----------|-------------|-----------------|------------|
| 0 | 1 | 26.34579623 | |
| 1 | 2 | 13.26462856 | 0.00006316 |
| 2 | 1 | 13.26322330 | 0.0000005 |
| 3 | 1 | 13.26322224 | 0.00000000 |

Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Estimate

USUBJID(SEQUENCE) 0.07738

Residual 0.02303

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.12; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-prim-anova.sas, 28JAN2020 12:59


# 16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.1: Statistical Output of Primary Analysis

Parameter: AUCO-t (h\*ng/mL) for Tepotinib

The Mixed Procedure

Fit Statistics

| -2 Res Log Likelihood | 13.3 |
|--------------------------|------|
| AIC (smaller is better) | 17.3 |
| AICC (smaller is better) | 17.7 |
| BIC (smaller is better) | 19.0 |

Type 3 Tests of Fixed Effects

| | Num | Den | | |
|----------|-----|-----|---------|--------|
| Effect | DF | DF | F Value | Pr > F |
| TRTA1 | 1 | 15 | 3.18 | 0.0947 |
| APERIOD | 1 | 15 | 6.09 | 0.0261 |
| SEQUENCE | 1 | 16 | 1.40 | 0.2546 |

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.12; SDTM package: 15JAN2020

Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-prim-anova.sas, 28JAN2020 12:59


16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.1: Statistical Output of Primary Analysis

Parameter: AUCO-t (h\*ng/mL) for Tepotinib

The Mixed Procedure

Least Squares Means

| Effect | TRTA1 | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper | |
|---|---|---|---|---|---|---|---|---|---|---|
| TRTA1<br>TRTA1 | R<br>T | 9.7125<br>9.6198 | 0.07469<br>0.07563 | 15<br>15 | 130.04<br>127.19 | <.0001<br><.0001 | 0.1<br>0.1 | 9.5816<br>9.4872 | 9.8434<br>9.7524 | |
| | | | | Difference | s of Least | . Squares Me | eans | | | |
| Effect | TRTA1 | _TRTA1 | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| TRTA1 | Т | R | -0.09269 | 0.05197 | 15 | -1.78 | 0.0947 | 0.1 | -0.1838 | -0.00159 |

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.12; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-prim-anova.sas, 28JAN2020 12:59


16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.1: Statistical Output of Primary Analysis

Parameter: Cmax (ng/mL) for Tepotinib

The Mixed Procedure

Model Information

Data Set WORK.PKPARS
Dependent Variable LOGAVAL

Covariance Structure Variance Components

Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Containment

Class Level Information

Class Levels Values
TRTA1 2 R T
APERIOD 2 1 2

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.12; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-prim-anova.sas, 28JAN2020 12:59


16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.1: Statistical Output of Primary Analysis

Parameter: Cmax (ng/mL) for Tepotinib

The Mixed Procedure

Class Level Information



T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.12; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-prim-anova.sas, 28JAN2020 12:59


16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.1: Statistical Output of Primary Analysis

Parameter: Cmax (ng/mL) for Tepotinib

The Mixed Procedure

Class Level Information

Class Levels Values

SEQUENCE 2 RT TR

Dimensions

Covariance Parameters 2
Columns in X 7
Columns in Z 18
Subjects 1
Max Obs Per Subject 36

Number of Observations

Number of Observations Read 36
Number of Observations Used 36
Number of Observations Not Used 0

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.12; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-prim-anova.sas, 28JAN2020 12:59


16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.1: Statistical Output of Primary Analysis

Parameter: Cmax (ng/mL) for Tepotinib

The Mixed Procedure

Iteration History

| Iteration | Evaluations | -2 Res Log Like | Criterion |
|-----------|-------------|-----------------|-----------|

1

7.31480767 2.58411332 0.00000000

Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Estimate

USUBJID (SEQUENCE) 0.02709 Residual 0.02645

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.12; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-prim-anova.sas, 28JAN2020 12:59


# 16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.1: Statistical Output of Primary Analysis

Parameter: Cmax (ng/mL) for Tepotinib

The Mixed Procedure

Fit Statistics

| -2 Res Log Likelihood | 2.6 |
|--------------------------|-----|
| AIC (smaller is better) | 6.6 |
| AICC (smaller is better) | 7.0 |
| BIC (smaller is better) | 8.4 |

Type 3 Tests of Fixed Effects

| | Num | Den | | |
|----------|-----|-----|---------|--------|
| Effect | DF | DF | F Value | Pr > F |
| TRTA1 | 1 | 16 | 0.69 | 0.4173 |
| APERIOD | 1 | 16 | 3.61 | 0.0754 |
| SEQUENCE | 1 | 16 | 0.38 | 0.5462 |

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.12; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-prim-anova.sas, 28JAN2020 12:59


16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.1: Statistical Output of Primary Analysis

Parameter: Cmax (ng/mL) for Tepotinib

The Mixed Procedure

Least Squares Means

| Effect | TRTA1 | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper | |
|---|---|---|---|---|---|---|---|---|---|---|
| TRTA1<br>TRTA1 | R<br>T | 5.4826<br>5.5277 | 0.05454<br>0.05454 | 16<br>16 | 100.52<br>101.35 | <.0001<br><.0001 | 0.1 | 5.3874<br>5.4325 | 5.5778<br>5.6230 | |
| | | | | Difference | s of Least | . Squares Me | ans | | | |
| Effect | TRTA1 | _TRTA1 | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| TRTA1 | Т | R | 0.04515 | 0.05422 | 16 | 0.83 | 0.4173 | 0.1 | -0.04951 | 0.1398 |

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.12; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-prim-anova.sas, 28JAN2020 12:59


16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.2: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571109A

Parameter: AUCO-inf (h\*ng/mL) for Metabolite MSC2571109A

The Mixed Procedure

Model Information

Data Set WORK.PKPARS Dependent Variable LOGAVAL

Covariance Structure Variance Components

Estimation Method REML Residual Variance Method Profile Fixed Effects SE Method Model-Based Degrees of Freedom Method Containment

Class Level Information

Class Levels Values TRTA1 R T 2 1 2 APERTOD

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3


Source: ADPP 22JAN2020 13:55; Listing 16.2.5.13; SDTM package: 15JAN2020

Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-expl-anova.sas, 28JAN2020 13:02

Page 47 of 331

16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.2: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571109A

Parameter: AUCO-inf (h\*ng/mL) for Metabolite MSC2571109A

The Mixed Procedure

Class Level Information

Class Levels Values

USUBJID 18



T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.13; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-expl-anova.sas, 28JAN2020 13:02


\_\_\_\_\_

## 16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.2: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571109A

Parameter: AUCO-inf (h\*ng/mL) for Metabolite MSC2571109A

The Mixed Procedure

Class Level Information

Class Levels Values

SEQUENCE 2 RT TR

Dimensions

Covariance Parameters 2
Columns in X 7
Columns in Z 18
Subjects 1
Max Obs Per Subject 35

Number of Observations

Number of Observations Read 35 Number of Observations Used 34 Number of Observations Not Used 1

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.13; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-expl-anova.sas, 28JAN2020 13:02


16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.2: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571109A

Parameter: AUCO-inf (h\*ng/mL) for Metabolite MSC2571109A

The Mixed Procedure

Iteration History

| Iteration | Evaluations | -2 Res Log Like | Criterion |
|-----------|-------------|-----------------|------------|
| 0 | 1 | 31.53030633 | |
| 1 | 2 | 16.76697914 | 0.00007090 |
| 2 | 1 | 16.76559433 | 0.0000005 |
| 3 | 1 | 16.76559328 | 0.0000000 |

Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Estimate

USUBJID(SEQUENCE) 0.09898

Residual 0.02278

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.13; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-expl-anova.sas, 28JAN2020 13:02


\_\_\_\_\_

- 16.1: Study Information
- 16.1.9: Documentation of Statistical Methods
- 16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.2: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571109A

Parameter: AUCO-inf (h\*ng/mL) for Metabolite MSC2571109A

The Mixed Procedure

Fit Statistics

| -2 Res Log Likelihood | 16.8 |
|--------------------------|------|
| AIC (smaller is better) | 20.8 |
| AICC (smaller is better) | 21.2 |
| BIC (smaller is better) | 22.5 |

Type 3 Tests of Fixed Effects

| | Num | Den | | |
|----------|-----|-----|---------|--------|
| Effect | DF | DF | F Value | Pr > F |
| TRTA1 | 1 | 14 | 2.11 | 0.1685 |
| APERIOD | 1 | 14 | 3.75 | 0.0731 |
| SEQUENCE | 1 | 16 | 0.71 | 0.4120 |

F = 100 mm HTQ = P = 2 mm HTQ

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.13; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-expl-anova.sas, 28JAN2020 13:02


16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.2: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571109A

Parameter: AUCO-inf (h\*ng/mL) for Metabolite MSC2571109A

The Mixed Procedure

Least Squares Means

| Effect | TRTA1 | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper | |
|---|---|---|---|---|---|---|---|---|---|---|
| TRTA1<br>TRTA1 | R<br>T | 9.3035<br>9.2264 | 0.08311 | 14<br>14 | 111.94<br>111.01 | <.0001<br><.0001 | 0.1 | 9.1571<br>9.0801 | 9.4499<br>9.3728 | |
| 11(1111 | 1 | J. 2201 | 0.00311 | 11 | 111.01 | 1.0001 | 0.1 | J.0001 | 3.3720 | |
| | | | | Difference | s of Least | Squares Me | eans | | | |
| Effect | TRTA1 | _TRTA1 | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| TRTA1 | Т | R | -0.07708 | 0.05308 | 14 | -1.45 | 0.1685 | 0.1 | -0.1706 | 0.01641 |

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.13; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-expl-anova.sas, 28JAN2020 13:02


\_\_\_\_\_

16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.2: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571109A

Parameter: AUCO-t (h\*ng/mL) for Metabolite MSC2571109A

The Mixed Procedure

Model Information

Data Set WORK.PKPARS
Dependent Variable LOGAVAL

Covariance Structure Variance Components

Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Containment

Class Level Information

Class Levels Values
TRTA1 2 R T
APERIOD 2 1 2

\_\_\_\_\_

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.13; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-expl-anova.sas, 28JAN2020 13:02


16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.2: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571109A

Parameter: AUCO-t (h\*ng/mL) for Metabolite MSC2571109A

The Mixed Procedure

Class Level Information

Class Levels Values
USUBJID 18

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.13; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-expl-anova.sas, 28JAN2020 13:02


\_\_\_\_\_

## 16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.2: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571109A

Parameter: AUCO-t (h\*ng/mL) for Metabolite MSC2571109A

The Mixed Procedure

Class Level Information

Class Levels Values

SEQUENCE 2 RT TR

Dimensions

Covariance Parameters 2
Columns in X 7
Columns in Z 18
Subjects 1
Max Obs Per Subject 35

Number of Observations

Number of Observations Read 35
Number of Observations Used 35
Number of Observations Not Used 0

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.13; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-expl-anova.sas, 28JAN2020 13:02


16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.2: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571109A

Parameter: AUCO-t (h\*ng/mL) for Metabolite MSC2571109A

The Mixed Procedure

Iteration History

| Iteration | Evaluations | -2 Res Log Like | Criterion |
|-----------|-------------|-----------------|------------|
| 0 | 1 | 26.81517413 | |
| 1 | 2 | 11.88675358 | 0.00035958 |
| 2 | 1 | 11.87830803 | 0.00000157 |
| 3 | 1 | 11.87827247 | 0.00000000 |

Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Estimate
USUBJID(SEQUENCE) 0.08272
Residual 0.02009

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.13; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-expl-anova.sas, 28JAN2020 13:02


\_\_\_\_\_

- 16.1: Study Information
- 16.1.9: Documentation of Statistical Methods
- 16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.2: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571109A

Parameter: AUCO-t (h\*ng/mL) for Metabolite MSC2571109A

The Mixed Procedure

Fit Statistics

| -2 Res Log Likelihood | 11.9 |
|--------------------------|------|
| AIC (smaller is better) | 15.9 |
| AICC (smaller is better) | 16.3 |
| BIC (smaller is better) | 17. |

Type 3 Tests of Fixed Effects

| | Num | Den | | |
|----------|-----|-----|---------|--------|
| Effect | DF | DF | F Value | Pr > F |
| TRTA1 | 1 | 15 | 2.29 | 0.1511 |
| APERIOD | 1 | 15 | 4.59 | 0.0491 |
| SEQUENCE | 1 | 16 | 0.68 | 0.4226 |

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.13; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-expl-anova.sas, 28JAN2020 13:02


16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.2: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571109A

Parameter: AUCO-t (h\*ng/mL) for Metabolite MSC2571109A

The Mixed Procedure

Least Squares Means

| Effect | TRTA1 | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper | |
|---|---|---|---|---|---|---|---|---|---|---|
| TRTA1<br>TRTA1 | R<br>T | 9.2341<br>9.1606 | 0.07558<br>0.07641 | 15<br>15 | 122.18<br>119.90 | <.0001<br><.0001 | 0.1<br>0.1 | 9.1016<br>9.0267 | 9.3666<br>9.2946 | |
| | | | | Di fifanan aa | <del>-</del> | Camana Ma | | | | |
| | | | | Standard | s of Least | : Squares Me | ans | | | |
| Effect | TRTA1 | _TRTA1 | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| TRTA1 | Т | R | -0.07348 | 0.04856 | 15 | -1.51 | 0.1511 | 0.1 | -0.1586 | 0.01166 |

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.13; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-expl-anova.sas, 28JAN2020 13:02


16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.2: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571109A

Parameter: Cmax (ng/mL) for Metabolite MSC2571109A

The Mixed Procedure

Model Information

Data Set WORK.PKPARS Dependent Variable LOGAVAL

Covariance Structure Variance Components

Estimation Method REML Residual Variance Method Profile Fixed Effects SE Method Model-Based Degrees of Freedom Method Containment

2 1 2

Class Level Information

Class Levels Values TRTA1 R T

APERTOD

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.13; SDTM package: 15JAN2020

Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-expl-anova.sas, 28JAN2020 13:02 

16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.2: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571109A

Parameter: Cmax (ng/mL) for Metabolite MSC2571109A

The Mixed Procedure

Class Level Information

Class Levels Values
USUBJID 18

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.13; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-expl-anova.sas, 28JAN2020 13:02


\_\_\_\_\_

### 16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.2: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571109A

Parameter: Cmax (ng/mL) for Metabolite MSC2571109A

The Mixed Procedure

Class Level Information

Class Levels Values

SEQUENCE 2 RT TR

Dimensions

Covariance Parameters 2
Columns in X 7
Columns in Z 18
Subjects 1
Max Obs Per Subject 36

Number of Observations

Number of Observations Read 36
Number of Observations Used 36
Number of Observations Not Used 0

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.13; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-expl-anova.sas, 28JAN2020 13:02


16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.2: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571109A

Parameter: Cmax (ng/mL) for Metabolite MSC2571109A

The Mixed Procedure

Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 15.17122702

1 6.48385334 0.00000000

Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Estimate

USUBJID(SEQUENCE) 0.04430 Residual 0.02414

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.13; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-expl-anova.sas, 28JAN2020 13:02


- 16.1: Study Information
- 16.1.9: Documentation of Statistical Methods
- 16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.2: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571109A

Parameter: Cmax (ng/mL) for Metabolite MSC2571109A

The Mixed Procedure

Fit Statistics

| -2 Res Log Likelihood | 6.5 |
|--------------------------|------|
| AIC (smaller is better) | 10.5 |
| AICC (smaller is better) | 10.9 |
| BIC (smaller is better) | 12.3 |

Type 3 Tests of Fixed Effects

| | Num | Den | | |
|----------|-----|-----|---------|--------|
| Effect | DF | DF | F Value | Pr > F |
| TRTA1 | 1 | 16 | 0.19 | 0.6704 |
| APERIOD | 1 | 16 | 4.23 | 0.0563 |
| SEQUENCE | 1 | 16 | 0.33 | 0.5736 |

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.13; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-expl-anova.sas, 28JAN2020 13:02


16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.2: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571109A

Parameter: Cmax (ng/mL) for Metabolite MSC2571109A

The Mixed Procedure

#### Least Squares Means

| Effect | TRTA1 | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | - | | | |
| TRTA1 | R | 4.7859 | 0.06166 | 16 | 77.61 | <.0001 | 0.1 | 4.6782 | 4.8935 | |
| TRTA1 | T | 4.7634 | 0.06166 | 16 | 77.25 | <.0001 | 0.1 | 4.6558 | 4.8711 | |
| Differences of Least Squares Means | | | | | | | | | | |
| | | | | Standard | | | | | | |
| Effect | TRTA1 | _TRTA1 | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| TRTA1 | Т | R | -0.02246 | 0.05179 | 16 | -0.43 | 0.6704 | 0.1 | -0.1129 | 0.06796 |

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.13; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-expl-anova.sas, 28JAN2020 13:02


16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.3: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571107A

Parameter: AUCO-inf (h\*ng/mL) for Metabolite MSC2571107A

The Mixed Procedure

Model Information

Data Set WORK.PKPARS Dependent Variable LOGAVAL

Covariance Structure Variance Components

Estimation Method REML Residual Variance Method Profile Fixed Effects SE Method Model-Based Degrees of Freedom Method Containment

Class Level Information

Class Levels Values TRTA1 R T 2 1 2 APERTOD

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.14; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-expl-anova.sas, 28JAN2020 13:02


16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.3: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571107A

Parameter: AUCO-inf (h\*ng/mL) for Metabolite MSC2571107A

The Mixed Procedure

Class Level Information

Class Levels Values
USUBJID 18

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.14; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-expl-anova.sas, 28JAN2020 13:02


\_\_\_\_\_\_

16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.3: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571107A

Parameter: AUCO-inf (h\*ng/mL) for Metabolite MSC2571107A

The Mixed Procedure

Class Level Information

Class Levels Values

SEQUENCE 2 RT TR

Dimensions

Covariance Parameters 2
Columns in X 7
Columns in Z 18
Subjects 1
Max Obs Per Subject 35

Number of Observations

Number of Observations Read 35 Number of Observations Used 34 Number of Observations Not Used 1

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.14; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-expl-anova.sas, 28JAN2020 13:02


16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.3: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571107A

Parameter: AUCO-inf (h\*ng/mL) for Metabolite MSC2571107A

The Mixed Procedure

Iteration History

| Iteration | Evaluations | -2 Res Log Like | Criterion |
|-----------|-------------|-----------------|------------|
| 0 | 1 | 39.33425405 | |
| 1 | 3 | 22.75268267 | 0.00020766 |
| 2 | 1 | 22.74922662 | 0.00000039 |
| 3 | 1 | 22.74922033 | 0.0000000 |

Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Estimate

USUBJID(SEQUENCE) 0.1279

Residual 0.02641

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.14; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-expl-anova.sas, 28JAN2020 13:02


# 16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.3: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571107A

Parameter: AUCO-inf (h\*ng/mL) for Metabolite MSC2571107A

The Mixed Procedure

Fit Statistics

| -2 Res Log Likelihood | 22. |
|--------------------------|------|
| AIC (smaller is better) | 26. |
| AICC (smaller is better) | 27.2 |
| BIC (smaller is better) | 28.5 |

Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|----------|-----------|-----------|---------|--------|
| TRTA1 | 1 | 14 | 1.97 | 0.1821 |
| APERIOD | 1 | 14 | 3.43 | 0.0854 |
| SEOUENCE | 1 | 16 | 1.19 | 0.2917 |

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.14; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-expl-anova.sas, 28JAN2020 13:02


16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.3: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571107A

Parameter: AUCO-inf (h\*ng/mL) for Metabolite MSC2571107A

The Mixed Procedure

Least Squares Means

| | | | Standard | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Effect | TRTA1 | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper | |
| TRTA1 | R | 6.5721 | 0.09348 | 14 | 70.30 | <.0001 | 0.1 | 6.4074 | 6.7367 | |
| TRTA1 | T | 6.4918 | 0.09348 | 14 | 69.44 | <.0001 | 0.1 | 6.3271 | 6.6564 | |
| | | | | Difference | s of Least | Squares Me | ans | | | |
| | | | | Standard | | | | | | |
| Effect | TRTA1 | _TRTA1 | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| TRTA1 | Т | R | -0.08030 | 0.05719 | 14 | -1.40 | 0.1821 | 0.1 | -0.1810 | 0.02042 |

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.14; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-expl-anova.sas, 28JAN2020 13:02


16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.3: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571107A

Parameter: AUCO-t (h\*ng/mL) for Metabolite MSC2571107A

The Mixed Procedure

Model Information

Data Set WORK.PKPARS Dependent Variable LOGAVAL

Covariance Structure Variance Components

Estimation Method REML Residual Variance Method Profile Fixed Effects SE Method Model-Based Degrees of Freedom Method Containment

Class Level Information

Class Levels Values TRTA1 R T 2 1 2 APERTOD

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.14; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-expl-anova.sas, 28JAN2020 13:02


16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.3: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571107A

Parameter: AUCO-t (h\*ng/mL) for Metabolite MSC2571107A

The Mixed Procedure

Class Level Information

Class Levels Values
USUBJID 18

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.14; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-expl-anova.sas, 28JAN2020 13:02


\_\_\_\_\_\_

## 16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.3: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571107A

Parameter: AUCO-t (h\*ng/mL) for Metabolite MSC2571107A

The Mixed Procedure

Class Level Information

Class Levels Values

SEQUENCE 2 RT TR

Dimensions

Covariance Parameters 2
Columns in X 7
Columns in Z 18
Subjects 1
Max Obs Per Subject 35

Number of Observations

Number of Observations Read 35 Number of Observations Used 35 Number of Observations Not Used 0

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.14; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-expl-anova.sas, 28JAN2020 13:02


16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.3: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571107A

Parameter: AUCO-t (h\*ng/mL) for Metabolite MSC2571107A

The Mixed Procedure

Iteration History

| Iteration | Evaluations | -2 Res Log Like | Criterion |
|-----------|-------------|-----------------|------------|
| 0 | 1 | 35.34606855 | |
| 1 | 2 | 18.61144132 | 0.00000217 |
| 2 | 1 | 18.61139966 | 0.00000000 |

Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Estimate
USUBJID(SEQUENCE) 0.1093
Residual 0.02369

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.14; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-expl-anova.sas, 28JAN2020 13:02


## 16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.3: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571107A

Parameter: AUCO-t (h\*ng/mL) for Metabolite MSC2571107A

The Mixed Procedure

Fit Statistics

| -2 Res Log Likelihood | 18.6 |
|--------------------------|------|
| AIC (smaller is better) | 22.6 |
| AICC (smaller is better) | 23.0 |
| BIC (smaller is better) | 24.4 |

Type 3 Tests of Fixed Effects

| | Num | Den | | |
|----------|-----|-----|---------|--------|
| Effect | DF | DF | F Value | Pr > F |
| TRTA1 | 1 | 15 | 2.60 | 0.1276 |
| APERIOD | 1 | 15 | 4.91 | 0.0425 |
| SEQUENCE | 1 | 16 | 1.38 | 0.2571 |

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.14; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-expl-anova.sas, 28JAN2020 13:02


16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.3: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571107A

Parameter: AUCO-t (h\*ng/mL) for Metabolite MSC2571107A

The Mixed Procedure

Least Squares Means

| Effect | TRTA1 | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper | |
|---|---|---|---|---|---|---|---|---|---|---|
| TRTA1<br>TRTA1 | R<br>T | 6.5079<br>6.4228 | 0.08596<br>0.08683 | 15<br>15 | 75.71<br>73.97 | <.0001<br><.0001 | 0.1 | 6.3572<br>6.2706 | 6.6586<br>6.5751 | |
| | | | | Difference | s of Least | Squares Me | ans | | | |
| Effect | TRTA1 | _TRTA1 | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| TRTA1 | Т | R | -0.08507 | 0.05274 | 15 | -1.61 | 0.1276 | 0.1 | -0.1775 | 0.007396 |

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.14; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-expl-anova.sas, 28JAN2020 13:02


\_\_\_\_\_

16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.3: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571107A

Parameter: Cmax (ng/mL) for Metabolite MSC2571107A

The Mixed Procedure

Model Information

Data Set WORK.PKPARS
Dependent Variable LOGAVAL

Covariance Structure Variance Components

Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Containment

Class Level Information

Class Levels Values
TRTA1 2 R T
APERIOD 2 1 2

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.14; SDTM package: 15JAN2020

Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-expl-anova.sas, 28JAN2020 13:02


16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.3: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571107A

Parameter: Cmax (ng/mL) for Metabolite MSC2571107A

The Mixed Procedure

Class Level Information

Class Levels Values

USUBJID 18



T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.14; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-expl-anova.sas, 28JAN2020 13:02


### 16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.3: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571107A

Parameter: Cmax (ng/mL) for Metabolite MSC2571107A

The Mixed Procedure

Class Level Information

Class Levels Values

SEQUENCE 2 RT TR

Dimensions

Covariance Parameters 2
Columns in X 7
Columns in Z 18
Subjects 1
Max Obs Per Subject 36

Number of Observations

Number of Observations Read 36
Number of Observations Used 36
Number of Observations Not Used 0

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.14; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-expl-anova.sas, 28JAN2020 13:02


\_\_\_\_\_\_

16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.3: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571107A

Parameter: Cmax (ng/mL) for Metabolite MSC2571107A

The Mixed Procedure

Iteration History

| Iteration | Evaluations | -2 Res Log Like | Criterion |
|-----------|-------------|-----------------|-----------|

0 1 18.54420114

1 6.94881662 0.00000000

Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Estimate

USUBJID(SEQUENCE) 0.05461 Residual 0.02145

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.14; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-expl-anova.sas, 28JAN2020 13:02


16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.3: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571107A

Parameter: Cmax (ng/mL) for Metabolite MSC2571107A

The Mixed Procedure

Fit Statistics

| -2 Res Log Likelihood | 6.9 |
|--------------------------|------|
| AIC (smaller is better) | 10.9 |
| AICC (smaller is better) | 11.4 |
| BIC (smaller is better) | 12.7 |

Type 3 Tests of Fixed Effects

| | Num | Den | | |
|----------|-----|-----|---------|--------|
| Effect | DF | DF | F Value | Pr > F |
| TRTA1 | 1 | 16 | 0.13 | 0.7220 |
| APERIOD | 1 | 16 | 5.50 | 0.0323 |
| SEQUENCE | 1 | 16 | 1.69 | 0.2126 |

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.14; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-expl-anova.sas, 28JAN2020 13:02


16.1: Study Information

16.1.9: Documentation of Statistical Methods

16.1.9.2: Statistical Analysis Output

Listing 16.1.9.2.3: Statistical Output of Exploratory Analysis - Tepotinib Metabolite MSC2571107A

Parameter: Cmax (ng/mL) for Metabolite MSC2571107A

The Mixed Procedure

Least Squares Means

| Effect | TRTA1 | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper | |
|---|---|---|---|---|---|---|---|---|---|---|
| TRTA1 | R | 2.1436 | 0.06500 | 16 | 32.98 | <.0001 | 0.1 | 2.0301 | 2.2571 | |
| TRTA1 | Т | 2.1260 | 0.06500 | 16 | 32.71 | <.0001 | 0.1 | 2.0125 | 2.2394 | |
| | Differences of Least Squares Means | | | | | | | | | |
| Effect | TRTA1 | _TRTA1 | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| TRTA1 | Т | R | -0.01768 | 0.04881 | 16 | -0.36 | 0.7220 | 0.1 | -0.1029 | 0.06755 |

T: 5 x 100 mg TF3; R: 2 x 250 mg TF3

Source: ADPP 22JAN2020 13:55; Listing 16.2.5.14; SDTM package: 15JAN2020 Program: J:\BIO\J19\N-A-PH1-19-070\tables\tr-expl-anova.sas, 28JAN2020 13:02


# WinNonlin Core Output - Tepotinib

WinNonlin 7.0.0.2535

PARAMCD=TEPO,SUBJID=PI ,APERIOD=1,TRTAN=2,TRTA=2 x 250 mg TF3

Date:

PI 09:23:24 Time:

#### WINNONLIN NONCOMPARTMENTAL ANALYSIS PROGRAM 7.0.0.2535 Core Version 04Jun2007

### Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

0.00 Dose time: 450.00 Dose amount:

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

## Summary Table

| Time | Conc. | Pred. | Residual | AUC | AUMC | Weight |
|---------|--------|-------|------------|--------------|-----------|--------|
| h | ng/mL | ng/mL | ng/mL | h*ng/mL | h*h*ng/mL | |
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.050 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.500 | 10.70 | | | 2.408 | 3.611 | |
| 2.000 | 14.50 | | | 8.708 | 14.87 | |
| 3.000 | 34.10 | | | 33.01 | 80.52 | |
| 4.000 | 48.20 | | | 74.16 | 228.1 | |
| 6.000 | 105.0 | | | 227.4 | 1051. | |
| 8.017 | 117.0 | | | 451.2 | 2632. | |
| 12.00 | 218.0 | | | 1118. | 9710. | |
| 16.03 | 222.0 | | | 2006. 2.216 | e+004 | |
| 24.00 | 257.0 | | | 3914. 6.091 | e+004 | |
| 36.07 * | 197.0 | 187.8 | 9.198 | 6637, 1,42 | 0e+005 | 1.000 |
| 48.00 * | 148.0 | 143.5 | 4.524 | 8681. 2.27 | 3e+005 | 1.000 |
| 60.00 * | 110.0 | 109.4 | 0.5533 1.0 | 022e+004 3.0 | 99e+005 | 1.000 |
| 72.00 * | 76.50 | 83.49 | -6.989 1.1 | 33e+004 3.82 | 25e+005 | 1.000 |
| 96.00 * | 45.90 | 48.58 | -2.682 1.2 | 76e+004 5.0° | 18e+005 | 1.000 |
| 120.0 * | 30.70 | 28.27 | 2.430 1.3 | 67e+004 5.9 | 90e+005 | 1.000 |
| 144.0 * | 15.10 | 16.45 | -1.350 1.4 | 20e+004 6.67 | 79e+005 | 1.000 |
| 168.0 * | 10.20 | 9.572 | 0.6275 1.4 | 150e+004 7.1 | 45e+005 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

### Final Parameters

| Rsq | | 0.9960 |
|--------------------|-------|----------|
| Rsq_adjusted | | 0.9953 |
| Corr_XY | | -0.9980 |
| No_points_lambda_z | | 8 |
| Lambda_z | 1/h | 0.0226 |
| Lambda_z_lower | h | 36.0667 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 30.7238 |
| Tlag | h | 1.0500 |
| Tmax | h | 24.0000 |
| Cmax | ng/mL | 257.0000 |

Cmax\_D ng/mL/mg 0.5711 168.0000 Tlast h Clast ng/mL 10.2000 AUClast 14497.1496 h\*ng/mL **AUCall** 14497.1496 h\*ng/mL AUCINF\_obs 14949.2650 h\*ng/mL AUCINF\_Dobs
AUCINF\_D\_obs
AUC\_%Extrap\_obs
Vz\_F\_obs
CI\_F\_obs
AUCINF\_pred
AUCINF\_D\_pred h\*ng/mL/mg 33.2206 % 3.0243 1334.2643 L L/h 30.1018 h\*ng/mL 14921.4501 h\*ng/mL/mg 33.1588 AUC\_%Extrap\_pred 2.8436 % Vz\_F\_pred L 1336.7515 CI\_F\_pred L/h 30.1579 **AUMClast** h\*h\*ng/mL 714474.9371 AUMCINF\_obs 810470.3763 h\*h\*ng/mL AUMC\_%Extrap\_obs 11.8444 AUMCINF\_pred AUMC\_%Extrap\_pred 804564.5644 h\*h\*ng/mL 11.1973 49.2838 MRTlast MRTINF\_obs 54.2147 h MRTINF\_pred h 53.9200 AUC0\_24 3913.7658 h\*ng/mL

WinNonlin 7.0.0.2535

PARAMCD=TEPO,SUBJID=PI ,APERIOD=2,TRTAN=2,TRTA=2 x 250 mg TF3

Date: PI Time: 09:23:24


## Settings

-----

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

| Conc. | Pred. | Residual | AUC | AUMC | Weight |
|---|---|---|---|---|---|
| ng/mL | ng/mL | ng/mL | h*ng/mL | h*h*ng/mL | |
| 0.0000 | | | 0.0000 | 0.0000 | |
| 0.0000 | | | 0.0000 | 0.0000 | |
| 0.0000 | | | 0.0000 | 0.0000 | |
| 5.860 | | | 0.7325 | .5494 | |
| 12.50 | | | 3.028 | 2.661 | |
| 24.70 | | | 12.33 | 15.05 | |
| 38.60 | | | 28.15 | 43.61 | |
| 76.10 | | | 85.50 | 196.4 | |
| 95.60 | | | 171.4 | 501.7 | |
| 256.0 | | | 523.0 | 2420. | |
| 228.0 | | | 1006. | 5795. | |
| 231.0 | | | 1924, 1,499 | e+004 | |
| 225.0 | | | 2836, 2,775 | e+004 | |
| 239.0 | | | 4696, 6,518 | e+004 | |
| 240.0 | | | 7566, 1,513 | e+005 | |
| | | 1.04 | | | |
| . 55.0 | | 1.0 | 0.02 | | |
| | ng/mL<br>0.0000<br>0.0000<br>0.0000<br>5.860<br>12.50<br>24.70<br>38.60<br>76.10<br>95.60<br>256.0<br>228.0<br>231.0<br>225.0 | ng/mL ng/mL 0.0000 0.0000 0.0000 5.860 12.50 24.70 38.60 76.10 95.60 256.0 228.0 231.0 225.0 239.0 240.0 232.0 249.0 | ng/mL ng/mL ng/mL ng/mL 0.0000 0.0000 0.0000 5.860 12.50 24.70 38.60 76.10 95.60 256.0 228.0 231.0 225.0 239.0 240.0 232.0 1.0 249.0 | ng/mL ng/mL ng/mL h*ng/mL 0.0000 0.0000 0.0000 0.0000 0.0000 0.0000 0.0000 0.0000 5.860 0.7325 0.000 0.0000 0. | ng/mL ng/mL ng/mL h*ng/mL h*ng/mL h*ng/mL 0.0000 0.0000 0.0000 0.0000 0.0000 0.0000 0.0000 0.0000 0.0000 5.860 0.7325 0.5494 12.50 3.028 2.661 24.70 12.33 15.05 38.60 28.15 43.61 76.10 85.50 196.4 95.60 171.4 501.7 256.0 523.0 2420. 228.0 1006. 5795. 231.0 1924. 1.499e+004 225.0 2836. 2.775e+004 239.0 4696. 6.518e+004 240.0 7566. 1.513e+005 232.0 1.040e+004 2.702e+005 249.0 1.328e+004 4.266e+005 |

| 96.00 | 137.0 | | 1.995e+004 9.345e+005 | |
|---------|-------|-------|-------------------------------|-------|
| 120.0 * | 76.30 | 75.83 | 0.4695 2.244e+004 1.200e+006 | 1.000 |
| 144.0 * | 47.20 | 47.79 | -0.5863 2.389e+004 1.391e+006 | 1.000 |
| 168.0 * | 30.30 | 30.11 | 0.1864 2.480e+004 1.533e+006 | 1.000 |

\*) Starred values were included in the estimation of Lambda\_z.

#### Final Parameters

| Rsq | | 0.9995 |
|--------------------|------------|--------------|
| Rsq_adjusted | | 0.9989 |
| Corr_XY | | -0.9997 |
| No points lambda z | | 3 |
| Lambda_z | 1/h | 0.0192 |
| Lambda_z_lower | h | 120.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 36.0262 |
| Tlag | h | 0.5000 |
| Tmax | h | 6.0000 |
| Cmax | ng/mL | 256.0000 |
| Cmax_D | ng/mL/mg | 0.5689 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 30.3000 |
| AUClast | h*ng/mL | 24804.7480 |
| AUCall | h*ng/mL | 24804.7480 |
| AUCINF_obs | h*ng/mL | 26379.5832 |
| AUCINF_D_obs | h*ng/mL/mg | 58.6213 |
| AUC_%Extrap_obs | % | 5.9699 |
| Vz_F_obs | L | 886.6191 |
| Cl_F_obs | L/h | 17.0586 |
| AUCINF_pred | h*ng/mL | 26369.8930 |
| AUCINF_D_pred | h*ng/mL/mg | 58.5998 |
| AUC_%Extrap_pred | % | 5.9353 |
| Vz_F_pred | L | 886.9449 |
| Cl_F_pred | L/h | 17.0649 |
| AUMClast | h*h*ng/mL | 1532953.4265 |
| AUMCINF_obs | h*h*ng/mL | 1879377.4103 |
| AUMC_%Extrap_obs | % | 18.4329 |
| AUMCINF_pred | h*h*ng/mL | 1877245.8165 |
| AUMC_%Extrap_pred | % | 18.3403 |
| MRTlast | h | 61.8008 |
| MRTINF_obs | h | 71.2436 |
| MRTINF_pred | h | 71.1890 |
| AUC0_24 | h*ng/mL | 4692.2430 |

WinNonlin 7.0.0.2535

PARAMCD=TEPO, SUBJID=PI ,APERIOD=2, TRTAN=2, TRTA=2 x 250 mg TF3

PI 09:23:22 Date: Time:


## Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 450.00 Dose amount:

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values
Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

| Time | Conc.<br>ng/mL | Pred.<br>ng/mL | Residual<br>ng/mL | AUC<br>h*ng/mL | AUMC<br>h*h*ng/mL | Weight |
|---|---|---|---|---|---|---|
| 0.0000<br>0.2500<br>0.5000<br>0.7500<br>1.000<br>1.500<br>2.000<br>3.000<br>4.000<br>6.000<br>8.000<br>12.00<br>16.00<br>24.00<br>36.00<br>48.00<br>60.00 * | 0.0000<br>0.0000<br>7.790<br>16.90<br>32.90<br>69.20<br>96.00<br>120.0<br>142.0<br>172.0<br>192.0<br>206.0<br>197.0<br>230.0<br>278.0<br>232.0<br>215.0<br>179.0 | 222.4<br>179.5<br>116.9 | 1.0<br>-7.439 1.3<br>-0.4744 1.5 | 0.0000<br>0.0000<br>0.9738<br>4.060<br>10.29<br>35.81<br>77.11<br>185.1<br>316.1<br>630.1 | 0.0000<br>0.0000<br>0.4869<br>2.558<br>8.255<br>42.43<br>116.4<br>392.4<br>856.4<br>2456.<br>5024.<br>e+004<br>e+004<br>le+005<br>88e+005<br>43e+005<br>97e+005 | 1.000<br>1.000 |
| 120.0 *<br>144.1 *<br>168.0 * | 87.70<br>46.30<br>31.70 | 76.18<br>49.56<br>32.32 | 11.52 2.1<br>-3.261 2.2 | 91e+004 8.60<br>33e+004 1.13<br>89e+004 1.3<br>81e+004 1.4 | 28e+006<br>32e+006 | 1.000<br>1.000<br>1.000<br>1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

## Final Parameters

| Rsq | | 0.9907 |
|--------------------|------------|--------------|
| Rsq_adjusted | | 0.9883 |
| Corr_XY | | -0.9953 |
| No_points_lambda_z | | 6 |
| Lambda_z | 1/h | 0.0179 |
| Lambda_z_lower | h | 60.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 38.8093 |
| Tlag | h | 0.2500 |
| Tmax | h | 36.0000 |
| Cmax | ng/mL | 278.0000 |
| Cmax_D | ng/mL/mg | 0.6178 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 31.7000 |
| AUClast | h*ng/mL | 23813.9884 |
| AUCall | h*ng/mL | 23813.9884 |
| AUCINF_obs | h*ng/mL | 25588.8703 |
| AUCINF_D_obs | h*ng/mL/mg | 56.8642 |
| AUC %Extrap obs | % | 6.9361 |
| Vz_F_obs | L | 984.6267 |
| CI F obs | L/h | 17.5858 |
| AUCINF_pred | h*ng/mL | 25623.6769 |
| AUCINF D pred | h*ng/mL/mg | 56.9415 |
| AUC_%Extrap_pred | % | 7.0626 |
| Vz_F_pred | L | 983.2892 |
| Cl_F_pred | L/h | 17.5619 |
| AUMClast | h*h*ng/mL | 1475092.5334 |
| AUMCINF_obs | h*h*ng/mL | 1872648.2664 |
| AUMC_%Extrap_obs | % | 21.2296 |
| AUMCINF_pred | h*h*ng/mL | 1880444.6104 |
| AUMC %Extrap pred | % | 21.5562 |
| MRTlast | h | 61.9423 |
| MRTINF_obs | h | 73.1821 |
| MRTINF_pred | h | 73.3870 |
| AUC0_24 | h*ng/mL | 4303.9760 |
| | • | |

WinNonlin 7.0.0.2535
PARAMCD=TEPO,SUBJID=PI ,APERIOD=2,TRTAN=2,TRTA=2 x 250 mg TF3

```
0 \ 0 \ 0000 \ 0 \ 0 \ 0
\begin{smallmatrix} 0 \end{smallmatrix} \ 0 \\ \ 0 \end{smallmatrix} \ 0 \end{smallmatrix} \ 0 \end{smallmatrix} \ 0 \\ \ 0 \end{smallmatrix} \ 0 \\ \ 0 \end{smallmatrix} \ 0 \\ \ 0 \end{smallmatrix} \ 0 \\ \ 0 
000000000000000000
0 00 0 00 0 00 0 0 0 0 00 0
```

| AUC_%Extrap_obs | % | 1.8710 |
|-------------------|------------|--------------|
| Vz_F_obs | L | 1008.3388 |
| Cl_F_obs | L/h | 25.9036 |
| AUCINF_pred | h*ng/mL | 17351.8162 |
| AUCINF_D_pred | h*ng/mL/mg | 38.5596 |
| AUC_%Extrap_pred | % | 1.7562 |
| Vz_F_pred | L | 1009.5189 |
| CI_F_pred | L/h | 25.9339 |
| AUMClast | h*h*ng/mL | 780914.2247 |
| AUMCINF_obs | h*h*ng/mL | 848 173.1252 |
| AUMC_%Extrap_obs | % | 7.9299 |
| AUMCINF_pred | h*h*ng/mL | 843970.8712 |
| AUMC_%Extrap_pred | % | 7.4714 |
| MRTlast | h | 45.8092 |
| MRTINF_obs | h | 48.8238 |
| MRTINF_pred | h | 48.6388 |
| AUC0_24 | h*ng/mL | 5224.6947 |

WinNonlin 7.0.0.2535

PARAMCD=TEPO,SUBJID=PI ,APERIOD=1,TRTAN=1,TRTA=5 x 100 mg TF3

Date: PI Time: 09:23:22


#### Settings

-----

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

| • | | | | | | |
|---|---|---|---|---|---|---|
| Time<br>h | Conc.<br>ng/mL | Pred.<br>ng/mL | Residual<br>ng/mL | AUC<br>h*ng/mL | AUMC<br>h*h*ng/mL | Weight |
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.000 | 16.30 | | | 2.038 | 2.038 | |
| 1.500 | 70.30 | | | 23.69 | 32.48 | |
| 2.000 | 135.0 | | | 75.01 | 126.3 | |
| 3.000 | 210.0 | | | 247.5 | 576.3 | |
| 4.000 | 263.0 | | | 484.0 | 1417. | |
| 6.000 | 273.0 | | | 1020. | 4107. | |
| 8.000 | 280.0 | | | 1573. | 7985. | |
| 12.00 | 227.0 | | | 2583. 1.802 | 2e+004 | |
| 16.00 | 196.0 | | | 3428. 2.980 | | |
| 24.02 * | 211.0 | 205.9 | 5.061 | 5059. 6.26 | 8e+004 | 1.000 |
| 36.00 * | 174.0 | 170.7 | 3.337 | 7359. 1.31 | l2e+005 | 1.000 |
| 48.00 * | 129.0 | 141.4 | -12.39 | 9163. 2.06 | 5e+005 | 1.000 |
| 60.00 * | 116.0 | 117.1 | | 63e+004 2.8 | | 1.000 |
| 72.02 * | 96.00 | 97.03 | | 90e+004 3.6 | | 1.000 |
| 96.00 * | 68.80 | 66.62 | 2.184 1.3 | 86e+004 5.3 | 24e+005 | 1.000 |
| 120.3 * | 51.50 | 45.52 | 5.978 1.5 | 31e+004 6.8 | 85e+005 | 1.000 |
| 144.0 * | 29.90 | 31.40 | -1.502 1.6 | 25e+004 8.1 | 18e+005 | 1.000 |
| 168.1 * | 20.70 | 21.50 | -0.8036 1.6 | 86e+004 9.0 | 56e+005 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

### Final Parameters

| Rsq | | 0.9940 |
|--------------------|------------|--------------|
| Rsq_adjusted | | 0.9931 |
| Corr_XY | | -0.9970 |
| No_points_lambda_z | | 9 |
| Lambda_z | 1/h | 0.0157 |
| Lambda_z_lower | h | 24.0167 |
| Lambda_z_upper | h | 168.1167 |
| HL_Lambda_z | h | 44.2083 |
| Tlag | h | 0.7500 |
| Tmax | h | 8.0000 |
| Cmax | ng/mL | 280.0000 |
| Cmax_D | ng/mL/mg | 0.6222 |
| Tlast | h | 168.1167 |
| Clast | ng/mL | 20.7000 |
| AUClast | h*ng/mL | 16855.7226 |
| AUCall | h*ng/mL | 16855.7226 |
| AUCINF obs | h*ng/mL | 18175.9510 |
| AUCINF_D_obs | h*ng/mL/mg | 40.3910 |
| AUC_%Extrap_obs | % | 7.2636 |
| Vz_F_obs | L | 1579.0435 |
| CI_F_obs | L/h | 24.7580 |
| AUCINF_pred | h*ng/mL | 18227.2059 |
| AUCINF_D_pred | h*ng/mL/mg | 40.5049 |
| AUC %Extrap pred | % | 7.5244 |
| Vz F pred | L | 1574.6032 |
| CI_F_pred | L/h | 24.6884 |
| AUMClast | h*h*ng/mL | 905589.6981 |
| AUMCINF_obs | h*h*ng/mL | 1211745.1415 |
| AUMC %Extrap obs | % | 25.2657 |
| AUMCINF_pred | h*h*ng/mL | 1223630.9399 |
| AUMC_%Extrap_pred | % | 25,9916 |
| MRTlast | h | 53.7259 |
| MRTINF_obs | h | 66.6675 |
| MRTINF_pred | h | 67.1321 |
| AUC0 24 | h*ng/mL | 5055.6666 |

WinNonlin 7.0.0.2535

PARAMCD=TEPO, SUBJID=PI ,APERIOD=1, TRTAN=1, TRTA=5 x 100 mg TF3

PI 09:23:23 Date: Time:

### WINNONLIN NONCOMPARTMENTAL ANALYSIS PROGRAM 7.0.0.2535 Core Version 04Jun2007

## Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

0.00 Dose time: 450.00 Dose amount:

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values
Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

| Time<br>h | Conc.<br>ng/mL | Pred.<br>ng/mL | Residual<br>ng/mL | AUC<br>h*ng/mL | AUMC<br>h*h*ng/mL | Weight |
|---|---|---|---|---|---|---|
| 0.0000<br>0.2500 | 0.0000 | | | | 0.0000<br>0.0000 | |
| 0.5000 | 0.0000 | | | | 0.0000 | |

| 0.7500<br>1.000 | 0.0000 | | 0.0000 0.0000<br>0.0000 0.0000 | |
|-----------------|--------|-------|--------------------------------|-------|
| 1.500 | 21.40 | | 5.350 8.025 | |
| 2.000 | 16.70 | | 14.83 24.51 | |
| 3.000 | 52.60 | | 49.48 120.1 | |
| 4.000 | 53.30 | | 102.4 305.6 | |
| 6.000 | 100.0 | | 255.7 1119. | |
| 8.000 | 107.0 | | 462.7 2575. | |
| 12.00 | 170.0 | | 1017. 8367. | |
| 16.00 | 175.0 | | 1707. 1.805e+004 | |
| 24.00 | 173.0 | | 3099. 4.588e+004 | |
| 36.00 | 208.0 | | 5385. 1.157e+005 | |
| 48.00 | 136.0 | | 7418. 2.003e+005 | |
| 60.03 | 103.0 | | 8847. 2.770e+005 | |
| 72.00 | 70.10 | | 9870. 3.442e+005 | |
| 96.00 * | 32.80 | 31.77 | 1.029 1.105e+004 4.414e+005 | 1.000 |
| 120.0 * | 17.20 | 18.28 | -1.081 1.163e+004 5.033e+005 | 1.000 |
| 144.0 * | 10.80 | 10.52 | 0.2805 1.196e+004 5.466e+005 | 1.000 |
| 168.0 * | 6.070 | 6.053 | 0.01687 1.216e+004 5.771e+005 | 1.000 |

## \*) Starred values were included in the estimation of Lambda\_z.

## Final Parameters

| Rsq | | 0.9965 |
|--------------------|------------|-------------|
| Rsq_adjusted | | 0.9947 |
| Corr_XY | | -0.9982 |
| No_points_lambda_z | | 4 |
| Lambda_z | 1/h | 0.0230 |
| Lambda_z_lower | h | 96.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 30.1010 |
| Tlag | h | 1.0000 |
| Tmax | h | 36.0000 |
| Cmax | ng/mL | 208.0000 |
| Cmax_D | ng/mL/mg | 0.4622 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 6.0700 |
| AUClast | h*ng/mL | 12155.8917 |
| AUCall | h*ng/mL | 12155.8917 |
| AUCINF_obs | h*ng/mL | 12419.4909 |
| AUCINF_D_obs | h*ng/mL/mg | 27.5989 |
| AUC_%Extrap_obs | % | 2.1225 |
| Vz_F_obs | L | 1573.4902 |
| Cl_F_obs | L/h | 36.2334 |
| AUCINF_pred | h*ng/mL | 12418.7581 |
| AUCINF_D_pred | h*ng/mL/mg | 27.5972 |
| AUC_%Extrap_pred | % | 2.1167 |
| Vz_F_pred | L | 1573.5831 |
| Cl_F_pred | L/h | 36.2355 |
| AUMClast | h*h*ng/mL | 577097.4841 |
| AUMCINF_obs | h*h*ng/mL | 632829.3454 |
| AUMC_%Extrap_obs | % | 8.8068 |
| AUMCINF_pred | h*h*ng/mL | 632674.4096 |
| AUMC_%Extrap_pred | % | 8.7844 |
| MRTlast | h | 47.4747 |
| MRTINF_obs | h | 50.9545 |
| MRTINF_pred | h | 50.9451 |
| AUC0_24 | h*ng/mL | 3098.7112 |

WinNonlin 7.0.0.2535

PARAMCD=TEPO,SUBJID=pj ,APERIOD=1,TRTAN=1,TRTA=5 x 100 mg TF3

Date: PI Time: 09:23:23

WINNONLIN NONCOMPARTMENTAL ANALYSIS PROGRAM 7.0.0.2535

```
0 0 0000 0 0 0
0 0 0 0 0 0000 0 00 0 0 0 0 0 0 0 0 0
\begin{smallmatrix} 0 \end{smallmatrix} \ 0 \\ \ 0 \end{smallmatrix} \ 0 \end{smallmatrix} \ 0 \\ \ 0 \end{smallmatrix} \ 0 \\ \ 0 \end{smallmatrix} \ 0 \\ \ 0 
0 0 0 0 0 00 00 0 0 0 0
000000000000000
0 00 0 00 0 00 0 0 0 0 0 0
```

CI\_F\_pred L/h 22.5195 **AUMClast** h\*h\*ng/mL 1080950.4897 1333031.7987 AUMCINF\_obs h\*h\*ng/mL AUMC\_%Extrap\_obs 18.9104 AUMCINF\_pred AUMC\_%Extrap\_pred h\*h\*ng/mL 1337815.7841 19.2003 57.4438 MRTlast MRTINF\_obs 66.7818 h MRTINF\_pred h 66.9487 AUC0\_24 h\*ng/mL 4766.7594

WinNonlin 7.0.0.2535

PARAMCD=TEPO,SUBJID=PI ,APERIOD=2,TRTAN=1,TRTA=5 x 100 mg TF3

Date: PI Time: 09:23:21


### Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

## Summary Table

| Time | Conc. | Pred. | Residual | AUC | AUMC | Weight |
|---------|--------|-------|--------------|--------------|-----------|--------|
| h | ng/mL | ng/mL | ng/mL | h*ng/mL | h*h*ng/mL | |
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5167 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 6.050 | | | 0.7058 ( | 0.5294 | |
| 1.000 | 7.990 | | | 2.461 | 2.095 | |
| 1.500 | 18.40 | | | 9.058 | 10.99 | |
| 2.000 | 89.20 | | | 35.96 | 62.49 | |
| 3.000 | 76.80 | | | 118.8 | 268.6 | |
| 4.000 | 122.0 | | | 218.2 | 627.8 | |
| 6.000 | 249.0 | | | 589.2 | 2610. | |
| 8.000 | 304.0 | | | 1142. | 6536. | |
| 12.00 | 351.0 | | | 2452. 1.982 | e+004 | |
| 16.00 | 309.0 | | | 3770. 3.822 | e+004 | |
| 24.00 | 255.0 | | | 6020. 8.292 | e+004 | |
| 36.00 | 193.0 | | | 8690. 1.623 | e+005 | |
| 48.00 | 162.0 | | 1.08 | 1e+004 2.51 | 2e+005 | |
| 60.00 | 122.0 | | 1.25 | 1e+004 3.42 | 1e+005 | |
| 72.00 | 75.50 | | 1.36 | 7e+004 4.18 | 3e+005 | |
| 96.00 | 59.00 | | 1.52 | 8e+004 5.52 | 4e+005 | |
| 120.0 * | 30.10 | 29.74 | 0.3605 1.6 | 31e+004 6.6 | 23e+005 | 1.000 |
| 144.0 * | 16.90 | 17.31 | -0.4122 1.68 | 36e+004 7.34 | 11e+005 | 1.000 |
| 168.0 * | 10.20 | 10.08 | 0.1221 1.7 | 17e+004 7.8 | 35e+005 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

#### Final Parameters

 Rsq
 0.9985

 Rsq\_adjusted
 0.9970

 Corr\_XY
 -0.9993

| Lambda_z 1/h 0.0225 Lambda_z_lower h 120.0000 Lambda_z_upper h 168.0000 HL_Lambda_z h 30.7457 Tlag h 0.5167 Tmax h 12.0000 Cmax ng/mL 351.0000 Cmax_D ng/mL/mg 0.7800 Tlast h 168.0000 | |
|---|---|
| Lambda_z_upper h 168.0000 HL_Lambda_z h 30.7457 Tlag h 0.5167 Tmax h 12.0000 Cmax ng/mL 351.0000 Cmax_D ng/mL/mg 0.7800 Tlast h 168.0000 | |
| Lambda_z_upper h 168.0000 HL_Lambda_z h 30.7457 Tlag h 0.5167 Tmax h 12.0000 Cmax ng/mL 351.0000 Cmax_D ng/mL/mg 0.7800 Tlast h 168.0000 | |
| HL_Lambda_z h 30.7457 Tlag h 0.5167 Tmax h 12.0000 Cmax ng/mL 351.0000 Cmax_D ng/mL/mg 0.7800 Tlast h 168.0000 | |
| Tmax h 12.0000 Cmax ng/mL 351.0000 Cmax_D ng/mL/mg 0.7800 Tlast h 168.0000 | |
| Tmax h 12.0000 Cmax ng/mL 351.0000 Cmax_D ng/mL/mg 0.7800 Tlast h 168.0000 | |
| Cmax_D ng/mL/mg 0.7800<br>Tlast h 168.0000 | |
| Cmax_D ng/mL/mg 0.7800<br>Tlast h 168.0000 | |
| Clast ng/mL 10.2000 | |
| AUClast h*ng/mL 17174.0467 | |
| AUCall h*ng/mL 17174.0467 | |
| AUCINF_obs h*ng/mL 17626.4846 | , |
| AUCINF_D_obs h*ng/mL/mg 39.170 | 0 |
| AUC_%Extrap_obs % 2.5668 | |
| Vz_F_obs L 1132.4150 | |
| CI_F_obs L/h 25.5298 | |
| AUCINF_pred h*ng/mL 17621.0665 | j |
| AUCINF_D_pred h*ng/mL/mg 39.157 | 9 |
| AUC_%Extrap_pred % 2.5368 | |
| Vz_F_pred L 1132.7632 | |
| CI_F_pred L/h 25.5376 | |
| AUMClast h*h*ng/mL 783474.7942 | |
| AUMCINF_obs h*h*ng/mL 879552.995 | 0 |
| AUMC_%Extrap_obs % 10.923 | 5 |
| AUMCINF_pred h*h*ng/mL 878402.427 | 2 |
| AUMC_%Extrap_pred % 10.806 | 9 |
| MRTlast h 45.6197 | |
| MRTINF_obs h 49.8995 | |
| MRTINF_pred h 49.8496 | |
| AUC0_24 h*ng/mL 6019.5094 | |

WinNonlin 7.0.0.2535

PARAMCD=TEPO,SUBJID=PI ,APERIOD=1,TRTAN=1,TRTA=5 x 100 mg TF3

PI 09:23:24 Date: Time:


## Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

0.00 Dose time: 450.00 Dose amount:

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values
Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

| Time<br>h | Conc.<br>ng/mL | Pred.<br>ng/mL | Residual<br>ng/mL | AUC<br>h*ng/m | AUMC<br>L h*h*ng/mL | Weight |
|---|---|---|---|---|---|---|
| 0.0000<br>0.2667<br>0.5000<br>0.7500<br>1.000<br>1.500<br>2.000<br>3.000<br>4.000<br>6.000 | 0.0000<br>0.0000<br>0.0000<br>7.380<br>9.900<br>26.40<br>51.40<br>9.570<br>126.0 | | | 0.0000<br>0.0000<br>0.0000<br>0.9225<br>3.083<br>12.16<br>31.61<br>105.2<br>216.0<br>516.0 | 0.0000<br>0.0000<br>0.0000<br>0.6919<br>2.621<br>15.00<br>50.60<br>245.5<br>641.1<br>2189. | |
| 0.000 | 4.0 | | | 0.0.0 | 2.00. | |

| 8.000 | 160.0 | | | 849.8 4521. | |
|---------|-------|-------|----------|------------------|-------|
| 12.00 * | 153.0 | 158.3 | -5.302 | 1476. 1.077e+004 | 1.000 |
| 16.00 * | 144.0 | 145.0 | -1.024 | 2070. 1.907e+004 | 1.000 |
| 24.00 * | 120.0 | 121.7 | -1.715 | 3123. 4.001e+004 | 1.000 |
| 36.00 * | 92.20 | 93.58 | -1.384 | 4388. 7.765e+004 | 1.000 |
| 48.00 * | 77.40 | 71.95 | 5.445 | 5404. 1.201e+005 | 1.000 |
| 60.00 * | 53.50 | 55.32 | -1.824 | 6180. 1.618e+005 | 1.000 |
| 72.00 * | 46.30 | 42.54 | 3.762 | 6778. 2.011e+005 | 1.000 |
| 96.00 * | 23.80 | 25.15 | -1.347 | 7589. 2.682e+005 | 1.000 |
| 120.2 * | 15.30 | 14.82 | 0.4824 | 8054. 3.180e+005 | 1.000 |
| 144.0 * | 8.630 | 8.789 | -0.1586 | 8332. 3.544e+005 | 1.000 |
| 168.0 * | 5.130 | 5.196 | -0.06559 | 8493. 3.794e+005 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

## Final Parameters

| Tillatt diditiolois | | |
|---------------------|------------|-------------|
| Rsq | | 0.9985 |
| Rsq_adjusted | | 0.9984 |
| Corr XY | | -0.9993 |
| No_points_lambda_z | | 11 |
| Lambda_z | 1/h | 0.0219 |
| Lambda_z_lower | h | 12.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 31.6478 |
| Tlag | h | 0.5000 |
| Tmax | h | 6.0000 |
| Cmax | ng/mL | 174.0000 |
| Cmax_D | ng/mL/mg | 0.3867 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 5.1300 |
| AUClast | h*ng/mL | 8493.2403 |
| AUCall | h*ng/mL | 8493.2403 |
| AUCINF_obs | h*ng/mL | 8727.4667 |
| AUCINF_D_obs | h*ng/mL/mg | 19.3944 |
| AUC_%Extrap_obs | % | 2.6838 |
| Vz_F_obs | L | 2354.1972 |
| CI_F_obs | L/h | 51.5614 |
| AUCINF_pred | h*ng/mL | 8730.4613 |
| AUCINF_D_pred | h*ng/mL/mg | 19.4010 |
| AUC_%Extrap_pred | % | 2.7172 |
| Vz_F_pred | L | 2353.3897 |
| Cl_F_pred | L/h | 51.5437 |
| AUMClast | h*h*ng/mL | 379413.2473 |
| AUMCINF_obs | h*h*ng/mL | 429457.6382 |
| AUMC_%Extrap_obs | % | 11.6529 |
| AUMCINF_pred | h*h*ng/mL | 430097.4552 |
| AUMC_%Extrap_pred | % | 11.7844 |
| MRTlast | h | 44.6724 |
| MRTINF_obs | h | 49.2076 |
| MRTINF_pred | h | 49.2640 |
| AUC0_24 | h*ng/mL | 3122.6100 |

WinNonlin 7.0.0.2535

PARAMCD=TEPO,SUBJID=pj ,APERIOD=1,TRTAN=1,TRTA=5 x 100 mg TF3

Date: PI Time: 09:23:23

## WINNONLIN NONCOMPARTMENTAL ANALYSIS PROGRAM 7.0.0.2535 Core Version 04Jun2007

## Settings

-----

Model: Plasma Data, Extravascular Administration Number of nonmissing observations: 22

Dose time: 0.00

```
\begin{smallmatrix} 0 \end{smallmatrix} \ 0 \\ \ 0 \end{smallmatrix} \ 0 \end{smallmatrix} \ 0 \end{smallmatrix} \ 0 \\ \ 0 \end{smallmatrix} \ 0 \\ \ 0 \end{smallmatrix} \ 0 \\ \ 0 \end{smallmatrix} \ 0 \\ \ 0 
00000000000000
0 00 0 00 0 00 0 0 0 0 00 0
^{\circ}
```

MRTINF\_obs MRTINF\_pred AUC0\_24 65.2297 h h 65.1955 h\*ng/mL 3422.5197

WinNonlin 7.0.0.2535

PARAMCD=TEPO,SUBJID=PI ,APERIOD=1,TRTAN=1,TRTA=5 x 100 mg TF3

> Date: PI 09:23:22 Time:


#### Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 450.00 Dose amount:

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

#### Summary Table

| Time<br>h | Conc.<br>ng/mL | Pred.<br>ng/mL | Residual<br>ng/mL | AUC<br>h*ng/mL | AUMC<br>h*h*ng/ml | Weight<br>L |
|---|---|---|---|---|---|---|
| 0.0000 | 0.0000 | | | 0.0000 | | |
| 0.0000 | 0.0000 | | | | 0.0000 | |
| 0.2500 | 0.0000 | | | | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.033 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.500 | 6.060 | | | 1.414 | 2.121 | |
| 2.000 | 13.30 | | | 6.254 | 11.04 | |
| 3.000 | 39.70 | | | 32.75 | 83.89 | |
| 4.000 | 49.00 | | | 77.10 | 241.4 | |
| 6.000 | 227.0 | | | 353.1 | 1799. | |
| 8.000 | 231.0 | | | 811.1 | 5009. | |
| 12.00 | 241.0 | | | 1755, 1,449 | e+004 | |
| 16.00 | 205.0 | | | 2645, 2,690 | | |
| 24.00 | 195.0 | | | 4245. 5.884 | | |
| 36.00 * | 181.0 | 185.7 | -4.703 | 6500, 1,26 | | 1.000 |
| 48.02 * | 145.0 | 147.9 | -2.936 | 8451, 2,078 | | 1.000 |
| 60.00 * | 125.0 | 117.9 | | 07e+004 2.94 | | 1.000 |
| | | | | 36e+004 3.79 | | |
| 72.00 * | 92.50 | 93.97 | | | | 1.000 |
| 96.00 * | 59.80 | 59.67 | | 16e+004 5.2 | | 1.000 |
| 120.0 * | 38.00 | 37.89 | | 31e+004 6.5 | | 1.000 |
| 144.0 * | 24.80 | 24.06 | | 06e+004 7.5 | | 1.000 |
| 168.0 * | 14.80 | 15.28 | -0.4801 1.5 | 52e+004 8.2 | 25e+005 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

## Final Parameters

| Rsq | | 0.9988 |
|--------------------|-----|----------|
| Rsq_adjusted | | 0.9986 |
| Corr_XY | | -0.9994 |
| No_points_lambda_z | | 8 |
| Lambda_z | 1/h | 0.0189 |
| Lambda_z_lower | h | 36.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 36.6333 |
| Tlag | h | 1.0333 |
| Tmax | h | 12.0000 |

241.0000 Cmax ng/mL ng/mL/mg Cmax D 0.5356 168.0000 Tlast h Clast ng/mL 14.8000 **AUClast** h\*ng/mL 15520.8814 AUCall h\*ng/mL 15520.8814 AUCINF\_obs 16303.0722 h\*ng/mL AUCINF\_D\_obs h\*ng/mL/mg 36.2290 AUC\_%Extrap\_obs Vz\_F\_obs 4.7978 1458,7943 CI\_F\_obs L/h 27.6022 AUCINF\_pred AUCINF\_D\_pred h\*ng/mL 16328.4450 h\*ng/mL/mg 36.2854 AUC\_%Extrap\_pred 4.9457 Vz\_F\_pred 1456.5275 L CI\_F\_pred L/h 27.5593 **AUMClast** h\*h\*ng/mL 822459.3369 AUMCINF\_obs h\*h\*ng/mL 995206.7539 AUMC\_%Extrap\_obs 17.3579 1000810.3660 AUMCINF\_pred h\*h\*ng/mL AUMC\_%Extrap\_pred 17.8207 MRTlast 52.9905 h MRTINF\_obs h 61.0441 MRTINF\_pred 61,2924 h AUC0\_24 h\*ng/mL 4244.8300

WinNonlin 7.0.0.2535

PARAMCD=TEPO,SUBJID=PI ,APERIOD=1,TRTAN=1,TRTA=5 x 100 mg TF3

Date: Time:

PI 09:23:22


## Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

## Summary Table

Pred. AUC AUMC Weight Time Conc. Residual h ng/mL ng/mL ng/mL h\*ng/mL h\*h\*ng/mL 0.0000 0.0000 0.0000 0.0000 0.2500 0.0000 0.0000 0.0000 0.5000 0.0000 0.0000 0.0000 0.7667 7.930 1.057 0.8106 1.000 10.20 3.173 2.710 1.500 41.80 16.17 20.93 2.000 67.90 43.60 70.56 3.000 102.0 128.5 291.5 4.000 130.0 244.5 704.5 186.0 6.000 560.5 2340. 8.017 234.0 984.0 5357. 12.00 222.0 1892. 1.443e+004 16.00 261.0 2858. 2.811e+004 24.02 267.0 4974. 7.055e+004 7619. 1.489e+005 36.00 \* 178.9 1.097 1.000 180.0 48.00 \* 142.0 139.5 2.496 9542. 2.292e+005 1.000 60.00 \* 108.8 2.219 1.105e+004 3.104e+005 1.000 111.0

| 72.00 * | 85.00 | 84.82 | 0.1753 1.222e+004 3.872e+005 | 1.000 |
|---------|-------|-------|------------------------------|-------|
| 96.00 * | 49.90 | 51.58 | -1.677 1.380e+004 5.184e+005 | 1.000 |
| 120.0 * | 29.10 | 31.36 | -2.261 1.473e+004 6.174e+005 | 1.000 |
| 144.0 * | 19.60 | 19.07 | 0.5309 1.531e+004 6.931e+005 | 1.000 |
| 168.0 * | 12.00 | 11.59 | 0.4051 1.568e+004 7.507e+005 | 1.000 |

\*) Starred values were included in the estimation of Lambda\_z.

## Final Parameters

| Rsq | | 0.9986 |
|--------------------|------------|-------------|
| Rsq_adjusted | | 0.9984 |
| Corr XY | | -0.9993 |
| No_points_lambda_z | | 8 |
| Lambda z | 1/h | 0.0207 |
| Lambda_z_lower | h | 36.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 33.4379 |
| Tlag | h | 0.5000 |
| Tmax | h | 24.0167 |
| Cmax | ng/mL | 267.0000 |
| Cmax D | ng/mL/mg | 0.5933 |
| Tlast | Ĭ h | 168.0000 |
| Clast | ng/mL | 12.0000 |
| AUClast | h*ng/mL | 15676.9265 |
| AUCall | h*ng/mL | 15676.9265 |
| AUCINF_obs | h*ng/mL | 16255.8149 |
| AUCINF_D_obs | h*ng/mL/mg | 36.1240 |
| AUC_%Extrap_obs | % | 3.5611 |
| Vz_F_obs | L | 1335.4184 |
| Cl_F_obs | L/h | 27.6824 |
| AUCINF_pred | h*ng/mL | 16236.2731 |
| AUCINF_D_pred | h*ng/mL/mg | 36.0806 |
| AUC_%Extrap_pred | % | 3.4450 |
| Vz_F_pred | L | 1337.0257 |
| Cl_F_pred | L/h | 27.7157 |
| AUMClast | h*h*ng/mL | 750689.4744 |
| AUMCINF_obs | h*h*ng/mL | 875868.7062 |
| AUMC_%Extrap_obs | % | 14.2920 |
| AUMCINF_pred | h*h*ng/mL | 871642.9765 |
| AUMC_%Extrap_pred | % | 13.8765 |
| MRTlast | h | 47.8850 |
| MRTINF_obs | h | 53.8803 |
| MRTINF_pred | h | 53.6849 |
| AUC0_24 | h*ng/mL | 4969.9879 |
| | _ | |

WinNonlin 7.0.0.2535

PARAMCD=TEPO,SUBJID=PI ,APERIOD=1,TRTAN=1,TRTA=5 x 100 mg TF3

Date: PI 09:23:21 Time:


## Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 450.00 Dose amount:

Calculation method: Linear Trapezoidal Rule for for Increasing Values, Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

```
000000000000000000
0 \ 00 \ 0 \ 000 \ 0 \ 000 \ 0 \ 000 \ 0
^\circ
0 00 0 0 0 000 00 00 00 00 0 0 0 0
```

Date: PI 09:23:24 Time:


### Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 45 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values, Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

### Summary Table

| Time | Conc. | Pred. | Residual | AUC | AUMC | Weight |
|---------|--------|-------|----------|-------------|-----------|--------|
| h | ng/mL | ng/mL | ng/mL | h*ng/mL | h*h*ng/mL | |
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.500 | 17.50 | | | 4.375 | 6.563 | |
| 2.000 | 20.20 | | | 13.80 | 23.23 | |
| 3.000 | 70.40 | | | 59.10 | 149.0 | |
| 4.000 | 106.0 | | | 147.3 | 466.6 | |
| 6.000 | 202.0 | | | 455.3 | 2103. | |
| 8.000 | 203.0 | | | 860.3 | 4939. | |
| 12.00 | 172.0 | | | 1609. 1.238 | 8e+004 | |
| 16.00 | 147.0 | | | 2245. 2.126 | e+004 | |
| 24.00 | 129.0 | | | 3348. 4.321 | e+004 | |
| 36.00 * | 122.0 | 119.3 | 2.733 | 4853. 8.83 | 0e+004 | 1.000 |
| 48.00 * | 86.30 | 87.78 | -1.479 | 6091. 1.39 | 8e+005 | 1.000 |
| 60.00 * | 64.40 | 64.60 | -0.2049 | 6989. 1.88 | 1e+005 | 1.000 |
| 72.00 * | 48.40 | 47.55 | 0.8514 | 7661. 2.32 | 2e+005 | 1.000 |
| 96.00 * | 25.30 | 25.76 | -0.4562 | 8515. 3.02 | 9e+005 | 1.000 |
| 120.0 * | 13.40 | 13.95 | -0.5517 | 8965. 3.50 | 9e+005 | 1.000 |
| 144.0 * | 7.850 | 7.557 | 0.2926 | 9214. 3.83 | Se+005 | 1.000 |
| 168.0 | 0.0000 | | | 9308. 3.97 | 1e+005 | |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

### Final Parameters

| Rsq | | 0.9993 |
|--------------------|----------|-----------|
| Rsq_adjusted | | 0.9991 |
| Corr XY | | -0.9996 |
| No_points_lambda_z | | 7 |
| Lambda_z | 1/h | 0.0255 |
| Lambda_z_lower | h | 36.0000 |
| Lambda_z_upper | h | 144.0000 |
| HL_Lambda_z | h | 27.1346 |
| Tlag | h | 1.0000 |
| Tmax | h | 8.0000 |
| Cmax | ng/mL | 203.0000 |
| Cmax_D | ng/mL/mg | 0.4511 |
| Tlast | h | 144.0000 |
| Clast | ng/mL | 7.8500 |
| AUClast | h*ng/mL | 9213.9288 |
| AUCall | h*ng/mL | 9308.1288 |
| AUCINF_obs | h*ng/mL | 9521.2320 |

AUCINF\_D\_obs 21.1583 h\*ng/mL/mg AUC\_%Extrap\_obs Vz\_F\_obs 3.2276 1850.1917 CI F obs L/h 47.2628 AUCINF\_pred AUCINF\_D\_pred h\*ng/mL 9509.7772 21.1328 h\*ng/mL/mg AUC\_%Extrap\_pred 3.1110 Vz\_F\_pred 1852.4203 L CI\_F\_pred AUMClast L/h 47.3197 h\*h\*ng/mL 383506.7812 AUMCINF\_obs h\*h\*ng/mL 439788.4020 AUMC %Extrap\_obs 12.7974 AUMCINF\_pred 437690.4856 h\*h\*ng/mL AUMC\_%Extrap\_pred 12.3795 MRTlast 41.6225 h MRTINF obs h 46.1903 MRTINF\_pred 46.0253 h AUC0\_24 h\*ng/mL 3347.7131

WinNonlin 7.0.0.2535

PARAMCD=TEPO, SUBJID=pj ,APERIOD=2, TRTAN=1, TRTA=5 x 100 mg TF3

Date: p Time:

09:23:23


## Settings

-----

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

## Summary Table

Weight AUC AUMC Time Conc. Pred. Residual h\*ng/mL h\*h\*ng/mL h ng/mL ng/mL ng/mL 0.0000 0.0000 0.0000 0.0000 0.2500 0.0000 0.0000 0.0000 0.5000 0.0000 0.0000 0.0000 0.7500 5.330 0.6663 0.4997 1.017 9.260 2.612 2.288 1.500 17.80 9.151 11.02 2.000 46.00 25.10 40.69 3.000 89.80 211.8 83.40 4.000 115.0 189.0 566.9 549.0 6.000 245.0 2497. 8.000 263.0 1057. 6071. 12.00 257.0 2097. 1.646e+004 16.00 3151. 3.127e+004 270.0 24.02 279.0 5352. 7.544e+004 36.00 8586. 1.723e+005 261.0 48.00 255.0 1.168e+004 3.022e+005 1.440e+004 4.486e+005 60.00 201.0 72.00 174.0 1.665e+004 5.966e+005 96.00 95.40 1.979e+004 8.565e+005 120.0 \* 48.84 0.1551 2.146e+004 1.035e+006 1.000 49.00 144.0 \* 30.80 31.00 -0.1956 2.240e+004 1.158e+006 1.000 168.1 \* 19.64 0.06215 2.300e+004 1.251e+006 1.000 19.70

### \*) Starred values were included in the estimation of Lambda\_z.

## Final Parameters

| Rsq | | 0.9999 |
|--------------------|------------|--------------|
| Rsq_adjusted | | 0.9997 |
| Corr XY | | -0.9999 |
| No_points_lambda_z | | 3 |
| Lambda z | 1/h | 0.0190 |
| Lambda_z_lower | h | 120.0333 |
| Lambda_z_upper | h | 168.0500 |
| HL_Lambda_z | h | 36.5265 |
| Tlag | h | 0.5000 |
| Tmax | h | 24.0167 |
| Cmax | ng/mL | 279.0000 |
| Cmax_D | ng/mL/mg | 0.6200 |
| Tlast | h | 168.0500 |
| Clast | ng/mL | 19.7000 |
| AUClast | h*ng/mL | 23000.4030 |
| AUCall | h*ng/mL | 23000.4030 |
| AUCINF_obs | h*ng/mL | 24038.5264 |
| AUCINF_D_obs | h*ng/mL/mg | 53.4189 |
| AUC_%Extrap_obs | % | 4.3186 |
| Vz_F_obs | L | 986.4780 |
| CI_F_obs | L/h | 18.7199 |
| AUCINF_pred | h*ng/mL | 24035.2514 |
| AUCINF_D_pred | h*ng/mL/mg | 53.4117 |
| AUC_%Extrap_pred | % | 4.3055 |
| Vz_F_pred | L | 986.6124 |
| Cl_F_pred | L/h | 18.7225 |
| AUMClast | h*h*ng/mL | 1250878.2518 |
| AUMCINF_obs | h*h*ng/mL | 1480040.4739 |
| AUMC_%Extrap_obs | % | 15.4835 |
| AUMCINF_pred | h*h*ng/mL | 1479317.5414 |
| AUMC_%Extrap_pred | % | 15.4422 |
| MRTlast | h | 54.3851 |
| MRTINF_obs | h | 61.5695 |
| MRTINF_pred | h | 61.5478 |
| AUC0_24 | h*ng/mL | 5346.8801 |

WinNonlin 7.0.0.2535

PARAMCD=TEPO, SUBJID=PI ,APERIOD=2,TRTAN=1,TRTA=5 x 100 mg TF3

Date: PI 09:23:21 Time:


## Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 18

Dose time: 0.00 450.00 Dose amount:

Calculation method: Linear Trapezoidal Rule for for Increasing Values, Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

| Time | Conc. | Pred. | Residual | AUC | AUMC | Weight |
|---|---|---|---|---|---|---|
| h | ng/mL | ng/mL | ng/mL | h*ng/mL | h*h*ng/mL | |
| 0.0000<br>0.2500 | 0.0000 | | | | 0.0000<br>0.0000 | |

| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
|---------|--------|-------|---------|----------|------------|-------|
| 0.7500 | 5.000 | | | 0.6250 | 0.4688 | |
| 1.000 | 10.30 | | | 2.538 | 2.225 | |
| 1.500 | 22.00 | | | 10.61 | 13.05 | |
| 2.000 | 38.80 | | | 25.81 | 40.70 | |
| 3.000 | 107.0 | | | 98.71 | 240.0 | |
| 4.000 | 143.0 | | | 223.7 | 686.5 | |
| 6.000 | 244.0 | | | 610.7 | 2723. | |
| 8.000 | 240.0 | | | 1095. | 6109. | |
| 12.00 | 201.0 | | | 1974. 1. | .485e+004 | |
| 16.00 | 147.0 | | | 2665.2. | .445e+004 | |
| 24.00 | 112.0 | | | 3694. 4. | .485e+004 | |
| 36.00 | 92.60 | | | 4918. 8. | .134e+004 | |
| 48.00 * | 68.80 | 68.47 | 0.3324 | 5880. 1 | 1.214e+005 | 1.000 |
| 60.00 * | 54.90 | 55.43 | -0.5344 | 6619. 1 | 1.612e+005 | 1.000 |
| 72.00 * | 45.10 | 44.88 | 0.2179 | 7217. 2 | 2.005e+005 | 1.000 |

\*) Starred values were included in the estimation of Lambda\_z.

#### Final Parameters

Rsq 0.9984 Rsq\_adjusted 0.9968 Corr\_XY -0.9992 No\_points\_lambda\_z 3 Lambda\_z 1/h 0.0176 48.0000 Lambda\_z\_lower h Lambda\_z\_upper h 72.0000 39.3907 HL\_Lambda\_z h Tlag h 0.5000 Tmax h 6.0000 Cmax ng/mL 244.0000 Cmax\_D ng/mL/mg 0.5422 72.0000 Tlast h Clast ng/mL 45.1000 AUClast h\*ng/mL 7216.8292 AUCall h\*ng/mL 7216.8292 9779.8055 AUCINF\_obs h\*ng/mL AUCINF\_D\_obs AUC\_%Extrap\_obs h\*ng/mL/mg 21.7329 26.2068 2614.8715 Vz\_F\_obs L CI\_F\_obs AUCINF\_pred L/h 46.0132 h\*ng/mL 9767.4225 AUCINF\_D\_pred h\*ng/mL/mg 21.7054 AUC\_%Extrap\_pred Vz\_F\_pred 26.1133 2618.1866 L CI\_F\_pred AUMClast L/h 46.0715 h\*h\*ng/mL 200528.3458 AUMCINF\_obs h\*h\*ng/mL 530713.3641 AUMC\_%Extrap\_obs 62.2153 AUMCINF\_pred h\*h\*ng/mL 529118.0731 AUMC\_%Extrap\_pred 62.1014 27.7862 MRTlast h MRTINF\_obs h 54.2662 MRTINF\_pred 54.1717 h AUC0 24 h\*ng/mL 3694.4375

WinNonlin 7.0.0.2535

PARAMCD=TEPO,SUBJID=pj ,APERIOD=1,TRTAN=2,TRTA=2 x 250 mg TF3

Date: pj Time: 09:23:23

WINNONLIN NONCOMPARTMENTAL ANALYSIS PROGRAM 7.0.0.2535 Core Version 04Jun2007

Settings

```
000000000
0 0 0 0 0 0 0 0 0 0 0 0 0
0000000000000000000
0\ 00\ 0\ 000\ 0\ 00\ 0\ 0\ 00
^{\,0} ^{\,0
```

AUMC\_%Extrap\_obs 11.6469 AUMCINF\_pred 474991.6570 h\*h\*ng/mL AUMC\_%Extrap\_pred 10.8133 MRTlast 43.9893 h MRTINF\_obs MRTINF\_pred 48.4922 h 48.1395 h AUC0\_24 h\*ng/mL 3639.0276

WinNonlin 7.0.0.2535

PARAMCD=TEPO,SUBJID=pj ,APERIOD=1,TRTAN=2,TRTA=2 x 250 mg TF3

Date: PI Time: 09:23:23


### Settings

----

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

## Summary Table

| Time | Conc. | Pred. | Residual | AUC | AUMC | Weight |
|---------|--------|-------|----------|-------------|-------------|--------|
| h | ng/mL | ng/mL | ng/mL | h*ng/mL | . h*h*ng/mL | |
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 2.000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 3.000 | 11.60 | | | 5.800 | 17.40 | |
| 4.000 | 30.20 | | | 26.70 | 95.20 | |
| 6.000 | 106.0 | | | 162.9 | 852.0 | |
| 8.000 | 109.0 | | | 377.9 | 2360. | |
| 12.00 | 100.0 | | | 795.6 | 6525. | |
| 16.00 | 90.50 | | | 1176. 1.184 | 4e+004 | |
| 24.00 | 100.0 | | | 1938. 2.72 | 3e+004 | |
| 36.00 * | 96.70 | 94.41 | 2.286 | 3118.6.26 | 0e+004 | 1.000 |
| 48.00 * | 68.60 | 71.08 | -2.480 | 4101. 1.03 | 5e+005 | 1.000 |
| 60.00 * | 51.90 | 53.51 | -1.613 | 4819. 1.42 | 1e+005 | 1.000 |
| 72.00 * | 41.00 | 40.29 | 0.7125 | 5374. 1.78 | 86e+005 | 1.000 |
| 96.00 * | 24.10 | 22.83 | 1.265 | 6137. 2.41 | 9e+005 | 1.000 |
| 120.0 * | 12.70 | 12.94 | -0.2424 | 6564. 2.87 | 75e+005 | 1.000 |
| 144.0 * | 7.260 | 7.336 | -0.07559 | 6798. 3.18 | 80e+005 | 1.000 |
| 168.0 | 0.0000 | | | 6885. 3.30 | 6e+005 | |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

## Final Parameters

| Rsq | | 0.9988 |
|--------------------|-----|---------|
| Rsq_adjusted | | 0.9985 |
| Corr_XY | | -0.9994 |
| No_points_lambda_z | | 7 |
| Lambda_z | 1/h | 0.0237 |
| Lambda_z_lower | h | 36.0000 |

| Lambda_z_upper | h | 144.0000 |
|-------------------|------------|-------------|
| HL_Lambda_z | h | 29.2999 |
| Tlag | h | 2.0000 |
| Tmax | h | 8.0000 |
| Cmax | ng/mL | 109.0000 |
| Cmax_D | ng/mL/mg | 0.2422 |
| Tlast | h | 144.0000 |
| Clast | ng/mL | 7.2600 |
| AUClast | h*ng/mL | 6797.6504 |
| AUCall | h*ng/mL | 6884.7704 |
| AUCINF_obs | h*ng/mL | 7104.5362 |
| AUCINF_D_obs | h*ng/mL/mg | 15.7879 |
| AUC_%Extrap_obs | % | 4.3196 |
| Vz_F_obs | L | 2677.4229 |
| Cl_F_obs | L/h | 63.3398 |
| AUCINF_pred | h*ng/mL | 7107.7313 |
| AUCINF_D_pred | h*ng/mL/mg | 15.7950 |
| AUC_%Extrap_pred | % | 4.3626 |
| Vz_F_pred | L | 2676.2193 |
| Cl_F_pred | L/h | 63.3113 |
| AUMClast | h*h*ng/mL | 318043.2142 |
| AUMCINF_obs | h*h*ng/mL | 375207.0721 |
| AUMC_%Extrap_obs | % | 15.2353 |
| AUMCINF_pred | h*h*ng/mL | 375802.2394 |
| AUMC_%Extrap_pred | % | 15.3695 |
| MRTlast | h | 46.7872 |
| MRTINF_obs | h | 52.8123 |
| MRTINF_pred | h | 52.8723 |
| AUC0_24 | h*ng/mL | 1938.3255 |

WinNonlin 7.0.0.2535 PARAMCD=TEPO,SUBJID=PI ,APERIOD=1,TRTAN=2,TRTA=2 x 250 mg TF3

> Date: PI 09:23:22 Time:


### Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

| Time | Conc. | Pred. | Residual | AUC | AUMC | Weight |
|--------|--------|-------|----------|------------|-------------|--------|
| h | ng/mL | ng/mL | ng/mL | h*ng/m | L h*h*ng/mL | |
| | | | | | • | |
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.000 | 7.290 | | | 0.9113 | 0.9113 | |
| 1.500 | 15.70 | | | 6.659 | 8.621 | |
| 2.000 | 35.70 | | | 19.51 | 32.36 | |
| 3.000 | 78.50 | | | 76.61 | 185.8 | |
| 4.000 | 106.0 | | | 168.9 | 515.6 | |
| 6.000 | 175.0 | | | 449.9 | 1990. | |
| 8.017 | 214.0 | | | 842.1 | 4778. | |
| 12.00 | 246.0 | | | 1758. 1.40 | 07e+004 | |
| 16.00 | 252.0 | | | 2754. 2.80 | 04e+004 | |

| 24.00 | 262.0 | | 4810. 6.932e+004 | |
|---------|-------|-------|-------------------------------|-------|
| 36.00 | 267.0 | | 7984. 1.647e+005 | |
| 48.00 | 281.0 | | 1.127e+004 3.033e+005 | |
| 60.03 | 245.0 | | 1.443e+004 4.736e+005 | |
| 72.00 | 201.0 | | 1.709e+004 6.486e+005 | |
| 96.03 * | 105.0 | 103.5 | 1.511 2.065e+004 9.426e+005 | 1.000 |
| 120.0 * | 64.50 | 65.17 | -0.6747 2.264e+004 1.156e+006 | 1.000 |
| 144.0 * | 40.10 | 41.02 | -0.9190 2.387e+004 1.317e+006 | 1.000 |
| 168.0 * | 26.30 | 25.82 | 0.4838 2.465e+004 1.439e+006 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

### Final Parameters

| Rsq | | 0.9989 |
|--------------------|------------|--------------|
| Rsq_adjusted | | 0.9984 |
| Corr XY | | -0.9995 |
| No_points_lambda_z | | 4 |
| Lambda_z | 1/h | 0.0193 |
| Lambda_z_lower | h | 96.0333 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 35.9271 |
| Tlag | h | 0.7500 |
| Tmax | h | 48.0000 |
| Cmax | ng/mL | 281.0000 |
| Cmax_D | ng/mL/mg | 0.6244 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 26.3000 |
| AUClast | h*ng/mL | 24654.2933 |
| AUCall | h*ng/mL | 24654.2933 |
| AUCINF_obs | h*ng/mL | 26017.4726 |
| AUCINF_D_obs | h*ng/mL/mg | 57.8166 |
| AUC_%Extrap_obs | % | 5.2395 |
| Vz_F_obs | L | 896.4883 |
| Cl_F_obs | L/h | 17.2961 |
| AUCINF_pred | h*ng/mL | 25992.3942 |
| AUCINF_D_pred | h*ng/mL/mg | 57.7609 |
| AUC_%Extrap_pred | % | 5.1480 |
| Vz_F_pred | L | 897.3533 |
| Cl_F_pred | L/h | 17.3128 |
| AUMClast | h*h*ng/mL | 1439103.8570 |
| AUMCINF_obs | h*h*ng/mL | 1738774.1565 |
| AUMC_%Extrap_obs | % | 17.2346 |
| AUMCINF_pred | h*h*ng/mL | 1733261.1376 |
| AUMC_%Extrap_pred | % | 16.9713 |
| MRTlast | h | 58.3713 |
| MRTINF_obs | h | 66.8310 |
| MRTINF_pred | h | 66.6834 |
| AUC0_24 | h*ng/mL | 4810.2671 |

WinNonlin 7.0.0.2535

PARAMCD=TEPO,SUBJID=PI ,APERIOD=2,TRTAN=2,TRTA=2 x 250 mg TF3

PI 09:23:22 Date: Time:


## Settings

Model: Plasma Data, Extravascular Administration Number of nonmissing observations: 22

Dose time:

450.00 Dose amount:

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

```
0\;0\;0\;0\;0\;0\;0\;0\;0\;0\;0
000000000000000000
0 \ 00 \ 0 \ 000 \ 0 \ 000 \ 0 \ 000 \ 0
0 \  \, \varpi \  \, 0 \  \, \varpi \  \, 0 \  \, \varpi \  \, 0 \  \, 
0 \  \, 
^{\circ}
```
PARAMCD=TEPO, SUBJID=pj ,APERIOD=2, TRTAN=2, TRTA=2 x 250 mg TF3

Date: Time:

09:23:22

## WINNONLIN NONCOMPARTMENTAL ANALYSIS PROGRAM 7.0.0.2535 Core Version 04Jun2007

## Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values, Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

## Summary Table

| Time<br>h | Conc.<br>ng/mL | Pred.<br>ng/mL | Residual<br>ng/mL | AUC<br>h*ng/mL | AUMC<br>h*h*ng/mL | Weight |
|---|---|---|---|---|---|---|
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.000 | 6.740 | | ( | 0.8425 0 | .8425 | |
| 1.500 | 15.70 | | | 6.453 | 3.415 | |
| 2.000 | 39.40 | | | 20.23 | 34.00 | |
| 3.000 | 88.80 | | | 84.33 | 206.6 | |
| 4.000 | 106.0 | | | 181.7 | 551.8 | |
| 6.017 | 168.0 | | | 458.0 | 1999. | |
| 8.000 | 178.0 | | | 801.1 | <b>14</b> 13. | |
| 12.00 | 182.0 | | | 1521. 1.163 | e+004 | |
| 16.10 | 190.0 | | | 2284. 2.238 | e+004 | |
| 24.07 | 187.0 | | | 3785. 5.252 | e+004 | |
| 36.00 | 179.0 | | | 5969. 1.180 | e+005 | |
| 48.00 * | 149.0 | 159.1 | -10.12 | 7931. 2.001 | e+005 | 1.000 |
| 60.02 * | 122.0 | 120.4 | 1.631 | 9554. 2.87 | <del>1e+</del> 005 | 1.000 |
| 72.00 * | 96.70 | 91.13 | 5.573 1.08 | 36e+004 3.73 | 2e+005 | 1.000 |
| 96.17 * | 55.70 | 51.99 | 3.713 1.26 | Se+004 5.22 | 2e+005 | 1.000 |
| 120.0 * | 28.40 | 29.89 | -1.489 1.36 | 2e+004 6.25 | 4e+005 | 1.000 |
| 146.9 * | 14.70 | 15.99 | -1.290 1.41 | 8e+004 6.99 | 3e+005 | 1.000 |
| 168.0 * | 10.40 | 9.803 | 0.5968 1.4 | 44e+004 7.40 | 04e+005 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

## Final Parameters

| Rsq | | 0.9961 |
|--------------------|----------|----------|
| Rsq_adjusted | | 0.9953 |
| Corr_XY | | -0.9981 |
| No_points_lambda_z | | 7 |
| Lambda_z | 1/h | 0.0232 |
| Lambda_z_lower | h | 48.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 29.8456 |
| Tlag | h | 0.7500 |
| Tmax | h | 16.1000 |
| Cmax | ng/mL | 190.0000 |
| Cmax_D | ng/mL/mg | 0.4222 |
| Tlast | h | 168.0000 |

Clast ng/mL 10.4000 **AUClast** h\*ng/mL 14442.9440 **AUCall** h\*ng/mL 14442.9440 AUCINF\_obs 14890.7483 h\*ng/mL AUCINF\_D\_obs AUC\_%Extrap\_obs h\*ng/mL/mg 33.0906 3.0073 Vz\_F\_obs Cl\_F\_obs L 1301.2206 30.2201 L/h AUCINF\_pred AUCINF\_D\_pred h\*ng/mL 14865.0506 h\*ng/mL/mg 33.0334 AUC\_%Extrap\_pred % 2.8396 Vz\_F\_pred Cl\_F\_pred L 1303.4700 L/h 30.2723 **AUMClast** h\*h\*ng/mL 740382.3484 AUMCINF\_obs h\*h\*ng/mL 834895.0777 AUMC %Extrap obs 11.3203 AUMCINF\_pred 829471.3823 h\*h\*ng/mL AUMC\_%Extrap\_pred 10.7405 MRTlast 51.2626 h MRTINF\_obs 56.0680 h MRTINF\_pred 55.8001 h AUC0\_24 h\*ng/mL 3772.9450

WinNonlin 7.0.0.2535

PARAMCD=TEPO, SUBJID=PI ,APERIOD=2, TRTAN=2, TRTA=2 x 250 mg TF3

Date: PI Time: 09:23:22


# Settings

-----

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00

Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

| Time | Conc. | Pred. | Residual | AUC | AUMC | Weight |
|---------|--------|-------|------------|--------------|-----------|--------|
| h | ng/mL | ng/mL | ng/mL | h*ng/mL | h*h*ng/mL | |
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | | 0.0000 | |
| 0.7500 | 0.0000 | | | | 0.0000 | |
| 1.000 | 7.880 | | | | .9850 | |
| 1.500 | 12.80 | | | | 7.755 | |
| 2.000 | 23.70 | | | | 24.41 | |
| 3.000 | 74.60 | | | | 160.0 | |
| 4.000 | 121.0 | | | | 513.9 | |
| 6.000 | 215.0 | | | | 2288. | |
| 8.000 | 231.0 | | | 944.2 | 5426. | |
| 12.00 | 210.0 | | | 1826. 1.421 | e+004 | |
| 16.00 | 186.0 | | | 2617, 2,525 | e+004 | |
| 24.02 | 166.0 | | | 4026, 5,335 | e+004 | |
| 36.00 | 189.0 | | | 6153, 1,180 | e+005 | |
| 48.00 | 175.0 | | | 8336, 2,095 | e+005 | |
| 60.00 | 156.0 | | 1.03 | 32e+004 3.16 | | |
| 72.00 | 118.0 | | | 95e+004 4.23 | | |
| 96.00 | 92.70 | | | 47e+004 6.33 | | |
| | | | | | | 4 000 |
| 120.0 * | 54.60 | 54.45 | 0.1531 1.6 | 20e+004 8.18 | 88e+005 | 1.000 |

144.0 \* 33.10 33.29 -0.1864 1.723e+004 9.538e+005 1.000 168.0 \* 20.40 20.34 0.05717 1.786e+004 1.051e+006 1.000

\*) Starred values were included in the estimation of Lambda\_z.

Final Parameters

Rsq 0.9999 Rsq\_adjusted 0.9998 Corr\_XY -1.0000 No\_points\_lambda\_z 3 Lambda z 0.0205 1/h Lambda\_z\_lower 120.0167 h Lambda\_z\_upper h 168.0000 HL\_Lambda\_z 33.7833 h Tlag h 0.7500 Tmax h 8.0000 231.0000 Cmax ng/mL 0.5133 Cmax\_D ng/mL/mg 168.0000 Tlast h Clast ng/mL 20.4000 **AUClast** 17858.0511 h\*ng/mL AUCall h\*ng/mL 17858.0511 AUCINF\_obs AUCINF\_D\_obs h\*ng/mL 18852.3253 h\*ng/mL/mg 41.8941 AUC\_%Extrap\_obs 5.2740 Vz\_F\_obs L 1163.3854 CI\_F\_obs L/h 23.8697 AUCINF\_pred 18849.5389 h\*ng/mL AUCINF\_D\_pred h\*ng/mL/mg 41.8879 AUC\_%Extrap\_pred Vz\_F\_pred % 5.2600 L 1163.5573 CI\_F\_pred AUMClast L/h 23.8733 h\*h\*ng/mL 1051407.0812 AUMCINF\_obs h\*h\*ng/mL 1266905.0092 AUMC\_%Extrap\_obs 17.0098 h\*h\*ng/mL AUMCINF\_pred 1266301.0863 AUMC\_%Extrap\_pred 16.9702 MRTlast 58.8758 MRTINF obs 67.2015 h MRTINF\_pred 67.1794 h AUC0 24 h\*ng/mL 4023.2390

WinNonlin 7.0.0.2535

PARAMCD=TEPO,SUBJID=PI ,APERIOD=2,TRTAN=2,TRTA=2 x 250 mg TF3

Date: pj Time: 09:23:23


Settings

-----

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00

Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

Summary Table

··---

Time Conc. Pred. Residual AUC AUMC Weight

| h | ng/mL | ng/mL | ng/mL | h*ng/mL | h*h*ng/r | nL |
|---------|--------|-------|--------------|--------------|----------|-------|
| 0.0000 | 0.0000 | | | | 0.0000 | |
| 0.2500 | 0.0000 | | | | 0.0000 | |
| 0.5000 | 0.0000 | | | | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.000 | 6.030 | | | 0.7538 ( | ).7538 | |
| 1.500 | 20.50 | | | 7.386 | 9.949 | |
| 2.000 | 35.80 | | | 21.46 | 35.54 | |
| 3.000 | 112.0 | | | 95.36 | 239.3 | |
| 4.000 | 176.0 | | | 239.4 | 759.3 | |
| 6.000 | 212.0 | | | 627.4 | 2735. | |
| 8.000 | 224.0 | | | 1063. | 5799. | |
| 12.00 | 233.0 | | | 1977. 1.498 | e+004 | |
| 16.00 | 213.0 | | | 2869. 2.743 | e+004 | |
| 24.02 | 231.0 | | | 4648. 6.333 | e+004 | |
| 36.00 | 225.0 | | | 7381. 1.452 | e+005 | |
| 48.00 | 175.0 | | | 9768. 2.449 | e+005 | |
| 60.00 | 176.0 | | 1.18 | 37e+004 3.58 | 37e+005 | |
| 72.00 | 164.0 | | 1.39 | 1e+004 4.93 | 31e+005 | |
| 96.00 | 112.0 | | 1.71 | 9e+004 7.65 | 5e+005 | |
| 120.0 * | 59.10 | 59.20 | -0.1041 1.91 | 17e+004 9.7 | 75e+005 | 1.000 |
| 144.0 * | 35.50 | 35.38 | 0.1248 2.0 | 28e+004 1.1 | 23e+006 | 1.000 |
| 168.0 * | 21.10 | 21.14 | -0.03717 2.0 | 95e+004 1.2 | 26e+006 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

| Rsq | | 1.0000 |
|--------------------|------------|--------------|
| Rsq_adjusted | | 0.9999 |
| Corr_XY | | -1.0000 |
| No_points_lambda_z | | 3 |
| Lambda z | 1/h | 0.0215 |
| Lambda_z_lower | h | 120.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 32.3033 |
| Tlag | h | 0.7500 |
| Tmax | h | 12.0000 |
| Cmax | ng/mL | 233.0000 |
| Cmax_D | ng/mL/mg | 0.5178 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 21.1000 |
| AUClast | h*ng/mL | 20947.0902 |
| AUCall | h*ng/mL | 20947.0902 |
| AUCINF_obs | h*ng/mL | 21930.4314 |
| AUCINF_D_obs | h*ng/mL/mg | 48.7343 |
| AUC_%Extrap_obs | % | 4.4839 |
| Vz_F_obs | L | 956.2845 |
| Cl_F_obs | L/h | 20.5194 |
| AUCINF_pred | h*ng/mL | 21932.1638 |
| AUCINF_D_pred | h*ng/mL/mg | 48.7381 |
| AUC_%Extrap_pred | % | 4.4915 |
| Vz_F_pred | L | 956.2089 |
| Cl_F_pred | L/h | 20.5178 |
| AUMClast | h*h*ng/mL | 1225971.4686 |
| AUMCINF_obs | h*h*ng/mL | 1437000.2689 |
| AUMC_%Extrap_obs | % | 14.6854 |
| AUMCINF_pred | h*h*ng/mL | 1437372.0569 |
| AUMC_%Extrap_pred | % | 14.7074 |
| MRTlast | h | 58.5271 |
| MRTINF_obs | h | 65.5254 |
| MRTINF_pred | h | 65.5372 |
| AUC0_24 | h*ng/mL | 4644.6133 |
| | _ | |

WinNonlin 7.0.0.2535 PARAMCD=TEPO, SUBJID= $\underline{PI}$  ,APERIOD=2, TRTAN=2, TRTA=2 x 250 mg TF3

Date: Pl

```
0 0 0000 0 0 0
000000000
00000000000000000
```

| Cl_F_obs | L/h | 37.8337 |
|-------------------|------------|-------------|
| AUCINF_pred | h*ng/mL | 11863.9452 |
| AUCINF_D_pred | h*ng/mL/mg | 26.3643 |
| AUC_%Extrap_pred | % | 2.5832 |
| Vz_F_pred | L | 1675.8349 |
| Cl_F_pred | L/h | 37.9300 |
| AUMClast | h*h*ng/mL | 541364.5996 |
| AUMCINF_obs | h*h*ng/mL | 612799.7356 |
| AUMC_%Extrap_obs | % | 11.6572 |
| AUMCINF_pred | h*h*ng/mL | 606390.8933 |
| AUMC_%Extrap_pred | % | 10.7235 |
| MRTlast | h | 46.8411 |
| MRTINF_obs | h | 51.5211 |
| MRTINF_pred | h | 51.1121 |
| AUC0_24 | h*ng/mL | 3679.1063 |

WinNonlin 7.0.0.2535 PARAMCD=TEPO,SUBJID=PI \_\_,APERIOD=1,TRTAN=1,TRTA=5 x 100 mg TF3

> Date: PI 09:23:21 Time:


# Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

| Time<br>h | Conc.<br>ng/mL | Pred.<br>ng/mL | Residual<br>ng/mL | AUC<br>h*ng/mL | AUMC<br>h*h*ng/mL | Weight |
|---|---|---|---|---|---|---|
| 0.0000 | 0.0000 | | | | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.033 | 11.10 | | | 1.572 | 1.625 | |
| 1.500 | 26.90 | | | 10.44 | 13.72 | |
| 2.017 | 34.20 | | | 26.22 | 41.96 | |
| 3.000 | 167.0 | | | 125.1 | 322.2 | |
| 4.000 | 154.0 | | | 285.6 | 882.6 | |
| 6.000 | 230.0 | | | 669.6 | 2879. | |
| 8.000 | 255.0 | | | 1155. | 6299. | |
| 12.00 | 291.0 | | | 2247. 1.736 | e+004 | |
| 16.00 | 298.0 | | | 3425. 3.388 | e+004 | |
| 24.03 | 312.0 | | | 5875. 8.315 | e+004 | |
| 36.00 * | 260.0 | 265.8 | -5.800 | 9288. 1.850 | e+005 | 1.000 |
| 48.00 * | 214.0 | 201.5 | 12.52 1.2 | 12e+004 3.03 | 35e+005 | 1.000 |
| 60.00 * | 144.0 | 152.7 | -8.726 1.42 | 24e+004 4.17 | '2e+005 | 1.000 |
| 72.00 * | 117.0 | 115.8 | 1.231 1.5 | 80e+004 5.19 | 98e+005 | 1.000 |
| 96.00 * | 62.60 | 66.52 | -3.920 1.78 | 89e+004 6.92 | 6e+005 | 1.000 |
| 120.3 * | 43.60 | 37.99 | 5.613 1.9 | 17e+004 8.29 | 95e+005 | 1.000 |
| 144.0 * | 20.90 | 21.96 | -1.062 1.99 | 90e+004 9.25 | 2e+005 | 1.000 |
| 168.0 * | 12.40 | 12.62 | -0.2189 2.0 | 29e+004 9.85 | 8e+005 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

Rsq 0.9961 Rsq\_adjusted 0.9954 -0.9980 Corr\_XY No\_points\_lambda\_z 8 Lambda\_z 0.0231 1/h Lambda\_z\_lower 36.0000 h Lambda\_z\_upper h 168.0000 30.0227 HL\_Lambda\_z h Tlag h 0.7500 Tmax h 24.0333 ng/mL 312.0000 Cmax ng/mL/mg 0.6933 Cmax\_D 168.0000 Tlast h Clast ng/mL 12.4000 **AUClast** 20289.2653 h\*ng/mL AUCall h\*ng/mL 20289.2653 AUCINF\_obs AUCINF\_D\_obs 20826.3535 h\*ng/mL h\*ng/mL/mg 46,2808 AUC\_%Extrap\_obs 2.5789 Vz\_F\_obs 935.8865 L CI\_F\_obs L/h 21.6072 AUCINF\_pred h\*ng/mL 20835.8369 AUCINF\_D\_pred h\*ng/mL/mg 46.3019 AUC\_%Extrap\_pred Vz\_F\_pred 2.6232 935.4606 L CI\_F\_pred L/h 21.5974 **AUM Clast** h\*h\*ng/mL 985802.1871 AUMCINF\_obs h\*h\*ng/mL 1099296.2082 AUMC\_%Extrap\_obs 10.3242 AUMCINF\_pred h\*h\*ng/mL 1101300.1855 AUMC\_%Extrap\_pred 10.4874 48.5874 MRTlast h MRTINF obs 52.7839 h MRTINF\_pred h 52.8561 AUC0\_24 h\*ng/mL 5864.3265

WinNonlin 7.0.0.2535

PARAMCD=TEPO,SUBJID=pj ,APERIOD=2,TRTAN=1,TRTA=5 x 100 mg TF3

Date: pj Time: 09:23:24


# Settings

\_\_\_\_

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

## Summary Table

AUC AUMC Time Conc. Pred. Residual Weight ng/mL ng/mL ng/mL h\*ng/mL h\*h\*ng/mL 0.0000 0.0000 0.0000 0.0000 0.2500 0.0000 0.0000 0.0000 0.5000 7.290 0.4556 0.9113 0.7500 16.00 3.823 2.411 1.000 21.90 8.560 6.649

| 1.500 | 39.40 | | 23.89 26.90 | |
|---------|-------|-------|------------------------------|-------|
| 2.000 | 69.90 | | 51.21 76.62 | |
| 3.000 | 97.10 | | 134.7 292.2 | |
| 4.000 | 195.0 | | 280.8 827.8 | |
| 6.000 | 343.0 | | 818.8 3666. | |
| 8.000 | 363.0 | | 1525. 8628. | |
| 12.00 | 301.0 | | 2849. 2.179e+004 | |
| 16.00 | 278.0 | | 4006. 3.796e+004 | |
| 24.00 * | 273.0 | 286.3 | -13.34 6210. 8.201e+004 | 1.000 |
| 36.00 * | 229.0 | 231.6 | -2.642 9214. 1.716e+005 | 1.000 |
| 48.00 * | 193.0 | 187.4 | 5.607 1.174e+004 2.773e+005 | 1.000 |
| 60.00 * | 149.0 | 151.6 | -2.596 1.378e+004 3.869e+005 | 1.000 |
| 72.00 * | 130.0 | 122.6 | 7.363 1.545e+004 4.970e+005 | 1.000 |
| 96.00 * | 78.70 | 80.26 | -1.559 1.791e+004 7.006e+005 | 1.000 |
| 120.0 * | 53.00 | 52.52 | 0.4752 1.947e+004 8.679e+005 | 1.000 |
| 144.0 * | 37.50 | 34.36 | 3.136 2.054e+004 1.009e+006 | 1.000 |
| 168.0 * | 20.60 | 22.50 | -1.896 2.122e+004 1.114e+006 | 1.000 |

\*) Starred values were included in the estimation of Lambda\_z.

## Final Parameters

| Rsq | | 0.9964 |
|--------------------|------------|--------------|
| Rsq_adjusted | | 0.9958 |
| Corr_XY | | -0.9982 |
| No_points_lambda_z | | 9 |
| Lambda_z | 1/h | 0.0177 |
| Lambda_z_lower | h | 24.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 39.2372 |
| Tlag | h | 0.2500 |
| Tmax | h | 8.0000 |
| Cmax | ng/mL | 363.0000 |
| Cmax_D | ng/mL/mg | 0.8067 |
| Tlast | Ď h | 168.0000 |
| Clast | ng/mL | 20.6000 |
| AUClast | h*ng/mL | 21218.2736 |
| AUCall | h*ng/mL | 21218,2736 |
| AUCINF obs | h*ng/mL | 22384.3851 |
| AUCINF_D_obs | h*ng/mL/mg | 49.7431 |
| AUC_%Extrap_obs | % | 5.2095 |
| Vz_F_obs | L | 1137.9946 |
| CI_F_obs | L/h | 20.1033 |
| AUCINF_pred | h*ng/mL | 22491.7155 |
| AUCINF_D_pred | h*ng/mL/mg | 49.9816 |
| AUC_%Extrap_pred | % | 5.6618 |
| Vz_F_pred | L | 1132.5641 |
| Cl_F_pred | L/h | 20.0074 |
| AUMClast | h*h*ng/mL | 1113944.4494 |
| AUMCINF_obs | h*h*ng/mL | 1375861.6680 |
| AUMC_%Extrap_obs | % | 19.0366 |
| AUMCINF_pred | h*h*ng/mL | 1399968.8604 |
| AUMC_%Extrap_pred | % | 20.4308 |
| MRTlast | h | 52.4993 |
| MRTINF obs | h | 61.4652 |
| MRTINF_pred | h | 62.2438 |
| AUC0_24 | h*ng/mL | 6210.2217 |

WinNonlin 7.0.0.2535 PARAMCD=TEPO,SUBJID=PI ,APERIOD=2,TRTAN=1,TRTA=5 x 100 mg TF3

> Date: Time: PI 09:23:23

WINNONLIN NONCOMPARTMENTAL ANALYSIS PROGRAM 7.0.0.2535 Core Version 04Jun2007

```
\Pi \Pi \Pi \Pi \Pi \Pi \Pi
0 0 0 0 0 00 00 0 0 0 0
\begin{smallmatrix}0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0
0 \  \, \varpi \, 0 \  \, \varpi
```

| AUMCINF_obs | h*h*ng/mL | 809099.4814 |
|-------------------|-----------|-------------|
| AUMC_%Extrap_obs | % | 13.5804 |
| AUMCINF_pred | h*h*ng/mL | 798791.8736 |
| AUMC_%Extrap_pred | % | 12.4653 |
| MRTlast | h | 49.9341 |
| MRTINF_obs | h | 55.7361 |
| MRTINF_pred | h | 55.2093 |
| AUC0 24 | h*ng/mL | 3865.0356 |

WinNonlin 7.0.0.2535 PARAMCD=TEPO, SUBJID=PI ,APERIOD=2,TRTAN=1,TRTA=5 x 100 mg TF3

> Date: PI 09:23:24 Time:


## Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

### Summary Table

| Time | Conc. | Pred. | Residual | AUC | AUMC | Weight |
|---------|--------|-------|--------------|--------------|-----------|--------|
| h | ng/mL | ng/mL | . ng/mL | h*ng/mL | h*h*ng/mL | |
| | | | | | • | |
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 2.000 | 8.690 | | | 2.173 | 4.345 | |
| 3.000 | 15.40 | | | 14.22 | 36.14 | |
| 4.000 | 37.30 | | | 40.57 | 133.8 | |
| 6.000 | 164.0 | | | 241.9 | 1267. | |
| 8.000 | 176.0 | | | 581.9 | 3659. | |
| 12.00 | 217.0 | | | 1368. 1.168 | e+004 | |
| 16.00 | 226.0 | | | 2254. 2.412 | e+004 | |
| 24.00 | 194.0 | | | 3931. 5.749 | e+004 | |
| 36.00 | 117.0 | | | 5758. 1.114 | e+005 | |
| 48.00 | 106.0 | | | 7095. 1.674 | e+005 | |
| 60.00 | 80.60 | | | 8207. 2.272 | e+005 | |
| 72.00 | 53.60 | | | 9002. 2.793 | e+005 | |
| 96.00 * | 42.20 | 40.78 | 1.415 1.0 | 15e+004 3.74 | 48e+005 | 1.000 |
| 120.0 * | 21.70 | 23.24 | -1.535 1.0 | 89e+004 4.53 | 88e+005 | 1.000 |
| 144.0 * | 13.70 | 13.24 | 0.4631 1.1 | 30e+004 5.0 | 85e+005 | 1.000 |
| 168.0 * | 7.540 | 7.541 | -0.001047 1. | 155e+004 5.4 | 68e+005 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

## Final Parameters

| Rsq | | 0.9956 |
|--------------------|-----|---------|
| Rsq_adjusted | | 0.9934 |
| Corr_XY | | -0.9978 |
| No_points_lambda_z | | 4 |
| Lambda z | 1/h | 0.0234 |

| Lambda_z_lower | ķ | 96.0000 |
|-------------------|------------|-------------|
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 29.5663 |
| Tlag | h | 1.5000 |
| Tmax | h | 16.0000 |
| Cmax | ng/mL | 226.0000 |
| Cmax_D | ng/mL/mg | 0.5022 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 7.5400 |
| AUClast | h*ng/mL | 11550.5353 |
| AUCall | h*ng/mL | 11550.5353 |
| AUCINF obs | h*ng/mL | 11872.1556 |
| AUCINF_D_obs | h*ng/mL/mg | 26.3826 |
| AUC %Extrap obs | % | 2.7090 |
| Vz F obs | L | 1616.7953 |
| CI F obs | L/h | 37.9038 |
| AUCINF pred | h*ng/mL | 11872,2003 |
| AUCINF D pred | h*ng/mL/mg | 26.3827 |
| AUC %Extrap pred | % | 2,7094 |
| Vz_F_pred | L | 1616.7892 |
| CI F pred | L/h | 37.9037 |
| AUMClast | h*h*ng/mL | 546801.8568 |
| AUMCINF obs | h*h*ng/mL | 614552.8489 |
| AUMC %Extrap obs | % | 11.0244 |
| AUMCINF_pred | h*h*ng/mL | 614562.2575 |
| AUMC %Extrap pred | % | 11.0258 |
| MRTlast | h | 47.3400 |
| MRTINF obs | h | 51.7642 |
| MRTINF_pred | h | 51.7648 |
| AUC0 24 | h*ng/mL | 3930.6117 |
| | ····g···· | 0000.0117 |

WinNonlin 7.0.0.2535

PARAMCD=TEPO, SUBJID=pj ,APERIOD=1,TRTAN=2,TRTA=2 x 250 mg TF3

PI 09:23:24 Date: Time:


## Settings

Model: Plasma Data, Extravascular Administration Number of nonmissing observations: 22

Dose time:

450.00 Dose amount:

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values
Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

| Time<br>h | Conc.<br>ng/mL | Pred.<br>ng/mL | Residual<br>ng/mL | AUC<br>h*ng/mL | AUMC<br>h*h*ng/mL | Weight |
|---|---|---|---|---|---|---|
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 2.000 | 16.20 | | | 4.050 | 8.100 | |
| 3.000 | 27.60 | | | 25.95 | 65.70 | |
| 4.000 | 57.30 | | | 68.40 | 221.7 | |
| 6.000 | 109.0 | | | 234.7 | 1105. | |
| 8.000 | 164.0 | | | 507.7 | 3071. | |
| 12.00 | 215.0 | | | 1266. 1.08 | 5e+004 | |

| 16.00 | 223.0 | | 2142. 2.315e+004 | |
|---------|-------|-------|------------------------------|-------|
| 24.00 | 272.0 | | 4122. 6.353e+004 | |
| 36.00 * | 234.0 | 225.3 | 8.735 7152. 1.540e+005 | 1.000 |
| 48.00 * | 172.0 | 174.1 | -2.053 9569. 2.548e+005 | 1.000 |
| 60.00 * | 131.0 | 134.5 | -3.484 1.138e+004 3.518e+005 | 1.000 |
| 72.00 * | 110.0 | 103.9 | 6.089 1.282e+004 4.468e+005 | 1.000 |
| 96.00 * | 56.20 | 62.04 | -5.835 1.474e+004 6.057e+005 | 1.000 |
| 120.0 * | 38.80 | 37.04 | 1.765 1.587e+004 7.266e+005 | 1.000 |
| 144.0 * | 20.90 | 22.11 | -1.210 1.656e+004 8.174e+005 | 1.000 |
| 168.0 * | 13.90 | 13.20 | 0.7000 1.697e+004 8.813e+005 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

| Rsq | | 0.9968 |
|--------------------|------------|--------------|
| Rsq_adjusted | | 0.9963 |
| Corr_XÝ | | -0.9984 |
| No_points_lambda_z | | 8 |
| Lambda_z | 1/h | 0.0215 |
| Lambda_z_lower | h | 36.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 32.2501 |
| Tlag | h | 1.5000 |
| Tmax | h | 24.0000 |
| Cmax | ng/mL | 272.0000 |
| Cmax_D | ng/mL/mg | 0.6044 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 13.9000 |
| AUClast | h*ng/mL | 16974.2217 |
| AUCall | h*ng/mL | 16974.2217 |
| AUCINF_obs | h*ng/mL | 17620.9485 |
| AUCINF_D_obs | h*ng/mL/mg | 39.1577 |
| AUC_%Extrap_obs | % | 3.6702 |
| Vz_F_obs | L | 1188.1994 |
| CI_F_obs | L/h | 25.5378 |
| AUCINF_pred | h*ng/mL | 17588.3816 |
| AUCINF_D_pred | h*ng/mL/mg | 39.0853 |
| AUC_%Extrap_pred | % | 3.4918 |
| Vz_F_pred | L | 1190.3995 |
| CI_F_pred | L/h | 25.5851 |
| AUMClast | h*h*ng/mL | 881344.2543 |
| AUMCINF_obs | h*h*ng/mL | 1020084.6943 |
| AUMC_%Extrap_obs | % | 13.6009 |
| AUMCINF_pred | h*h*ng/mL | 1013098.1999 |
| AUMC_%Extrap_pred | % | 13.0051 |
| MRTlast | h | 51.9225 |
| MRTINF_obs | h | 57.8905 |
| MRTINF_pred | h | 57.6004 |
| AUC0_24 | h*ng/mL | 4121.7000 |
| | _ | |

WinNonlin 7.0.0.2535

PARAMCD=TEPO, SUBJID=PI ,APERIOD=1,TRTAN=2,TRTA=2 x 250 mg TF3

Date: PI Time: 09:23:22


# Settings

-----

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00

Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

```
00000000000000000
0 00 0 00 0 0 00 0 0 0 0 0
0 \  \, 
0 \  \, \varpi \  \, 0 \  \, \varpi \  \, 0 \  \,
```

AUC0\_24 h\*ng/mL 3882.1260

WinNonlin 7.0.0.2535 PARAMCD=TEPO,SUBJID=PI ,APERIOD=1,TRTAN=2,TRTA=2 x 250 mg TF3

> Date: PI 09:23:23 Time:


# Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

## Summary Table

| Time<br>h | Conc.<br>ng/mL | Pred.<br>ng/mL | Residual<br>ng/mL | AUC<br>h*ng/mL | AUMC<br>h*h*ng/mL | Weight |
|---|---|---|---|---|---|---|
| | | | | | • | |
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | | 0.0000 | |
| 0.5000 | 7.060 | | | 0.8825 | 0.4413 | |
| 0.7500 | 17.20 | | | 3.915 | 2.495 | |
| 1.000 | 25.50 | | | 9.253 | 7.295 | |
| 1.500 | 38.30 | | | 25.20 | 28.03 | |
| 2.000 | 39.40 | | | 44.63 | 62.10 | |
| 3.000 | 67.20 | | | 97.93 | 202.3 | |
| 4.000 | 109.0 | | | 186.0 | 521.1 | |
| 6.000 | 173.0 | | | 468.0 | 1995. | |
| 8.000 | 218.0 | | | 859.0 | 4777. | |
| 12.00 | 227.0 | | | 1749. 1.37 | le+004 | |
| 16.00 | 237.0 | | | 2677. 2.675 | 5e+004 | |
| 24.00 | 290.0 | | | 4785. 6.975 | 5e+004 | |
| 36.00 | 267.0 | | | 8125. 1.697 | 7e+005 | |
| 48.00 | 234.0 | | 1.11 | 13e+004 2.9 | 54e+005 | |
| 60.00 * | 195.0 | 199.7 | -4.686 1.36 | 59e+004 4.3 | 35e+005 | 1.000 |
| 72.00 * | 166.0 | 159.4 | 6.581 1.5 | 86e+004 5.7 | 58e+005 | 1.000 |
| 96.00 * | 100.0 | 101.6 | -1.608 1.89 | 98e+004 8.3 | 52e+005 | 1.000 |
| 120.0 * | 65.80 | 64.76 | 1.039 2.09 | 94e+004 1.0 | 45e+006 | 1.000 |
| 144.0 * | 39.70 | 41.28 | -1.576 2.21 | 18e+004 1.2 | 08e+006 | 1.000 |
| 168.0 * | 26.90 | 26.31 | 0.5922 2.2 | 97e+004 1.3 | 30e+006 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

## Final Parameters

| Rsq | | 0.9985 |
|--------------------|----------|----------|
| Rsq_adjusted | | 0.9981 |
| Corr_XY | | -0.9992 |
| No_points_lambda_z | | 6 |
| Lambda_z | 1/h | 0.0188 |
| Lambda_z_lower | h | 60.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 36.9336 |
| Tlag | h | 0.2500 |
| Tmax | h | 24.0000 |
| Cmax | ng/mL | 290.0000 |
| Cmax_D | ng/mL/mg | 0.6444 |

| Tlast | h | 168.0000 |
|-------------------|------------|--------------|
| Clast | ng/mL | 26.9000 |
| AUClast | h*ng/mL | 22970.4375 |
| AUCall | h*ng/mL | 22970.4375 |
| AUCINF_obs | h*ng/mL | 24403.7739 |
| AUCINF_D_obs | h*ng/mL/mg | 54.2306 |
| AUC_%Extrap_obs | % | 5.8734 |
| Vz_F_obs | L | 982.5426 |
| CI_F_obs | L/h | 18.4398 |
| AUCINF_pred | h*ng/mL | 24372.2207 |
| AUCINF_D_pred | h*ng/mL/mg | 54.1605 |
| AUC_%Extrap_pred | % | 5.7516 |
| Vz_F_pred | L | 983.8146 |
| Cl_F_pred | L/h | 18.4636 |
| AUMClast | h*h*ng/mL | 1330242.4556 |
| AUMCINF_obs | h*h*ng/mL | 1647416.7110 |
| AUMC_%Extrap_obs | % | 19.2528 |
| AUMCINF_pred | h*h*ng/mL | 1640434.4943 |
| AUMC_%Extrap_pred | % | 18.9091 |
| MRTlast | h | 57.9111 |
| MRTINF_obs | h | 67.5066 |
| MRTINF_pred | h | 67.3076 |
| AUC0_24 | h*ng/mL | 4785.0275 |

WinNonlin 7.0.0.2535

PARAMCD=TEPO,SUBJID=PI ,APERIOD=2,TRTAN=2,TRTA=2 x 250 mg TF3

PI 09:23:22 Date: Time:

## WINNONLIN NONCOMPARTMENTAL ANALYSIS PROGRAM 7.0.0.2535 Core Version 04Jun2007

# Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 450.00 Dose amount:

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values
Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

| Time | Conc. | Pred. | Residual | AUC | AUMC | Weight |
|--------|--------|-------|----------|--------------|-----------|--------|
| h | ng/mL | ng/mL | ng/mL | h*ng/mL | h*h*ng/mL | |
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2667 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.017 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.500 | 14.20 | | | 3.432 | 5.147 | |
| 2.000 | 38.30 | | | 16.56 | 29.62 | |
| 3.000 | 73.90 | | | 72.66 | 178.8 | |
| 4.000 | 129.0 | | | 174.1 | 547.6 | |
| 6.000 | 233.0 | | | 536.1 | 2462. | |
| 8.000 | 274.0 | | | 1043. | 6052. | |
| 12.00 | 297.0 | | | 2185, 1,756 | e+004 | |
| 16.00 | 290.0 | | | 3359. 3.399 | e+004 | |
| 24.00 | 299.0 | | | 5715, 8,125 | e+004 | |
| 36.00 | 268.0 | | | 9114, 1,828 | e+005 | |
| 48.00 | 223.0 | | 1.20 | 05e+004 3.05 | 7e+005 | |
| 60.00 | 170.0 | | 1.44 | 10e+004 4.31 | 6e+005 | |
| 72.73 | 125.0 | | | 26e+004 5.54 | | |
| 96.03 | 81.80 | | | 3e+004 7.53 | | |
| 30.00 | | | | | | |

| 120.0 * | 42.50 | 42.21 | 0.2920 2.007e+004 9.065e+005 | 1.000 |
|---------|-------|-------|-------------------------------|-------|
| 144.0 * | 24.40 | 24.74 | -0.3387 2.085e+004 1.009e+006 | 1.000 |
| 168.0 * | 14.60 | 14.50 | 0.1003 2.131e+004 1.080e+006 | 1.000 |

\*) Starred values were included in the estimation of Lambda\_z.

### Final Parameters

0.9995 Rsq Rsq\_adjusted 0.9990 Corr\_XY -0.9998 No\_points\_lambda\_z 3 Lambda\_z 1/h 0.0223 Lambda z lower h 120.0000 Lambda\_z\_upper 168.0000 h HL\_Lambda\_z h 31.1386 Tlag 1.0167 h 24.0000 Tmax h ng/mL Cmax 299.0000 Cmax\_D ng/mL/mg 0.6644 Tlast h 168.0000 14.6000 Clast ng/mL AUClast h\*ng/mL 21311.5822 AUCall h\*ng/mL 21311.5822 AUCINF\_obs 21967.4656 h\*ng/mL AUCINF\_D\_obs h\*ng/mL/mg 48.8166 AUC\_%Extrap\_obs Vz\_F\_obs CI\_F\_obs AUCINF\_pred 2.9857 L 920.2511 L/h 20.4848 h\*ng/mL 21962.9600 AUCINF\_D\_pred h\*ng/mL/mg 48.8066 AUC\_%Extrap\_pred % 2.9658 Vz\_F\_pred L 920.4399 CI\_F\_pred L/h 20.4890 **AUM**Clast h\*h\*ng/mL 1079987.9763 AUMCINF obs h\*h\*ng/mL 1219640.9871 AUMC\_%Extrap\_obs 11.4503 AUMCINF\_pred h\*h\*ng/mL 1218681.6380 AUMC\_%Extrap\_pred 11.3806 MRTlast 50.6761 MRTINF\_obs 55.5203 h MRTINF\_pred h 55.4880 5715.0510 AUC0\_24 h\*ng/mL

WinNonlin 7.0.0.2535

PARAMCD=TEPO,SUBJID=PI ,APERIOD=1,TRTAN=2,TRTA=2 x 250 mg TF3

Date: PI Time: 09:23:22


Settings

----

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

Summary Table

-----

| Time<br>h | Conc.<br>ng/mL | Pred.<br>ng/mL | Residual<br>ng/mL | AUC<br>h*ng/mL | AUMC<br>h*h*ng/ml | Weight |
|---|---|---|---|---|---|---|
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7333 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.500 | 11.00 | | | 2.750 | 4.125 | |
| 2.000 | 27.00 | | | 12.25 | 21.75 | |
| 3.000 | 75.70 | | | 63.60 | 162.3 | |
| 4.000 | 111.0 | | | 157.0 | 497.9 | |
| 6.000 | 153.0 | | | 421.0 | 1860. | |
| 8.050 | 176.0 | | | 758.2 | 4253. | |
| 12.00 | 211.0 | | | 1523. 1.205 | e+004 | |
| 16.05 | 211.0 | | | 2377. 2.404 | e+004 | |
| 24.02 | 218.0 | | | 4086. 5.838 | e+004 | |
| 36.00 | 194.0 | | | 6552. 1.321 | e+005 | |
| 48.00 * | 149.0 | 151.1 | -2.125 | 8598. 2.175 | 5e+005 | 1.000 |
| 60.00 * | 109.0 | 106.2 | 2.809 1.0 | 13e+004 2.99 | 99e+005 | 1.000 |
| 72.00 * | 75.20 | 74.62 | 0.5832 1.1 | 23e+004 3.7 | 16e+005 | 1.000 |
| 95.73 * | 37.20 | 37.13 | 0.06842 1.2 | 251e+004 4.7 | 73e+005 | 1.000 |
| 120.0 * | 17.10 | 18.19 | -1.090 1.3 | 13e+004 5.44 | l0e+005 | 1.000 |
| 144.0 * | 9.350 | 8.981 | 0.3687 1.3 | 344e+004 5.8 | 43e+005 | 1.000 |
| 168.0 | 0.0000 | | 1.3 | 56e+004 6.00 | )5e+005 | |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

| Rsq | | 0.9989 |
|--------------------|------------|-------------|
| Rsq_adjusted | | 0.9987 |
| Corr_XY | | -0.9995 |
| No_points_lambda_z | | 6 |
| Lambda_z | 1/h | 0.0294 |
| Lambda_z_lower | h | 48.0000 |
| Lambda_z_upper | h | 144.0000 |
| HL Lambda z | h | 23.5718 |
| Tlag | h | 1.0000 |
| Tmax | h | 24.0167 |
| Cmax | ng/mL | 218.0000 |
| Cmax_D | ng/mL/mg | 0.4844 |
| Tlast | h | 144.0000 |
| Clast | ng/mL | 9.3500 |
| AUClast | h*ng/mL | 13443.0163 |
| AUCall | h*ng/mL | 13555.2163 |
| AUCINF_obs | h*ng/mL | 13760.9804 |
| AUCINF_D_obs | h*ng/mL/mg | 30.5800 |
| AUC_%Extrap_obs | % | 2.3106 |
| Vz_F_obs | L | 1112.0636 |
| Cl_F_obs | L/h | 32.7012 |
| AUCINF_pred | h*ng/mL | 13748.4425 |
| AUCINF_D_pred | h*ng/mL/mg | 30.5521 |
| AUC_%Extrap_pred | % | 2.2215 |
| Vz_F_pred | L | 1113.0777 |
| Cl_F_pred | L/h | 32.7310 |
| AUMClast | h*h*ng/mL | 584346.9180 |
| AUMCINF_obs | h*h*ng/mL | 640946.7075 |
| AUMC_%Extrap_obs | % | 8.8307 |
| AUMCINF_pred | h*h*ng/mL | 638714.8799 |
| AUMC_%Extrap_pred | % | 8.5121 |
| MRTlast | h | 43.4684 |
| MRTINF_obs | h | 46.5771 |
| MRTINF_pred | h | 46.4573 |
| AUC0_24 | h*ng/mL | 4082.2668 |

WinNonlin 7.0.0.2535 PARAMCD=TEPO,SUBJID= $\mathbf{p_I}$  ,APERIOD=1,TRTAN=2,TRTA=2 x 250 mg TF3

```
00000000
0 \ 0 \ 0 \ 0 \ 0 \ 00 \ 00 \ 0 \ 00 \ 0
0000000000000000
0\ 00\ 0\ 000\ 0\ 00\ 0\ 0\ 0
00000000000000000
```

| Vz_F_obs | L | 1493.7034 |
|-------------------|------------|--------------|
| CI_F_obs | L/h | 27.4937 |
| AUCINF_pred | h*ng/mL | 16370.7366 |
| AUCINF_D_pred | h*ng/mL/mg | 36.3794 |
| AUC_%Extrap_pred | % | 5.2307 |
| Vz_F_pred | L | 1493.3982 |
| CI_F_pred | L/h | 27.4881 |
| AUMClast | h*h*ng/mL | 822206.6838 |
| AUMCINF_obs | h*h*ng/mL | 1011845.4005 |
| AUMC_%Extrap_obs | % | 18.7419 |
| AUMCINF_pred | h*h*ng/mL | 1012588.9412 |
| AUMC_%Extrap_pred | % | 18.8015 |
| MRTlast | h | 52.9963 |
| MRTINF_obs | h | 61.8208 |
| MRTINF_pred | h | 61.8536 |
| AUC0_24 | h*ng/mL | 4081.4941 |

WinNonlin 7.0.0.2535

PARAMCD=TEPO, SUBJID=pj ,APERIOD=2, TRTAN=1, TRTA=5 x 100 mg TF3

PI 09:23:22 Date: Time:

## WINNONLIN NONCOMPARTMENTAL ANALYSIS PROGRAM 7.0.0.2535 Core Version 04Jun2007

# Settings

Model: Plasma Data, Extravascular Administration Number of nonmissing observations: 22

Dose time: 450.00 Dose amount:

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values
Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

| Time<br>h | Conc.<br>ng/mL | Pred.<br>ng/mL | Residual<br>ng/mL | AUC<br>h*ng/mL | AUMC<br>h*h*ng/mL | Weight |
|---|---|---|---|---|---|---|
| 0.0000 | 0.0000 | | | 0.0000 | .0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | .0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | .0000 | |
| 0.7500 | 0.0000 | | | 0.0000 0 | .0000 | |
| 1.000 | 0.0000 | | | 0.0000 0 | .0000 | |
| 1.500 | 7.410 | | | 1.853 2 | 2.779 | |
| 2.000 | 10.80 | | | 6.405 | 0.96 | |
| 3.000 | 37.80 | | | 30.71 7 | 8.46 | |
| 4.000 | 68.10 | | | 83.66 2 | 71.4 | |
| 6.000 | 198.0 | | | 349.8 | 732. | |
| 8.067 | 221.0 | | | 782.7 | 1802. | |
| 12.00 | 202.0 | | | 1614. 1.312 | | |
| 16.00 | 190.0 | | | 2398. 2.407 | +004 | |
| 24.02 | 203.0 | | | 3973. 5.580 | e+004 | |
| 36.00 * | 172.0 | 175.3 | -3.261 | 6215. 1.227 | e+005 | 1.000 |
| 48.00 * | 146.0 | 137.0 | 9.014 | 81 19. 2.023 | 8e+005 | 1.000 |
| 60.00 * | 108.0 | 107.1 | 0.9303 | 9631. 2.836 | | 1.000 |
| 72.00 * | 81.60 | 83.69 | -2.087 1.0 | 76e+004 3.57 | 8e+005 | 1.000 |
| 96.07 * | 51.90 | 51.06 | 0.8442 1.2 | 34e+004 4.89 | 2e+005 | 1.000 |
| 120.0 * | 27.70 | 31.22 | -3.523 1.3 | 26e+004 5.87 | 7e+005 | 1.000 |
| 144.0 * | 19.80 | 19.08 | | 83e+004 6.61 | | 1.000 |
| 168.0 * | 12.10 | 11.65 | 0.4510 1.4 | 20e+004 7.20 | )1e+005 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

| Rsq | | 0.9966 |
|--------------------|------------|-------------|
| Rsq_adjusted | | 0.9961 |
| Corr_XÝ | | -0.9983 |
| No_points_lambda_z | | 8 |
| Lambda_z | 1/h | 0.0205 |
| Lambda_z_lower | h | 36.0000 |
| Lambda_z_upper | h | 168.0333 |
| HL_Lambda_z | h | 33.7575 |
| Tlag | h | 1.0000 |
| Tmax | h | 8.0667 |
| Cmax | ng/mL | 221.0000 |
| Cmax_D | ng/mL/mg | 0.4911 |
| Tlast | h | 168.0333 |
| Clast | ng/mL | 12.1000 |
| AUClast | h*ng/mL | 14204.1004 |
| AUCall | h*ng/mL | 14204.1004 |
| AUCINF_obs | h*ng/mL | 14793.3920 |
| AUCINF_D_obs | h*ng/mL/mg | 32.8742 |
| AUC_%Extrap_obs | % | 3.9835 |
| Vz_F_obs | L | 1481.4590 |
| CI F obs | L/h | 30.4190 |
| AUCINF_pred | h*ng/mL | 14771.4261 |
| AUCINF_D_pred | h*ng/mL/mg | 32.8254 |
| AUC_%Extrap_pred | % | 3.8407 |
| Vz_F_pred | L | 1483.6620 |
| CI F pred | L/h | 30.4642 |
| AUMClast | h*h*ng/mL | 720112.4562 |
| AUMCINF_obs | h*h*ng/mL | 847832.6414 |
| AUMC_%Extrap_obs | % | 15.0643 |
| AUMCINF_pred | h*h*ng/mL | 843071.8634 |
| AUMC_%Extrap_pred | % | 14.5847 |
| MRTlast | h | 50.6975 |
| MRTINF_obs | h | 57.3116 |
| MRTINF_pred | h | 57.0745 |
| AUC0_24 | h*ng/mL | 3969.7088 |
| | • | |

WinNonlin 7.0.0.2535

PARAMCD=TEPO,SUBJID=PI ,APERIOD=2,TRTAN=1,TRTA=5 x 100 mg TF3

> PI 09:23:23 Date: Time:


## Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 450.00 Dose amount:

Calculation method: Linear Trapezoidal Rule for for Increasing Values, Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

| Time | Conc. | Pred. | Residual | AUC | AUMC | Weight |
|---|---|---|---|---|---|---|
| h | ng/mL | ng/mL | ng/mL | h*ng/mL | h*h*ng/mL | |
| 0.0000<br>0.2500<br>0.5000<br>0.7500 | 0.0000<br>0.0000<br>0.0000<br>7.590 | | | 0.0000 | 0.0000<br>0.0000<br>0.0000<br>0.7116 | |

```
^{\circ}
0 \  \, 
0 \  \,
```

# WinNonlin Core Output - Tepotinib Metabolite MSC2571107A

WinNonlin 7.0.0.2535

PARAMCD=M7A,SUBJID=PI ,APERIOD=2,TRTAN=2,TRTA=2 x 250 mg TF3

Date: PI Time: 09:27:24


## Settings

\_\_\_\_

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

## Summary Table

| Time | Conc. | Pred. | Residual | AUC | AUMC | Weight |
|---------|--------|--------|----------|-------------|-----------|--------|
| h | ng/mL | ng/mL | ng/mL | h*ng/mL | h*h*ng/mL | |
| | | | | | • | |
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2667 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.017 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.500 | 0.2140 | | | 0.05172 0 | .07757 | |
| 2.000 | 0.4690 | | | 0.2225 | 0.3923 | |
| 3.000 | 1.240 | | | 1.077 | 2.721 | |
| 4.000 | 2.380 | | | 2.887 | 9.341 | |
| 6.000 | 2.850 | | | 8.117 | 35.96 | |
| 8.000 | 4.150 | | | 15.12 | 86.26 | |
| 12.00 | 4.780 | | | 32.98 | 267.4 | |
| 16.00 | 6.450 | | | 55.44 | 588.5 | |
| 24.00 | 7.650 | | | 111.8 | 1736. | |
| 36.00 | 5.910 | | | 192.7 | 4142. | |
| 48.00 | 6.360 | | | 266.4 | 7250. | |
| 60.00 | 4.160 | | | 328.6 1.058 | e+004 | |
| 72.73 | 3.870 | | | 379.7 1.397 | e+004 | |
| 96.03 | 3.130 | | | 460.9 2.079 | e+004 | |
| 120.0 * | 2.060 | 2.025 | 0.03491 | 522.2 2.73 | 36e+004 | 1.000 |
| 144.0 * | 1.050 | 1.087 | -0.03652 | 558.2 3.20 | 6e+004 | 1.000 |
| 168.0 * | 0.5930 | 0.5829 | 0.01005 | 577.4 3.5 | | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

# Final Parameters

| Rsq | | 0.9977 |
|--------------------|-------|----------|
| Rsq_adjusted | | 0.9955 |
| Corr_XY | | -0.9989 |
| No_points_lambda_z | | 3 |
| Lambda_z | 1/h | 0.0259 |
| Lambda z lower | h | 120.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 26.7180 |
| Tlag | h | 1.0167 |
| Tmax | h | 24.0000 |
| Cmax | ng/mL | 7.6500 |

Cmax\_D ng/mL/mg 0.0170 168.0000 Tlast h ng/mL Clast 0.5930 AUClast h\*ng/mL 577.3723 **AUCall** 577.3723 h\*ng/mL AUCINF\_obs h\*ng/mL 600.2301 AUCINF\_Dobs
AUC\_%Extrap\_obs
Vz\_F\_obs
CI\_F\_obs
AUCINF\_pred h\*ng/mL/mg 1.3338 % 3.8082 28898.3851 L L/h 749.7125 h\*ng/mL 599.8427 AUCINF\_D\_pred h\*ng/mL/mg 1.3330 AUC\_%Extrap\_pred 3.7460 % Vz\_F\_pred L 28917.0494 CI\_F\_pred L/h 750.1967 **AUMClast** h\*h\*ng/mL 35035.3710 39756.5470 AUMCINF\_obs h\*h\*ng/mL AUMC\_%Extrap\_obs 11.8752 AUMCINF\_pred AUMC\_%Extrap\_pred h\*h\*ng/mL 39676.5285 11.6975 60.6807 MRTlast MRTINF\_obs 66.2355 h MRTINF\_pred h 66.1449 AUC0\_24 111.8370 h\*ng/mL

WinNonlin 7.0.0.2535

PARAMCD=M7A,SUBJID=PI ,APERIOD=1,TRTAN=2,TRTA=2 x 250 mg TF3

Date: PI Time: 09:27:26


### Settings

-----

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

| Time | Conc. | Pred. | Residual | AUC | AUMC | Weight |
|--------|--------|-------|----------|-----------|-----------|--------|
| h | ng/mL | ng/mL | ng/mL | h*ng/m | L h*h*ng/ | mL |
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.000 | 0.1010 | | ( | 0.01263 | 0.01263 | |
| 1.500 | 0.1960 | | ( | 0.08688 | 0.1114 | |
| 2.000 | 0.3280 | | | 0.2179 | 0.3489 | |
| 3.000 | 0.7880 | | | 0.7759 | 1.859 | |
| 4.000 | 1.350 | | | 1.845 | 5.741 | |
| 6.000 | 2.130 | | | 5.325 | 23.92 | |
| 8.000 | 3.030 | | | 10.48 | 60.94 | |
| 12.00 | 3.960 | | | 24.46 | 204.5 | |
| 16.00 | 4.790 | | | 41.96 | 452.8 | |
| 24.00 | 9.560 | | | 99.36 | 1677. | |
| 36.00 | 8.510 | | | 207.7 | 4913. | |
| 48.00 | 11.20 | | | 325.9 | 9977. | |
| 60.00 | 10.10 | | | 453.6 1.6 | 86e+004 | |
| 72.00 | 12.20 | | | 587.4 2.5 | 77e+004 | |
| 72.00 | | | | | | |

| 96.00 * | 10.50 | 10.78 | -0.2835 | 859.3 4.852e+004 | 1.000 |
|---------|-------|-------|-----------|------------------|-------|
| 120.0 * | 7.720 | 7.328 | 0.3921 | 1076. 7.182e+004 | 1.000 |
| 144.0 * | 4.860 | 4.980 | -0.1197 | 1225. 9.126e+004 | 1.000 |
| 168.0 * | 3.380 | 3.384 | -0.003920 | 1322, 1,064e+005 | 1.000 |

\*) Starred values were included in the estimation of Lambda\_z.

## Final Parameters

| Rsq | | 0.9946 |
|--------------------|------------|-------------|
| Rsq_adjusted | | 0.9920 |
| Corr XY | | -0.9973 |
| No points lambda z | | 4 |
| Lambda z | 1/h | 0.0161 |
| Lambda_z_lower | h | 96.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL Lambda z | h | 43.0607 |
| Tlag | h | 0.7500 |
| Tmax | h | 72.0000 |
| Cmax | ng/mL | 12.2000 |
| Cmax D | ng/mL/mg | 0.0271 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 3.3800 |
| AUClast | h*ng/mL | 1322.3614 |
| AUCall | h*ng/mL | 1322.3614 |
| AUCINF_obs | h*ng/mL | 1532.3387 |
| AUCINF D obs | h*ng/mL/mg | 3.4052 |
| AUC_%Extrap_obs | % | 13.7031 |
| Vz_F_obs | L | 18243.7204 |
| Cl_F_obs | L/h | 293.6688 |
| AUCINF_pred | h*ng/mL | 1532.5822 |
| AUCINF_D_pred | h*ng/mL/mg | 3.4057 |
| AUC_%Extrap_pred | % | 13.7168 |
| Vz F pred | L | 18240.8217 |
| CI F pred | L/h | 293.6221 |
| AUMClast | h*h*ng/mL | 106446.9712 |
| AUMCINF_obs | h*h*ng/mL | 154767.6771 |
| AUMC %Extrap obs | % | 31.2214 |
| AUMCINF_pred | h*h*ng/mL | 154823.7155 |
| AUMC_%Extrap_pred | % | 31.2463 |
| MRTlast | h | 80.4976 |
| MRTINF_obs | h | 101.0010 |
| MRTINF pred | h | 101.0215 |
| AUC0_24 | h*ng/mL | 99.3649 |

WinNonlin 7.0.0.2535

PARAMCD=M7A,SUBJID=PI ,APERIOD=1,TRTAN=2,TRTA=2 x 250 mg TF3

PI 09:27:25 Date: Time:


## Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 450.00 Dose amount:

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values
Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

| Time | Conc.<br>ng/mL | Pred.<br>ng/mL | Residual<br>ng/mL | AUC<br>h*ng/mL | AUMC<br>h*h*ng/mL | Weight |
|---|---|---|---|---|---|---|
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.033 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 2.000 | 0.2340 | | | 0.05850 | 0.1170 | |
| 3.000 | 0.6310 | | | 0.4910 | 1.298 | |
| 4.000 | 1.170 | | | 1.392 | 4.584 | |
| 6.000 | 2.050 | | | 4.612 | 21.56 | |
| 8.000 | 2.730 | | | 9.392 | 55.70 | |
| 12.00 | 3.830 | | | 22.51 | 191.3 | |
| 16.00 | 4.180 | | | 38.53 | 417.0 | |
| 24.00 | 6.540 | | | 81.41 | 1312. | |
| 36.00 | 5.230 | | | 151.7 | 3406. | |
| 48.00 | 5.570 | | | 216.5 | 6140. | |
| 60.00 | 3.810 | | | 272.2 | 9122. | |
| 72.00 | 4.250 | | | 320.5 1.233 | 3e+004 | |
| 96.00 * | 3.040 | 2.942 | 0.09836 | 407.2 1.9 | 55e+004 | 1.000 |
| 120.0 * | 1.670 | 1.708 | -0.03760 | 462.1 2.54 | 41e+004 | 1.000 |
| 144.0 * | 0.9390 | 0.9912 | -0.05224 | 492.5 2.9 | 40e+004 | 1.000 |
| 168.0 * | 0.6010 | 0.5754 | 0.02559 | 510.7 3.2 | 22e+004 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

| Rsq | | 0.9957 |
|--------------------|------------|------------|
| Rsq_adjusted | | 0.9935 |
| Corr_XY | | -0.9978 |
| No_points_lambda_z | | 4 |
| Lambda_z | 1/h | 0.0227 |
| Lambda_z_lower | h | 96.0000 |
| Lambda_z_upper | h | 168,0000 |
| HL Lambda z | h | 30.5867 |
| Tlag | h | 1.5000 |
| Tmax | h | 24.0000 |
| Cmax | ng/mL | 6.5400 |
| Cmax D | ng/mL/mg | 0.0145 |
| Tlast | Ď h | 168.0000 |
| Clast | ng/mL | 0.6010 |
| AUClast | h*ng/mL | 510.7214 |
| AUCall | h*ng/mL | 510.7214 |
| AUCINF_obs | h*ng/mL | 537.2419 |
| AUCINF_D_obs | h*ng/mL/mg | 1.1939 |
| AUC_%Extrap_obs | % | 4.9364 |
| Vz_F_obs | L | 36961.4899 |
| Cl_F_obs | L/h | 837.6116 |
| AUCINF_pred | h*ng/mL | 536.1125 |
| AUCINF_D_pred | h*ng/mL/mg | 1.1914 |
| AUC_%Extrap_pred | % | 4.7362 |
| Vz_F_pred | L | 37039.3505 |
| Cl_F_pred | L/h | 839.3760 |
| AUMClast | h*h*ng/mL | 32221.9479 |
| AUMCINF_obs | h*h*ng/mL | 37847.6627 |
| AUMC_%Extrap_obs | % | 14.8641 |
| AUMCINF_pred | h*h*ng/mL | 37608.0990 |
| AUMC_%Extrap_pred | % | 14.3218 |
| MRTlast | h | 63.0910 |
| MRTINF_obs | h | 70.4481 |
| MRTINF_pred | h | 70.1496 |
| AUC0_24 | h*ng/mL | 81.4115 |

WinNonlin 7.0.0.2535

PARAMCD=M7A,SUBJID=PI ,APERIOD=1,TRTAN=2,TRTA=2 x 250 mg TF3

```
^{\circ} 0 ^{\circ}
                                                             000000000
0000000000000
                                       0000000000000000
П
П
 \  \  \, 0\  \  \, 0\ \  \, 0\  \  \, 0\
0 0 0 0 0 0 0 00000000 0 0 0 0 0
П
П
00000000000000000000000
Π
П
П
```

| AUC_%Extrap_obs | % | 6.0859 |
|-------------------|------------|------------|
| Vz_F_obs | L | 27115.4992 |
| Cl_F_obs | L/h | 591.9313 |
| AUCINF_pred | h*ng/mL | 760.0826 |
| AUCINF_D_pred | h*ng/mL/mg | 1.6891 |
| AUC_%Extrap_pred | % | 6.0685 |
| Vz_F_pred | L | 27120.5212 |
| Cl_F_pred | L/h | 592.0410 |
| AUMClast | h*h*ng/mL | 47483.5017 |
| AUMCINF_obs | h*h*ng/mL | 57375.6966 |
| AUMC_%Extrap_obs | % | 17.2411 |
| AUMCINF_pred | h*h*ng/mL | 57345.5984 |
| AUMC_%Extrap_pred | % | 17.1977 |
| MRTlast | h | 66.5075 |
| MRTINF_obs | h | 75.4722 |
| MRTINF_pred | h | 75.4465 |
| AUC0_24 | h*ng/mL | 86.3275 |

WinNonlin 7.0.0.2535

PARAMCD=M7A,SUBJID=PI ,APERIOD=2,TRTAN=1,TRTA=5 x 100 mg TF3

Date: P| Time: 09:27:27


## Settings

-----

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

| - | Time<br>h | Conc.<br>ng/mL | Pred.<br>ng/mL | Residual<br>ng/mL | AUC<br>h*ng/ml | AUMC<br>h*h*ng/m | Weight<br>L |
|---|---|---|---|---|---|---|---|
| | 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| | 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| | 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| | 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| | 1.000 | 0.0000 | | | 0.0000 | 0.0000 | |
| | 1.500 | 0.0000 | | | 0.0000 | 0.0000 | |
| | 2.000 | 0.2530 | | | 0.06325 | 0.1265 | |
| | 3.000 | 0.4760 | | | 0.4278 | 1.094 | |
| | 4.000 | 0.9520 | | | 1.142 | 3.712 | |
| | 6.000 | 1.690 | | | 3.784 | 17.66 | |
| | 8.000 | 2.800 | | | 8.274 | 50.20 | |
| | 12.00 | 4.360 | | | 22.59 | 199.6 | |
| | 16.00 | 6.300 | | | 43.91 | 505.9 | |
| | 24.00 | 7.890 | | | 100.7 | 1667. | |
| | 36.00 | 4.610 | | | 173.9 | 3825. | |
| | 48.00 | 5.970 | | | 237.4 | 6540. | |
| | 60.00 | 3.580 | | | 293.5 | 9540. | |
| | 72.00 * | 3.430 | 3.624 | -0.1935 | 335.5 1.23 | 31e+004 | 1.000 |
| | 96.00 * | 2.510 | 2.346 | 0.1636 | 406.2 1.8 | 21e+004 | 1.000 |
| | 120.0 * | 1.430 | 1.519 | -0.08936 | 452.3 2.3 | 13e+004 | 1.000 |
| | 144.0 * | 1.130 | 0.9838 | 0.1462 | 482.9 2.7 | 15e+004 | 1.000 |
| | 168.0 * | 0.5820 | 0.6371 | -0.05508 | 502.7 3.0 | | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

| Dee | | 0.9800 |
|---------------------|------------|------------|
| Rsq<br>Rsq_adjusted | | 0.9733 |
| | | -0.9899 |
| Corr_XY | | |
| No_points_lambda_z | 1/h | 5 |
| Lambda_z | | 0.0181 |
| Lambda_z_lower | h | 72.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | . h | 38.2800 |
| Tlag | h | 1.5000 |
| Tmax | h | 24.0000 |
| Cmax | ng/mL | 7.8900 |
| Cmax_D | ng/mL/mg | 0.0175 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 0.5820 |
| AUClast | h*ng/mL | 502.7147 |
| AUCall | h*ng/mL | 502.7147 |
| AUCINF_obs | h*ng/mL | 534.8564 |
| AUCINF_D_obs | h*ng/mL/mg | 1.1886 |
| AUC %Extrap obs | % | 6.0094 |
| Vz_F_obs | L | 46464.5032 |
| CI_F_obs | L/h | 841.3473 |
| AUCINF_pred | h*ng/mL | 537.8982 |
| AUCINF D pred | h*ng/mL/mg | 1.1953 |
| AUC %Extrap pred | % | 6.5409 |
| Vz_F_pred | L | 46201.7451 |
| Cl_F_pred | L/h | 836,5895 |
| AUMClast | h*h*ng/mL | 30221.0222 |
| AUMCINF_obs | h*h*ng/mL | 37395.8970 |
| AUMC %Extrap obs | % | 19,1863 |
| AUMCINF_pred | h*h*ng/mL | 38074.9136 |
| AUMC_%Extrap_pred | % | 20.6275 |
| MRTlast | h | 60.1157 |
| MRTINF_obs | " h | 69.9176 |
| MRTINF_pred | h<br>h | 70.7846 |
| AUC0_24 | h*ng/mL | 100.6738 |
| E4 | ng-mc | 100.0700 |

WinNonlin 7.0.0.2535

PARAMCD=M7A,SUBJID=PI ,APERIOD=2,TRTAN=1,TRTA=5 x 100 mg TF3

PI 09:27:25 Date: Time:


# Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 450.00 Dose amount:

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values
Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

# Summary Table

AUC AUMC Time Conc. Pred. Residual Weight h ng/mL ng/mL ng/mL h\*ng/mL h\*h\*ng/mL 0.0000 0.0000 0.0000 0.0000 0.2500 0.0000 0.0000 0.0000 0.5333 0.0000 0.0000 0.0000

| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
|---------|--------|--------|---------|-----------|------------|-------|
| 1.000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 2.000 | 0.2030 | | | 0.05075 | 0.1015 | |
| 3.000 | 0.5050 | | | 0.4048 | 1.062 | |
| 4.000 | 1.110 | | | 1.212 | 4.040 | |
| 6.000 | 1.630 | | | 3.952 | 18.26 | |
| 8.000 | 2.750 | | | 8.332 | 50.04 | |
| 12.00 | 4.120 | | | 22.07 | 192.9 | |
| 16.00 | 5.480 | | | 41.27 | 467.2 | |
| 24.02 | 8.200 | | | 96.11 | 1608. | |
| 36.00 | 6.740 | | | 185.3 | 4268. | |
| 48.00 | 7.440 | | | 270.4 | 7867. | |
| 60.02 | 4.510 | | | 340.8 1.1 | 163e+004 | |
| 72.00 * | 4.640 | 4.819 | -0.1787 | 395.6 1. | 525e+004 | 1.000 |
| 96.00 * | 3.090 | 3.021 | 0.06895 | | .287e+004 | 1.000 |
| 120.0 * | 2.100 | 1.894 | 0.2060 | | .946e+004 | 1.000 |
| 144.0 * | 1.050 | 1.187 | -0.1375 | | 421e+004 | 1.000 |
| 168.0 * | 0.7710 | 0.7445 | 0.02653 | 606.63 | 3.758e+004 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

| Rsq | | 0.9869 |
|--------------------|------------|------------|
| Rsq_adjusted | | 0.9825 |
| Corr XY | | -0.9934 |
| No_points_lambda_z | | 5 |
| Lambda_z | 1/h | 0.0195 |
| Lambda_z_lower | h | 72.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 35.6302 |
| Tlag | h | 1.5000 |
| Tmax | h | 24.0167 |
| Cmax | ng/mL | 8.2000 |
| Cmax_D | ng/mL/mg | 0.0182 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 0.7710 |
| AUClast | h*ng/mL | 606.6329 |
| AUCall | h*ng/mL | 606.6329 |
| AUCINF_obs | h*ng/mL | 646.2650 |
| AUCINF_D_obs | h*ng/mL/mg | 1.4361 |
| AUC_%Extrap_obs | % | 6.1325 |
| Vz_F_obs | L | 35792.7014 |
| Cl_F_obs | L/h | 696.3087 |
| AUCINF_pred | h*ng/mL | 644.9014 |
| AUCINF_D_pred | h*ng/mL/mg | 1.4331 |
| AUC_%Extrap_pred | % | 5.9340 |
| Vz_F_pred | L | 35868.3832 |
| Cl_F_pred | L/h | 697.7811 |
| AUMClast | h*h*ng/mL | 37580.0970 |
| AUMCINF_obs | h*h*ng/mL | 46275.5166 |
| AUMC_%Extrap_obs | % | 18.7905 |
| AUMCINF_pred | h*h*ng/mL | 45976.3356 |
| AUMC_%Extrap_pred | % | 18.2621 |
| MRTlast | h | 61.9487 |
| MRTINF_obs | h | 71.6045 |
| MRTINF_pred | h | 71.2920 |
| AUC0_24 | h*ng/mL | 95.9696 |

WinNonlin 7.0.0.2535

PARAMCD=M7A,SUBJID=PI ,APERIOD=2,TRTAN=1,TRTA=5 x 100 mg TF3

Date: PI Time: 09:27:26

WINNONLIN NONCOMPARTMENTAL ANALYSIS PROGRAM 7.0.0.2535

```
00000000 0
00000000
П
0000000000000000
00000000000000000
П
П
П
П
Π
П
```

CI\_F\_pred L/h 330.0405 **AUMClast** h\*h\*ng/mL 87479.5168 AUMCINF\_obs h\*h\*ng/mL 130072.5656 AUMC\_%Extrap\_obs 32.7456 AUMCINF\_pred AUMC\_%Extrap\_pred h\*h\*ng/mL 131143.1515 33.2946 MRTlast 74.2963 MRTINF\_obs 95.7185 h MRTINF\_pred h 96.1835 AUC0\_24 h\*ng/mL 132.7461

WinNonlin 7.0.0.2535

PARAMCD=M7A,SUBJID=PI ,APERIOD=1,TRTAN=1,TRTA=5 x 100 mg TF3

Date: PI Time: 09:27:24


## Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

## Summary Table

| Time | Conc. | Pred. | Residual | AUC | AUMC | Weight |
|---------|--------|--------|-----------|------------|----------|--------|
| h | ng/mL | ng/mL | ng/ml | _ h*ng/ml | h*h*ng/n | nL |
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.033 | 0.1370 | | | 0.01941 | 0.02006 | |
| 1.500 | 0.3340 | | | 0.1293 | 0.1700 | |
| 2.017 | 0.6180 | | | 0.3752 | 0.6214 | |
| 3.000 | 1.760 | | | 1.544 | 3.830 | |
| 4.000 | 2.430 | | | 3.639 | 11.33 | |
| 6.000 | 3.230 | | | 9.299 | 40.43 | |
| 8.000 | 3.700 | | | 16.23 | 89.41 | |
| 12.00 | 4.640 | | | 32.91 | 260.0 | |
| 16.00 | 5.720 | | | 53.63 | 554.4 | |
| 24.03 | 8.570 | | | 111.0 | 1749. | |
| 36.00 | 6.430 | | | 200.2 | 4399. | |
| 48.00 | 6.360 | | | 276.9 | 7622. | |
| 60.00 | 4.490 | | | 341.4 1.10 | 8e+004 | |
| 72.00 * | 4.330 | 4.450 | -0.1201 | 394.3 1.4 | 57e+004 | 1.000 |
| 96.00 * | 3.060 | 2.841 | 0.2195 | 482.1 2.1 | 88e+004 | 1.000 |
| 120.3 * | 1.680 | 1.804 | -0.1241 | 537.9 2.7 | 86e+004 | 1.000 |
| 144.0 * | 1.190 | 1.157 | 0.03269 | | 29e+004 | 1.000 |
| 168.0 * | 0.7360 | 0.7387 | -0.002710 | 594.3 3.5 | 581e+004 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

### Final Parameters

Rsq 0.9940 Rsq\_adjusted 0.9920 Corr\_XY -0.9970

| No_points_lambda_z | | 5 |
|--------------------|------------|------------|
| Lambda_z | 1/h | 0.0187 |
| Lambda_z_lower | h | 72.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 37.0548 |
| Tlag | h | 0.7500 |
| Tmax | h | 24.0333 |
| Cmax | ng/mL | 8.5700 |
| Cmax_D | ng/mL/mg | 0.0190 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 0.7360 |
| AUClast | h*ng/mL | 594.3188 |
| AUCall | h*ng/mL | 594.3188 |
| AUCINF_obs | h*ng/mL | 633.6645 |
| AUCINF_D_obs | h*ng/mL/mg | 1.4081 |
| AUC_%Extrap_obs | % | 6.2092 |
| Vz_F_obs | L | 37964.0342 |
| Cl_F_obs | L/h | 710.1550 |
| AUCINF_pred | h*ng/mL | 633.8094 |
| AUCINF_D_pred | h*ng/mL/mg | 1.4085 |
| AUC_%Extrap_pred | % | 6.2307 |
| Vz_F_pred | L | 37955.3550 |
| Cl_F_pred | L/h | 709.9927 |
| AUMClast | h*h*ng/mL | 35805.1167 |
| AUMCINF_obs | h*h*ng/mL | 44518.5627 |
| AUMC_%Extrap_obs | % | 19.5726 |
| AUMCINF_pred | h*h*ng/mL | 44550.6517 |
| AUMC_%Extrap_pred | % | 19.6305 |
| MRTlast | h | 60.2456 |
| MRTINF_obs | h | 70.2557 |
| MRTINF_pred | h | 70.2903 |
| AUC0_24 | h*ng/mL | 110.7421 |

WinNonlin 7.0.0.2535

PARAMCD=M7A,SUBJID=pj ,APERIOD=2,TRTAN=1,TRTA=5 x 100 mg TF3


## Settings

----

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

### Summary Table

Pred. AUC AUMC Weight Time Conc. Residual ng/mL ng/mL h\*ng/mL h\*h\*ng/mL h ng/mL 0.0000 0.0000 0.0000 0.0000 0.2500 0.0000 0.0000 0.0000 0.5000 0.0000 0.0000 0.0000 0.0000 0.7500 0.0000 0.0000 1.000 0.0000 0.0000 0.0000 1.500 0.0000 0.0000 0.0000 2.000 0.1420 0.03550 0.07100 0.3935 3.000 0.5740 1.074 4.000 0.9620 1.162 3.859 6.000 2.620 4.744 23.43

| 8.067 | 3.960 | | | 11.54 | 72.68 | |
|---------|--------|--------|-----------|----------|------------|-------|
| 12.00 | 4.660 | | | 28.50 | 245.5 | |
| 16.00 | 5.570 | | | 48.96 | 535.6 | |
| 24.02 | 8.080 | | | 103.7 | 1671. | |
| 36.00 * | 6.450 | 7.315 | -0.8655 | 190.4 | 4253. | 1.000 |
| 48.00 * | 7.090 | 5.952 | 1.138 | 271.6 | 7688. | 1.000 |
| 60.00 * | 4.450 | 4.842 | -0.3921 | 339.6 1. | 133e+004 | 1.000 |
| 72.00 * | 4.170 | 3.939 | 0.2306 | 391.3 1. | 474e+004 | 1.000 |
| 96.07 * | 2.890 | 2.604 | 0.2856 | 475.3 2. | 174e+004 | 1.000 |
| 120.0 * | 1.390 | 1.725 | -0.3353 | 524.4 2. | 697e+004 | 1.000 |
| 144.0 * | 1.250 | 1.142 | 0.1077 | 556.0 3. | 114e+004 | 1.000 |
| 168.0 * | 0.7560 | 0.7557 | 0.0003353 | 579.7 | 3.480e+004 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

| rinarraiameters | | |
|--------------------|------------|------------|
| Rsq | | 0.9744 |
| Rsq_adjusted | | 0.9701 |
| Corr_XY | | -0.9871 |
| No_points_lambda_z | | 8 |
| Lambda_z | 1/h | 0.0172 |
| Lambda_z_lower | h | 36.0000 |
| Lambda_z_upper | h | 168.0333 |
| HL_Lambda_z | h | 40.3139 |
| Tlag | h | 1.5000 |
| Tmax | h | 24.0167 |
| Cmax | ng/mL | 8.0800 |
| Cmax_D | ng/mL/mg | 0.0180 |
| Tlast | h | 168.0333 |
| Clast | ng/mL | 0.7560 |
| AUClast | h*ng/mL | 579.6538 |
| AUCall | h*ng/mL | 579.6538 |
| AUCINF obs | h*ng/mL | 623.6233 |
| AUCINF D obs | h*ng/mL/mg | 1.3858 |
| AUC %Extrap obs | % | 7.0506 |
| Vz_F_obs | L | 41968.1021 |
| CI_F_obs | L/h | 721.5895 |
| AUCINF pred | h*ng/mL | 623.6038 |
| AUCINF_D_pred | h*ng/mL/mg | 1.3858 |
| AUC_%Extrap_pred | % | 7.0477 |
| Vz_F_pred | L | 41969.4145 |
| Cl_F_pred | L/h | 721.6121 |
| AUMClast | h*h*ng/mL | 34796.5459 |
| AUMCINF_obs | h*h*ng/mL | 44742.1674 |
| AUMC_%Extrap_obs | % | 22.2287 |
| AUMCINF pred | h*h*ng/mL | 44737.7564 |
| AUMC %Extrap pred | % | 22.2211 |
| MRTlast | h | 60.0299 |
| MRTINF_obs | h | 71.7455 |
| MRTINF_pred | h | 71.7407 |
| AUCO 24 | h*ng/mL | 103.5346 |
| - | • | |

WinNonlin 7.0.0.2535

PARAMCD=M7A,SUBJID=pj ,APERIOD=2,TRTAN=1,TRTA=5 x 100 mg TF3

Date: Time: PI 09:27:26


# Settings

Model: Plasma Data, Extravascular Administration Number of nonmissing observations: 22

Dose time: 0.00

```
000000000000000
П
Π
П
.
П
```

MRTINF\_obs MRTINF\_pred AUC0\_24 h 57.6716 57.7456 h 99.1593 h\*ng/mL

WinNonlin 7.0.0.2535

PARAMCD=M7A, SUBJID=PI ,APERIOD=1,TRTAN=2,TRTA=2 x 250 mg TF3

> Date: PI 09:27:25 Time:


### Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 450.00 Dose amount:

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

### Summary Table

| Time | Conc.<br>ng/mL | Pred.<br>ng/mL | Residual<br>ng/ml | | AUMC<br>L h*h*ng/r | Weight |
|---|---|---|---|---|---|---|
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7333 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.000 | 0.1030 | | | 0.01373 | 0.01373 | |
| 1.500 | 0.2560 | | | 0.1035 | 0.1355 | |
| 2.000 | 0.5180 | | | 0.2970 | 0.4905 | |
| 3.000 | 1.390 | | | 1.251 | 3.093 | |
| 4.000 | 2.120 | | | 3.006 | 9.418 | |
| 6.000 | 2.510 | | | 7.636 | 32.96 | |
| 8.050 | 3.240 | | | 13.53 | 75.13 | |
| 12.00 | 3.820 | | | 27.47 | 217.2 | |
| 16.05 | 4.580 | | | 44.48 | 458.9 | |
| 24.02 | 6.260 | | | 87.66 | 1351. | |
| 36.00 | 4.660 | | | 152.6 | 3281. | |
| 48.00 * | 4.790 | 4.434 | 0.3562 | 209.3 | 5667. | 1.000 |
| 60.00 * | 2.660 | 3.282 | -0.6221 | 252.8 | 7988. | 1.000 |
| 72.00 * | 3.010 | 2.430 | 0.5805 | 286.8 1.0 | 25e+004 | 1.000 |
| 95.73 * | 1.360 | 1.340 | 0.01979 | 336.1 1.4 | 130e+004 | 1.000 |
| 120.0 * | 0.6590 | 0.7295 | -0.07048 | 359.6 1.6 | 680e+004 | 1.000 |
| 144.0 * | 0.3480 | 0.3997 | -0.05173 | 371.3 1.8 | 333e+004 | 1.000 |
| 168.0 * | 0.2530 | 0.2190 | 0.03397 | 378.4 1.9 | 944e+004 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

# Final Parameters

| Rsq | | 0.9810 |
|--------------------|-----|----------|
| Rsq_adjusted | | 0.9772 |
| Corr_XY | | -0.9905 |
| No_points_lambda_z | | 7 |
| Lambda_z | 1/h | 0.0251 |
| Lambda_z_lower | h | 48.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 27.6541 |
| Tlag | h | 0.7333 |
| Tmax | h | 24.0167 |

Cmax ng/mL 6.2600 Cmax D ng/mL/mg 0.0139 Tlast 168.0000 h ng/mL Clast 0.2530 **AUClast** h\*ng/mL 378.4066 AUCall h\*ng/mL 378.4066 AUCINF\_obs AUCINF\_D\_obs h\*ng/mL 388.5004 h\*ng/mL/mg 0.8633 AUC\_%Extrap\_obs Vz\_F\_obs Cl\_F\_obs 2.5981 46212.0324 1158.2999 L/h AUCINF\_pred AUCINF\_D\_pred h\*ng/mL 387,1453 h\*ng/mL/mg 0.8603 AUC\_%Extrap\_pred 2.2572 Vz\_F\_pred 46373.7922 L CI\_F\_pred AUMClast L/h 1162.3544 19440.8740 h\*h\*ng/mL AUMCINF\_obs h\*h\*ng/mL 21539.3383 AUMC\_%Extrap\_obs AUMCINF\_pred 9.7425 h\*h\*ng/mL 21257.6061 AUMC\_%Extrap\_pred 8.5463 MRTlast 51.3756 h MRTINF\_obs h 55.4423 MRTINF\_pred AUC0\_24 54.9086 h 87.5583 h\*ng/mL

WinNonlin 7.0.0.2535

PARAMCD=M7A,SUBJID=pj ,APERIOD=1,TRTAN=2,TRTA=2 x 250 mg TF3

Date: pj Time: 09:27:25


# Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

| Summary rable | | | | | | | |
|---|---|---|---|---|---|---|---|
| T | 0 | Dood | Desident | A110 | A1.0 | | 18/-: |
| Time | Conc. | Pred. | Residual | AUC | AUI | | Weight |
| h | ng/mL | ng/mL | ng/mL | h*ng/n | nL h"h" | 'ng/mL | |
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | | |
| 1.000 | 0.1250 | | | 0.01563 | 0.01563 | | |
| 1.600 | 0.2270 | | | 0.1212 | 0.1621 | | |
| 2.217 | 0.4870 | | | 0.3414 | 0.6069 | | |
| 3.000 | 1.370 | | | 1.069 | 2.639 | | |
| 4.000 | 2.050 | | | 2.779 | 8.794 | | |
| 6.000 | 2.970 | | | 7.799 | 34.81 | | |
| 8.000 | 3.980 | | | 14.75 | 84.47 | | |
| 12.00 | 4.200 | | | 31.11 | 249.0 | | |
| 16.00 | 5.090 | | | 49.69 | 512.6 | | |
| 24.02 | 7.640 | | | 100.7 | 1575. | | |
| 36.00 | 5.950 | | | 181.7 | 3985. | | |
| 48.02 | 6.530 | | | 256.7 | 7156. | | |
| 60.00 | 4.320 | | | 320.8 1.0 | 159e+004 | | |
| 72.00 * | 4.640 | 4.654 | -0.01418 | 374.6 1.415e+004 | 1.000 |
|---------|-------|-------|----------|------------------|-------|
| 96.02 * | 3.330 | 3.176 | 0.1541 | 469.4 2.206e+004 | 1.000 |
| 120.0 * | 2.010 | 2.168 | -0.1582 | 532.1 2.877e+004 | 1.000 |
| 144.1 * | 1.510 | 1.478 | 0.03242 | 574.2 3.430e+004 | 1.000 |
| 168.0 * | 1.020 | 1.010 | 0.009878 | 604.1 3.894e+004 | 1.000 |

### Final Parameters

| Rsq | | 0.9942 |
|--------------------|------------|------------|
| Rsq_adjusted | | 0.9922 |
| Corr XY | | -0.9971 |
| No_points_lambda_z | | 5 |
| Lambda z | 1/h | 0.0159 |
| Lambda_z_lower | h | 72.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 43.5572 |
| Tlag | h | 0.7500 |
| Tmax | h | 24.0167 |
| Cmax | ng/mL | 7.6400 |
| Cmax_D | ng/mL/mg | 0.0170 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 1.0200 |
| AUClast | h*ng/mL | 604.0927 |
| AUCall | h*ng/mL | 604.0927 |
| AUCINF_obs | h*ng/mL | 668.1893 |
| AUCINF_D_obs | h*ng/mL/mg | 1.4849 |
| AUC_%Extrap_obs | % | 9.5926 |
| Vz_F_obs | L | 42320.1954 |
| Cl_F_obs | L/h | 673.4618 |
| AUCINF_pred | h*ng/mL | 667.5686 |
| AUCINF_D_pred | h*ng/mL/mg | 1.4835 |
| AUC_%Extrap_pred | % | 9.5085 |
| Vz_F_pred | L | 42359.5480 |
| Cl_F_pred | L/h | 674.0881 |
| AUMClast | h*h*ng/mL | 38939.8758 |
| AUMCINF_obs | h*h*ng/mL | 53735.9159 |
| AUMC_%Extrap_obs | % | 27.5347 |
| AUMCINF_pred | h*h*ng/mL | 53592.6206 |
| AUMC_%Extrap_pred | % | 27.3410 |
| MRTlast | h | 64.4601 |
| MRTINF_obs | h | 80.4202 |
| MRTINF_pred | h | 80.2803 |
| AUC0_24 | h*ng/mL | 100.5875 |

WinNonlin 7.0.0.2535

PARAMCD=M7A,SUBJID=PI ,APERIOD=2,TRTAN=1,TRTA=5 x 100 mg TF3

Date: PI 09:27:24 Time:


## Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 450.00 Dose amount:

Calculation method: Linear Trapezoidal Rule for for Increasing Values, Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

```
ПППП
00000000000000000
П
П
Π
Π
תחתום חום חום התחתות התחתות המוחום הווחום הווחום הווחום התחתות החתות
    0000000000000000000
Π
П
П
0 0 0 000000000
П
П
П
Π
```

Date: PI 09:27:26 Time:


### Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 450.00 Dose amount:

Calculation method: Linear Trapezoidal Rule for for Increasing Values, Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

### Summary Table

| Time | Conc.<br>ng/mL | Pred.<br>ng/mL | Residual<br>ng/ml | | AUMC | |
|---|---|---|---|---|---|---|
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.500 | 0.2120 | | | 0.05300 | 0.07950 | |
| 2.000 | 0.3270 | | | 0.1878 | 0.3225 | |
| 3.000 | 0.6210 | | | 0.6618 | 1.581 | |
| 4.000 | 0.9700 | | | 1.457 | 4.453 | |
| 6.000 | 1.590 | | | 4.017 | 17.87 | |
| 8.000 | 1.960 | | | 7.567 | 43.09 | |
| 12.00 | 2.990 | | | 17.47 | 146.2 | |
| 16.00 | 3.520 | | | 30.49 | 330.6 | |
| 24.00 | 5.850 | | | 67.97 | 1117. | |
| 36.00 | 6.530 | | | 142.2 | 3370. | |
| 48.00 * | 6.200 | 5.763 | 0.4373 | 218.6 | 6574. | 1.000 |
| 60.03 * | 3.890 | 4.333 | -0.4435 | 278.2 | 9767. | 1.000 |
| 72.00 * | 3.440 | 3.264 | 0.1762 | 322.0 1. | 265e+004 | 1.000 |
| 96.00 * | 1.660 | 1.849 | -0.1885 | 380.7 1.7 | 749e+004 | 1.000 |
| 120.0 * | 1.190 | 1.047 | 0.1431 | 414.6 2. | 113e+004 | 1.000 |
| 144.0 * | 0.5790 | 0.5929 | -0.01395 | 434.92 | .379e+004 | 1.000 |
| 168.0 * | 0.3310 | 0.3358 | -0.004825 | 445.62 | .544e+004 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

### Final Parameters

| Rsq | | 0.9929 |
|--------------------|----------|----------|
| Rsq_adjusted | | 0.9915 |
| Corr_XY | | -0.9964 |
| No_points_lambda_z | | 7 |
| Lambda_z | 1/h | 0.0237 |
| Lambda_z_lower | h | 48.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 29.2614 |
| Tlag | h | 1.0000 |
| Tmax | h | 36.0000 |
| Cmax | ng/mL | 6.5300 |
| Cmax_D | ng/mL/mg | 0.0145 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 0.3310 |
| AUClast | h*ng/mL | 445.5607 |
| AUCall | h*ng/mL | 445.5607 |
| AUCINF_obs | h*ng/mL | 459.5339 |

AUCINF\_D\_obs 1.0212 h\*ng/mL/mg AUC\_%Extrap\_obs Vz\_F\_obs 3.0407 41339.3706 979.2530 CI\_F\_obs L/h AUCINF\_pred AUCINF\_D\_pred h\*ng/mL 459.7376 1.0216 h\*ng/mL/mg AUC\_%Extrap\_pred 3.0837 Vz\_F\_pred 41321.0542 L CI\_F\_pred AUMClast L/h 978.8191 h\*h\*ng/mL 25437.2620 AUMCINF\_obs h\*h\*ng/mL 28374.6483 AUMC %Extrap\_obs 10.3522 AUMCINF\_pred h\*h\*ng/mL 28417.4685 AUMC\_%Extrap\_pred 10.4872 MRTlast 57.0905 h MRTINF obs h 61.7466 MRTINF\_pred 61.8124 h AUC0\_24 h\*ng/mL 67.9673

WinNonlin 7.0.0.2535

PARAMCD=M7A,SUBJID=pj ,APERIOD=1,TRTAN=1,TRTA=5 x 100 mg TF3

Date: pj Time: 09:27:25


## Settings

-----

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

## Summary Table

AUC AUMC Weight Time Conc. Pred. Residual h\*ng/mL h\*h\*ng/mL h ng/mL ng/mL ng/mL 0.0000 0.0000 0.0000 0.0000 0.2500 0.0000 0.0000 0.0000 0.5000 0.0000 0.0000 0.0000 0.7500 0.0000 0.0000 0.0000 1.000 0.0000 0.0000 0.0000 0.1450 0.5800 1.500 0.2175 2.000 1.280 0.6100 1.075 3.000 3.020 6.885 2.760 4.000 4.860 6.700 21.14 5.460 17.02 73.34 6.000 8.000 6.340 28.82 156.8 12.00 6.020 53.53 403.5 16.00 7.440 80.45 786.1 24.02 8.680 145.1 2099. 7.300 36.00 240.6 4948. 48.00 4.870 312.6 7945. 60.00 3.910 365.1 1.077e+004 72.02 4.110 413.3 1.395e+004 96.00 3.730 507.2 2.183e+004 120.3 \* 1.000 3.900 3.740 0.1599 599.9 3.187e+004 144.0 \* 2.292 -0.1825 668.9 4.091e+004 1.000 2.110 168.1 \* 1.392 0.05834 1.450 711.4 4.750e+004 1.000

## Final Parameters

| Rsq | | 0.9793 |
|--------------------|------------|------------|
| Rsq_adjusted | | 0.9586 |
| Corr_XY | | -0.9896 |
| No_points_lambda_z | | 3 |
| Lambda_z | 1/h | 0.0207 |
| Lambda_z_lower | h | 120.2833 |
| Lambda_z_upper | h | 168.1167 |
| HL_Lambda_z | h | 33.5377 |
| Tlag | h | 1.0000 |
| Tmax | h | 24.0167 |
| Cmax | ng/mL | 8.6800 |
| Cmax_D | ng/mL/mg | 0.0193 |
| Tlast | h | 168.1167 |
| Clast | ng/mL | 1.4500 |
| AUClast | h*ng/mL | 711.3561 |
| AUCall | h*ng/mL | 711.3561 |
| AUCINF_obs | h*ng/mL | 781.5139 |
| AUCINF_D_obs | h*ng/mL/mg | 1.7367 |
| AUC_%Extrap_obs | % | 8.9772 |
| Vz_F_obs | L | 27860.1940 |
| Cl_F_obs | L/h | 575.8055 |
| AUCINF_pred | h*ng/mL | 778.6913 |
| AUCINF_D_pred | h*ng/mL/mg | 1.7304 |
| AUC_%Extrap_pred | % | 8.6472 |
| Vz_F_pred | L | 27961.1811 |
| CI_F_pred | L/h | 577.8926 |
| AUMClast | h*h*ng/mL | 47504.9820 |
| AUMCINF_obs | h*h*ng/mL | 62694.2573 |
| AUMC_%Extrap_obs | % | 24.2275 |
| AUMCINF_pred | h*h*ng/mL | 62083.1634 |
| AUMC_%Extrap_pred | % | 23.4817 |
| MRTlast | h | 66.7809 |
| MRTINF_obs | h | 80.2215 |
| MRTINF_pred | h | 79.7276 |
| AUC0_24 | h*ng/mL | 144.9242 |

WinNonlin 7.0.0.2535

PARAMCD=M7A,SUBJID=PI ,APERIOD=1,TRTAN=1,TRTA=5 x 100 mg TF3

Date: PI 09:27:26 Time:


### Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 450.00 Dose amount:

Calculation method: Linear Trapezoidal Rule for for Increasing Values, Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

| Time | Conc. | Pred. | Residual | AUC | AUMC | Weight |
|---|---|---|---|---|---|---|
| h | ng/mL | ng/mL | ng/mL | h*ng/mL | h*h*ng/mL | |
| 0.0000<br>0.2500 | 0.0000<br>0.0000 | | | | .0000 | |

| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
|---------|--------|-------|---------|----------|-----------|-------|
| 0.7833 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 2.000 | 0.1960 | | | 0.04900 | 0.09800 | |
| 3.000 | 0.7990 | | | 0.5465 | 1.493 | |
| 4.000 | 1.930 | | | 1.911 | 6.551 | |
| 6.000 | 3.630 | | | 7.471 | 36.05 | |
| 8.000 | 4.620 | | | 15.72 | 94.79 | |
| 12.00 | 5.790 | | | 36.54 | 307.7 | |
| 16.00 | 6.000 | | | 60.12 | 638.6 | |
| 24.00 | 8.500 | | | 118.1 | 1839. | |
| 36.00 | 5.930 | | | 203.8 | 4378. | |
| 48.00 | 6.750 | | | 279.9 | 7602. | |
| 60.00 | 5.750 | | | 354.7 1. | 163e+004 | |
| 72.00 * | 6.700 | 6.909 | -0.2088 | 429.4 1 | .660e+004 | 1.000 |
| 96.00 * | 4.920 | 4.753 | 0.1673 | 567.7 2 | .813e+004 | 1.000 |
| 120.0 * | 3.070 | 3.270 | -0.1996 | 661.93 | .821e+004 | 1.000 |
| 144.0 * | 2.600 | 2.249 | 0.3508 | 729.8 4 | .715e+004 | 1.000 |
| 168.0 * | 1.420 | 1.547 | -0.1273 | 776.6 5 | .440e+004 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

| Tillatt diditiolois | | |
|---------------------|------------|------------|
| Rsq | | 0.9760 |
| Rsq_adjusted | | 0.9679 |
| Corr XY | | -0.9879 |
| No points lambda z | | 5 |
| Lambda_z | 1/h | 0.0156 |
| Lambda z lower | ''h | 72.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL Lambda z | h | 44.4717 |
| Tlag | h | 1.5000 |
| Tmax | "h | 24.0000 |
| Cmax | ng/mL | 8.5000 |
| Cmax_D | ng/mL/mg | 0.0189 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 1,4200 |
| AUClast | h*ng/mL | 776.5863 |
| AUCall | h*ng/mL | 776.5863 |
| AUCINF_obs | h*ng/mL | 867.6923 |
| AUCINF D obs | h*ng/mL/mg | 1.9282 |
| AUC_%Extrap_obs | % | 10.4998 |
| Vz_F_obs | L | 33274.0250 |
| CI_F_obs | L/h | 518.6170 |
| AUCINF_pred | h*ng/mL | 875.8598 |
| AUCINF_D_pred | h*ng/mL/mg | 1.9464 |
| AUC_%Extrap_pred | % | 11.3344 |
| Vz_F_pred | L | 32963.7376 |
| CI_F_pred | L/h | 513.7808 |
| AUMClast | h*h*ng/mL | 54396.3729 |
| AUMCINF_obs | h*h*ng/mL | 75547.4595 |
| AUMC_%Extrap_obs | % | 27.9971 |
| AUMCINF_pred | h*h*ng/mL | 77443.6381 |
| AUMC_%Extrap_pred | % | 29.7600 |
| MRTlast | h. | 70.0455 |
| MRTINF_obs | h | 87.0671 |
| MRTINF_pred | h | 88.4201 |
| AUC0_24 | h*ng/mL | 118.1210 |

WinNonlin 7.0.0.2535

PARAMCD=M7A,SUBJID=PI ,APERIOD=2,TRTAN=2,TRTA=2 x 250 mg TF3

Date: **PI** Time: 09:27:27

```
00000000
П
П
                0000000000000000
00000000000000000
П
 \  \, 0 \ \, 0 \  \, 0 \ \, 0 \  \, 0 \ \, 0 \  \, 0 \  \, 0 \ \, 0 \  \, 0 \ \,
П
П
П
П
П
0000000
```

Vz\_F\_pred Cl\_F\_pred AUMClast L 39739.4753 L/h 376.8262 h\*h\*ng/mL 67713.0139 133753.1096 AUMCINF\_obs h\*h\*ng/mL AUMC\_%Extrap\_obs AUMCINF\_pred 49.3746 h\*h\*ng/mL 133942.2754 AUMC\_%Extrap\_pred 49.4461 MRTlast h 71.1276 MRTINF\_obs h 112.0687 MRTINF\_pred 112.1621 h AUC0\_24 128.1248 h\*ng/mL

WinNonlin 7.0.0.2535

PARAMCD=M7A,SUBJID=pj ,APERIOD=2,TRTAN=2,TRTA=2 x 250 mg TF3

Date: pj Time: 09:27:26


## Settings

-----

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting

Lambda\_z method: Find best fit for lambda\_z, Log regression

## Summary Table

| Time | Conc. | Pred. | Residual | AUC | AUMC | Weight |
|---------|--------|--------|-----------|-----------|------------|--------|
| h | ng/mL | ng/mL | | | | |
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.500 | 0.2060 | | | 0.05150 | 0.07725 | |
| 2.000 | 0.4930 | | | 0.2263 | 0.4010 | |
| 3.000 | 1.030 | | | 0.9878 | 2.439 | |
| 4.000 | 1.810 | | | 2.408 | 7.604 | |
| 6.000 | 2.680 | | | 6.898 | 30.92 | |
| 8.000 | 3.650 | | | 13.23 | 76.20 | |
| 12.00 | 5.840 | | | 32.21 | 274.8 | |
| 16.00 | 7.130 | | | 58.15 | 643.1 | |
| 24.00 | 10.20 | | | 127.5 | 2079. | |
| 36.03 | 9.030 | | | 243.0 | 5533. | |
| 48.00 | 8.760 | | | 349.5 1.0 | 000e+004 | |
| 60.00 | 5.560 | | | 433.9 1.4 | 53e+004 | |
| 72.00 | 4.820 | | | 496.1 1.8 | 62e+004 | |
| 96.00 | 3.130 | | | 590.1 2.6 | 43e+004 | |
| 120.0 * | 1.390 | 1.399 | -0.008729 | 641.53 | .190e+004 | 1.000 |
| 144.0 * | 0.9030 | 0.8918 | 0.01124 | 668.63 | 3.546e+004 | 1.000 |
| 168.0 * | 0.5650 | 0.5685 | -0.003548 | 685.9 3 | 3.814e+004 | 1.000 |
| | | | | 300.00 | | |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

#### Final Parameters

-----

Rsq 0.9994 Rsq\_adjusted 0.9988

| Corr_XY | | -0.9997 |
|--------------------|------------|------------|
| No_points_lambda_z | | 3 |
| Lambda z | 1/h | 0.0188 |
| Lambda_z_lower | h | 120.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 36.9583 |
| Tlag | h | 1.0000 |
| Tmax | h | 24.0000 |
| Cmax | ng/mL | 10.2000 |
| Cmax_D | ng/mL/mg | 0.0227 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 0.5650 |
| AUClast | h*ng/mL | 685.8936 |
| AUCall | h*ng/mL | 685.8936 |
| AUCINF_obs | h*ng/mL | 716.0191 |
| AUCINF_D_obs | h*ng/mL/mg | 1.5912 |
| AUC_%Extrap_obs | % | 4.2074 |
| Vz_F_obs | L | 33509.9715 |
| Cl_F_obs | L/h | 628.4748 |
| AUCINF_pred | h*ng/mL | 716.2083 |
| AUCINF_D_pred | h*ng/mL/mg | 1.5916 |
| AUC_%Extrap_pred | % | 4.2327 |
| Vz_F_pred | L | 33501.1202 |
| Cl_F_pred | L/h | 628.3088 |
| AUMClast | h*h*ng/mL | 38139.9732 |
| AUMCINF_obs | h*h*ng/mL | 44807.3395 |
| AUMC_%Extrap_obs | % | 14.8801 |
| AUMCINF_pred | h*h*ng/mL | 44849.2085 |
| AUMC_%Extrap_pred | % | 14.9595 |
| MRTlast | h | 55.6063 |
| MRTINF_obs | h | 62.5784 |
| MRTINF_pred | h | 62.6203 |
| AUC0_24 | h*ng/mL | 127.4678 |

WinNonlin 7.0.0.2535

PARAMCD=M7A,SUBJID=PI ,APERIOD=2,TRTAN=2,TRTA=2 x 250 mg TF3

Date: PI 09:27:25 Time:


## Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 450.00 Dose amount:

Calculation method: Linear Trapezoidal Rule for for Increasing Values, Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

| Time<br>h | Conc.<br>ng/mL | Pred.<br>ng/mL | Residual<br>ng/mL | AUC<br>h*ng/n | AUM<br>nL h*h*n | C Weight<br>g/mL |
|---|---|---|---|---|---|---|
| 0.0000 | 0.0000 | | ( | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | ( | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | ( | 0.0000 | 0.0000 | |
| 0.7500 | 0.1400 | | 0. | 01750 | 0.01313 | |
| 1.000 | 0.2360 | | 0. | 06450 | 0.05575 | |
| 1.500 | 0.6430 | | 0 | .2843 | 0.3559 | |
| 2.000 | 1.030 | | 0 | .7025 | 1.112 | |
| 3.000 | 1.830 | | | 2.133 | 4.887 | |
| 4.000 | 2.730 | | | 4.413 | 13.09 | |

| 6.000 | 3.290 | | | 10.43 | 43.75 | |
|---------|-------|-------|---------|-----------|------------|-------|
| 8.000 | 4.070 | | | 17.79 | 96.05 | |
| 12.00 | 5.010 | | | 35.95 | 281.4 | |
| 16.00 | 6.230 | | | 58.43 | 601.0 | |
| 24.00 | 8.700 | | | 118.2 | 1835. | |
| 36.00 | 7.870 | | | 217.5 | 4805. | |
| 48.00 | 9.130 | | | 319.5 | 9134. | |
| 60.00 | 7.900 | | | 421.5 1.4 | 163e+004 | |
| 72.02 | 7.720 | | | 515.3 2.0 | 082e+004 | |
| 96.00 | 5.010 | | | 665.7 3.3 | 332e+004 | |
| 120.0 * | 5.270 | 5.068 | 0.2022 | 789.04 | .668e+004 | 1.000 |
| 144.1 * | 2.680 | 2.899 | -0.2188 | 881.2 5. | 873e+004 | 1.000 |
| 168.0 * | 1.730 | 1.663 | 0.06675 | 933.1 6 | 6.679e+004 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

| · marr alameters | | |
|--------------------|------------|------------|
| Rsq | | 0.9853 |
| Rsq_adjusted | | 0.9707 |
| Corr_XY | | -0.9926 |
| No_points_lambda_z | | 3 |
| Lambda_z | 1/h | 0.0232 |
| Lambda_z_lower | h | 120.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 29.8629 |
| Tlag | h | 0.5000 |
| Tmax | h | 48.0000 |
| Cmax | ng/mL | 9.1300 |
| Cmax_D | ng/mL/mg | 0.0203 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 1.7300 |
| AUClast | h*ng/mL | 933.1420 |
| AUCall | h*ng/mL | 933.1420 |
| AUCINF_obs | h*ng/mL | 1007.6757 |
| AUCINF_D_obs | h*ng/mL/mg | 2.2393 |
| AUC_%Extrap_obs | % | 7.3966 |
| Vz_F_obs | L | 19239.7000 |
| CI_F_obs | L/h | 446.5723 |
| AUCINF_pred | h*ng/mL | 1004.8000 |
| AUCINF_D_pred | h*ng/mL/mg | 2.2329 |
| AUC_%Extrap_pred | % | 7.1316 |
| Vz_F_pred | L | 19294.7628 |
| Cl_F_pred | L/h | 447.8503 |
| AUMClast | h*h*ng/mL | 66785.9287 |
| AUMCINF_obs | h*h*ng/mL | 82518.7298 |
| AUMC_%Extrap_obs | % | 19.0657 |
| AUMCINF_pred | h*h*ng/mL | 81911.7235 |
| AUMC_%Extrap_pred | % | 18.4660 |
| MRTlast | h | 71.5710 |
| MRTINF_obs | h | 81.8902 |
| MRTINF pred | h | 81.5204 |
| AUC0_24 | h*ng/mL | 118.1525 |
| _ | - | |

WinNonlin 7.0.0.2535 PARAMCD=M7A,SUBJID= $p_1$ ,APERIOD=1,TRTAN=2,TRTA=2 x 250 mg TF3

Date: Time:


### Settings

Model: Plasma Data, Extravascular Administration Number of nonmissing observations: 22

```
0 0 0 0 0 0 0 000000 0
0000000000
00000000000000000
Π
0 0 0 0 0 00000000 0 0 0 0 0000000
П
0 0 0 0 0 0 0 0 0 0 0 0 0 0 000000000
00000000 \\
   П
00000000
0\,0\,0\,0\,0\,0\,0\,0\,0\,0\,0\,0\,0000000
```

MRTlast h 63.5371 MRTINF\_obs h 71.4680 MRTINF\_pred AUC0\_24 71.8122 h h\*ng/mL 95.9402

WinNonlin 7.0.0.2535

PARAMCD=M7A,SUBJID=pj ,APERIOD=2,TRTAN=2,TRTA=2 x 250 mg TF3

Date: PI 09:27:27 Time:


## Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values
Weighting for lambda\_z calculations: Uniform weighting

Lambda\_z method: Find best fit for lambda\_z, Log regression

## Summary Table

| Time | Conc. | Pred. | Residual | AUC | AUMC | Weight |
|---------|--------|--------|----------|----------|----------|--------|
| h | ng/mL | ng/mL | ng/mL | h*ng/m | | |
| | | | | | • | |
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 2.000 | 0.1130 | | | 0.02825 | 0.05650 | |
| 3.000 | 0.2980 | | | 0.2338 | 0.6165 | |
| 4.000 | 0.6840 | | | 0.7248 | 2.432 | |
| 6.000 | 1.910 | | | 3.319 | 16.63 | |
| 8.000 | 2.730 | | | 7.959 | 49.93 | |
| 12.03 | 4.330 | | | 22.20 | 199.0 | |
| 16.00 | 5.310 | | | 41.32 | 470.9 | |
| 24.00 | 7.840 | | | 93.92 | 1563. | |
| 36.00 | 5.480 | | | 173.0 | 3907. | |
| 48.00 * | 5.960 | 5.814 | 0.1456 | 241.6 | 6808. | 1.000 |
| 60.00 * | 3.910 | 4.436 | -0.5265 | 300.0 | 9934. | 1.000 |
| 72.00 * | 3.750 | 3.385 | 0.3649 | | 297e+004 | 1.000 |
| 96.07 * | 2.060 | 1.968 | 0.09214 | | 359e+004 | 1.000 |
| 120.1 * | 1.160 | 1.146 | 0.01389 | | 261e+004 | 1.000 |
| 144.0 * | 0.5890 | 0.6680 | -0.07902 | | 525e+004 | 1.000 |
| 168.0 * | 0.4160 | 0.3889 | 0.02708 | 483.5 2. | 710e+004 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

### Final Parameters

| Rsq | | 0.9920 |
|--------------------|-----|----------|
| Rsq_adjusted | | 0.9903 |
| Corr_XY | | -0.9960 |
| No_points_lambda_z | | 7 |
| Lambda_z | 1/h | 0.0225 |
| Lambda_z_lower | h | 48.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 30.7528 |
| Tlag | h | 1.5000 |

| Tmax | h | 24.0000 |
|-------------------|------------|------------|
| Cmax | ng/mL | 7.8400 |
| Cmax_D | ng/mL/mg | 0.0174 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 0.4160 |
| AUClast | h*ng/mL | 483.5428 |
| AUCall | h*ng/mL | 483.5428 |
| AUCINF_obs | h*ng/mL | 501.9995 |
| AUCINF_D_obs | h*ng/mL/mg | 1.1156 |
| AUC_%Extrap_obs | % | 3.6766 |
| Vz_F_obs | L | 39771.2079 |
| CI_F_obs | L/h | 896.4152 |
| AUCINF_pred | h*ng/mL | 500.7980 |
| AUCINF_D_pred | h*ng/mL/mg | 1.1129 |
| AUC_%Extrap_pred | % | 3.4455 |
| Vz_F_pred | L | 39866.6228 |
| CI_F_pred | L/h | 898.5658 |
| AUMClast | h*h*ng/mL | 27099.5522 |
| AUMCINF_obs | h*h*ng/mL | 31019.1346 |
| AUMC_%Extrap_obs | % | 12.6360 |
| AUMCINF_pred | h*h*ng/mL | 30763.9841 |
| AUMC_%Extrap_pred | % | 11.9114 |
| MRTlast | h | 56.0437 |
| MRTINF_obs | h | 61.7912 |
| MRTINF_pred | h | 61.4299 |
| AUC0_24 | h*ng/mL | 93.9158 |

WinNonlin 7.0.0.2535

PARAMCD=M7A,SUBJID=PI ,APERIOD=2,TRTAN=2,TRTA=2 x 250 mg TF3

Date: PI 09:27:26 Time:


## Settings

Model: Plasma Data, Extravascular Administration Number of nonmissing observations: 22

Dose time: 0.00 450.00 Dose amount:

Calculation method: Linear Trapezoidal Rule for for Increasing Values, Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

| Summary Table | | | | | | |
|---|---|---|---|---|---|---|
| Time | Conc. | Pred. | Residual | AUC | AUMC | Weight |
| h | ng/mL | ng/mL | ng/mL | h*ng/n | nL h*h*ng/mL | |
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.500 | 0.2630 | | ( | 0.06575 | 0.09863 | |
| 2.000 | 0.3670 | | | 0.2233 | 0.3808 | |
| 3.000 | 1.010 | | | 0.9118 | 2.263 | |
| 4.000 | 1.950 | | | 2.392 | 7.678 | |
| 6.000 | 3.120 | | | 7.462 | 34.20 | |
| 8.000 | 4.360 | | | 14.94 | 87.80 | |
| 12.00 | 5.840 | | | 35.34 | 297.7 | |
| 16.00 | 7.500 | | | 62.02 | 677.9 | |
| 24.02 | 11.30 | | | 137.4 | 2247. | |
| 36.00 | 10.10 | | | 265.5 | 6076. | |
| 48.00 | 11.00 | | | 392.1 1.1 | 43e+004 | |

| 60.00 | 8.970 | | | 511.5 1.785e+004 | |
|---------|-------|-------|----------|------------------|-------|
| 72.00 | 9.890 | | | 624.6 2.535e+004 | |
| 96.00 | 8.430 | | | 844.0 4.371e+004 | |
| 120.0 * | 5.550 | 5.592 | -0.04182 | 1009. 6.143e+004 | 1.000 |
| 144.0 * | 3.500 | 3.448 | 0.05215 | 1116. 7.542e+004 | 1.000 |
| 168.0 * | 2.110 | 2.126 | -0.01590 | 1182, 8,563e+004 | 1.000 |

#### Final Parameters

| Rsq | | 0.9993 |
|--------------------|------------|-------------|
| Rsq_adjusted | | 0.9986 |
| Corr_XY | | -0.9996 |
| No_points_lambda_z | | 3 |
| Lambda_z | 1/h | 0.0201 |
| Lambda_z_lower | h | 120.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 34.4026 |
| Tlag | h | 1.0000 |
| Tmax | h | 24.0167 |
| Cmax | ng/mL | 11.3000 |
| Cmax_D | ng/mL/mg | 0.0251 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 2.1100 |
| AUClast | h*ng/mL | 1182.0003 |
| AUCall | h*ng/mL | 1182.0003 |
| AUCINF_obs | h*ng/mL | 1286.7247 |
| AUCINF_D_obs | h*ng/mL/mg | 2.8594 |
| AUC_%Extrap_obs | % | 8.1388 |
| Vz_F_obs | L | 17357.7026 |
| Cl_F_obs | L/h | 349.7252 |
| AUCINF_pred | h*ng/mL | 1287.5138 |
| AUCINF_D_pred | h*ng/mL/mg | 2.8611 |
| AUC_%Extrap_pred | % | 8.1951 |
| Vz_F_pred | L | 17347.0644 |
| Cl_F_pred | L/h | 349.5108 |
| AUMClast | h*h*ng/mL | 85634.6553 |
| AUMCINF_obs | h*h*ng/mL | 108426.0761 |
| AUMC_%Extrap_obs | % | 21.0202 |
| AUMCINF_pred | h*h*ng/mL | 108597.8077 |
| AUMC_%Extrap_pred | % | 21.1451 |
| MRTlast | h | 72.4489 |
| MRTINF_obs | h | 84.2652 |
| MRTINF_pred | h | 84.3469 |
| AUC0_24 | h*ng/mL | 137.1901 |

WinNonlin 7.0.0.2535

PARAMCD=M7A,SUBJID=PI ,APERIOD=2,TRTAN=2,TRTA=2 x 250 mg TF3

Date: pj Time: 09:27:25


### Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

```
00000000
П
\\
0000000 0 0 0 0 0000000
Π
П
0000000000000000000000
П
П
П
П
0000000
Π
П
```

Date: Time: PI 09:27:24


## Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

0.00 Dose time: 450.00 Dose amount:

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values
Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

### Summary Table

| Time | Conc. | Pred. | Residual | AUC | AUMC | Weight |
|---------|--------|--------|----------|-------------|-----------|--------|
| h | ng/mL | ng/mL | ng/mL | h*ng/mL | h*h*ng/mL | |
| | | | | | • | |
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.500 | 0.1430 | | | 0.03575 | .05363 | |
| 2.000 | 0.4110 | | | 0.1743 | 0.3128 | |
| 3.000 | 0.9090 | | | 0.8343 | 2.087 | |
| 4.000 | 1.650 | | | 2.114 | 6.751 | |
| 6.017 | 2.300 | | | 6.097 | 27.36 | |
| 8.000 | 3.110 | | | 11.46 | 65.76 | |
| 12.00 | 4.290 | | | 26.26 | 218.5 | |
| 16.10 | 5.790 | | | 46.93 | 515.1 | |
| 24.07 | 7.830 | | | 101.2 | 1637. | |
| 36.00 | 5.950 | | | 182.9 | 4069. | |
| 48.00 | 6.410 | | | 257.0 | 7200. | |
| 60.02 | 4.190 | | | 319.8 1.056 | e+004 | |
| 72.00 * | 5.150 | 5.541 | -0.3912 | 375.8 1.42 | 9e+004 | 1.000 |
| 96.17 * | 3.410 | 3.241 | 0.1689 | 477.7 2.27 | 8e+004 | 1.000 |
| 120.0 * | 1.940 | 1.910 | 0.03020 | 539.9 2.94 | 13e+004 | 1.000 |
| 146.9 * | 1.190 | 1.051 | 0.1395 | 581.2 3.49 | 0e+004 | 1.000 |
| 168.0 * | 0.5850 | 0.6582 | -0.07322 | 599.1 3.7 | 70e+004 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

#### Final Parameters

| i marr alamotors | | |
|--------------------|----------|----------|
| Rsq | | 0.9872 |
| Rsq_adjusted | | 0.9829 |
| Corr_XY | | -0.9936 |
| No points lambda z | | 5 |
| Lambda_z | 1/h | 0.0222 |
| Lambda_z_lower | h | 72.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 31.2343 |
| Tlag | h | 1.0000 |
| Tmax | h | 24.0667 |
| Cmax | ng/mL | 7.8300 |
| Cmax_D | ng/mL/mg | 0.0174 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 0.5850 |
| AUClast | h*ng/mL | 599.1435 |
| AUCall | h*ng/mL | 599.1435 |

AUCINF\_obs AUCINF\_D\_obs h\*ng/mL 625.5045 h\*ng/mL/mg 1.3900 AUC\_%Extrap\_obs % 4.2144 32418.1193 Vz\_F\_obs L CI\_F\_obs AUCINF\_pred L/h 719.4193 h\*ng/mL 628.8041 AUCINF\_D\_pred h\*ng/mL/mg 1.3973 AUC\_%Extrap\_pred Vz\_F\_pred CI\_F\_pred AUMClast 4.7170 % L 32248.0091 L/h 715.6442 h\*h\*ng/mL 37701.8848 h\*h\*ng/mL 43318.3955 AUMCINF\_obs AUMC\_%Extrap\_obs 12.9656 AUMCINF\_pred h\*h\*ng/mL 44021.4077 AUMC\_%Extrap\_pred 14.3556 MRTlast h 62.9263 MRTINF\_obs 69.2535 h MRTINF\_pred h 70.0081 AUC0\_24 100.6572 h\*ng/mL

WinNonlin 7.0.0.2535

PARAMCD=M7A,SUBJID=PI ,APERIOD=2,TRTAN=2,TRTA=2 x 250 mg TF3

Date: PI Time: 09:27:25


#### Settings

\_\_\_\_

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting

Lambda\_z method: Find best fit for lambda\_z, Log regression

| | ' | | | | | |
|---------|--------|----------|----------|-----------|------------|--------|
| Time | Conc. | Pred. | Residual | AUC | AUMC | Weight |
| h | ng/mL | ng/mL | ng/mL | | nL h*h*ng/ | |
| | | <u>-</u> | | | | |
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2667 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.000 | 0.1140 | | | 0.01425 | 0.01425 | |
| 1.500 | 0.3890 | | | 0.1400 | 0.1886 | |
| 2.000 | 0.7540 | | | 0.4258 | 0.7115 | |
| 3.000 | 1.500 | | | 1.553 | 3.716 | |
| 4.000 | 2.770 | | | 3.688 | 11.51 | |
| 6.000 | 4.180 | | | 10.64 | 47.67 | |
| 8.000 | 7.520 | | | 22.34 | 132.9 | |
| 12.00 | 9.070 | | | 55.52 | 470.9 | |
| 16.00 | 12.20 | | | 98.06 | 1079. | |
| 24.00 | 20.40 | | | 228.5 | 3818. | |
| 36.00 | 13.60 | | | 429.7 | 9774. | |
| 48.00 | 16.20 | | | 608.5 1.7 | | |
| 60.00 | 10.20 | | | 764.1 2.5 | | |
| 72.00 * | 9.940 | 9.861 | 0.07859 | | .368e+004 | 1.000 |
| 96.00 * | 6.410 | 6.340 | 0.06952 | | .973e+004 | 1.000 |
| 120.0 * | 4.160 | 4.077 | 0.08334 | | .312e+004 | 1.000 |
| 144.0 * | 2.360 | 2.621 | -0.2611 | | 309e+004 | 1.000 |
| 168.0 * | 1.800 | 1.685 | 0.1147 | 1329. 8. | .080e+004 | 1.000 |

#### Final Parameters

| Rsq | | 0.9919 |
|--------------------|------------|-------------|
| Rsq_adjusted | | 0.9892 |
| Corr XY | | -0.9959 |
| No_points_lambda_z | | 5 |
| Lambda_z | 1/h | 0.0184 |
| Lambda z lower | h | 72.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL Lambda z | h | 37.6646 |
| Tlag | h | 0.7500 |
| Tmax | h | 24.0000 |
| Cmax | ng/mL | 20.4000 |
| Cmax_D | ng/mL/mg | 0.0453 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 1.8000 |
| AUClast | h*ng/mL | 1328.8158 |
| AUCall | h*ng/mL | 1328.8158 |
| AUCINF_obs | h*ng/mL | 1426.6251 |
| AUCINF_D_obs | h*ng/mL/mg | 3.1703 |
| AUC_%Extrap_obs | % | 6.8560 |
| Vz_F_obs | L | 17139.9782 |
| Cl_F_obs | L/h | 315.4298 |
| AUCINF_pred | h*ng/mL | 1420.3908 |
| AUCINF_D_pred | h*ng/mL/mg | 3.1564 |
| AUC_%Extrap_pred | % | 6.4472 |
| Vz_F_pred | L | 17215.2070 |
| Cl_F_pred | L/h | 316.8142 |
| AUMClast | h*h*ng/mL | 80803.2468 |
| AUMCINF_obs | h*h*ng/mL | 102550.0171 |
| AUMC_%Extrap_obs | % | 21.2060 |
| AUMCINF_pred | h*h*ng/mL | 101163.9117 |
| AUMC_%Extrap_pred | % | 20.1264 |
| MRTlast | h | 60.8085 |
| MRTINF_obs | h | 71.8829 |
| MRTINF_pred | h | 71.2226 |
| AUC0_24 | h*ng/mL | 228.4578 |
| | - | |

WinNonlin 7.0.0.2535

PARAMCD=M7A,SUBJID=PI ,APERIOD=1,TRTAN=2,TRTA=2 x 250 mg TF3

Date: pj Time: 09:27:25


## Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

## Summary Table

Time Conc. Pred. Residual AUC AUMC Weight ng/mL ng/mL h\*ng/mL h\*h\*ng/mL h ng/mL 0.0000 0.0000 0.0000 0.0000

| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
|---------|--------|-------|----------|----------|------------|-------|
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.500 | 0.1910 | | | 0.04775 | 0.07163 | |
| 2.000 | 0.5420 | | | 0.2310 | 0.4143 | |
| 3.000 | 1.190 | | | 1.097 | 2.741 | |
| 4.000 | 2.030 | | | 2.707 | 8.586 | |
| 6.000 | 3.610 | | | 8.347 | 38.37 | |
| 8.017 | 4.360 | | | 16.38 | 95.45 | |
| 12.00 | 5.270 | | | 35.56 | 291.0 | |
| 16.00 | 6.310 | | | 58.72 | 619.4 | |
| 24.00 | 8.520 | | | 118.0 | 1841. | |
| 36.00 | 6.670 | | | 208.7 | 4540. | |
| 48.00 | 9.440 | | | 305.4 | 8699. | |
| 60.03 | 7.370 | | | 406.0 1. | 411e+004 | |
| 72.00 * | 7.300 | 7.075 | 0.2253 | 493.8 1 | .990e+004 | 1.000 |
| 96.03 * | 4.520 | 4.603 | -0.08263 | 633.2 3 | .148e+004 | 1.000 |
| 120.0 * | 2.940 | 2.998 | -0.05792 | 721.2 4 | .091e+004 | 1.000 |
| 144.0 * | 1.890 | 1.952 | -0.06153 | 778.2 4 | .839e+004 | 1.000 |
| 168.0 * | 1.320 | 1.270 | 0.04963 | 816.4 5 | 5.431e+004 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

| Rsq | | 0.9977 |
|-------------------------------|------------|------------|
| Rsq_adjusted | | 0.9970 |
| Corr_XY | | -0.9989 |
| No_points_lambda_z | | 5 |
| Lambda_z | 1/h | 0.0179 |
| Lambda_z_lower | h | 72.0000 |
| Lambda z upper | h | 168.0000 |
| HL_Lambda_z | h | 38.7500 |
| Tlag | h | 1.0000 |
| Tmax | h | 48.0000 |
| Cmax | ng/mL | 9.4400 |
| Cmax_D | ng/mL/mg | 0.0210 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 1.3200 |
| AUClast | h*ng/mL | 816.3601 |
| AUCall | h*ng/mL | 816.3601 |
| AUCINF_obs | h*ng/mL | 890.1539 |
| AUCINF_D_obs | h*ng/mL/mg | 1.9781 |
| AUC %Extrap obs | % | 8.2900 |
| Vz_F_obs | L | 28261.3909 |
| CI F obs | L/h | 505.5306 |
| AUCINF_pred | h*ng/mL | 887.3796 |
| AUCINF_D_pred | h*ng/mL/mg | 1.9720 |
| AUC %Extrap pred | % | 8.0033 |
| AUC_%Extrap_pred<br>Vz_F_pred | L | 28349.7466 |
| Cl_F_pred | L/h | 507.1110 |
| AUMClast | h*h*ng/mL | 54311.3950 |
| AUMCINF_obs | h*h*ng/mL | 70834.1596 |
| AUMC_%Extrap_obs | % | 23.3260 |
| AUMCINF_pred | h*h*ng/mL | 70212.9858 |
| AUMC %Extrap pred | % | 22.6476 |
| MRTlast | h | 66.5287 |
| MRTINF_obs | h | 79.5752 |
| MRTINF_pred | h | 79.1240 |
| AUC0_24 | h*ng/mL | 118.0432 |

WinNonlin 7.0.0.2535

PARAMCD=M7A,SUBJID=PI ,APERIOD=1,TRTAN=2,TRTA=2 x 250 mg TF3

Date: P| 09:27:26

```
П
000000000
00000000
П
0000000000000000
00000000000000000
000000 0 0 0 0 0 000000
                              \  \, 0\  
                      Π
П
П
П
П
П
П
П
```

AUC\_%Extrap\_pred Vz\_F\_pred CI\_F\_pred AUMClast 4.2327 65833.1146 L L/h 1413.8941 h\*h\*ng/mL 18127.7153 AUMCINF\_obs h\*h\*ng/mL 20845.0826 AUMC\_%Extrap\_obs 13.0360 AUMCINF\_pred h\*h\*ng/mL 21018.1307 AUMC\_%Extrap\_pred 13.7520 MRTlast h 59.4744 MRTINF\_obs 65.6614 h MRTINF\_pred h 66.0387 AUC0\_24 h\*ng/mL 50.2685

WinNonlin 7.0.0.2535

PARAMCD=M7A,SUBJID=PI ,APERIOD=1,TRTAN=2,TRTA=2 x 250 mg TF3

Date: PI Time: 09:27:26


### Settings

\_\_\_\_

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

## Summary Table

| Time | Conc. | Pred. | Residual | AUC | AUMC | Weight |
|---------|--------|--------|-----------|-------------|-----------|--------|
| h | ng/mL | ng/mL | ng/mL | . h*ng/mL | h*h*ng/mL | |
| | | | | | • | |
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.8167 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.017 | 0.1080 | | | 0.01080 0 | .01098 | |
| 1.500 | 0.2230 | | | 0.09079 | 0.1184 | |
| 2.000 | 0.4240 | | | 0.2525 | 0.4140 | |
| 3.000 | 1.390 | | | 1.160 | 2.923 | |
| 4.000 | 2.450 | | | 3.080 | 9.908 | |
| 6.000 | 3.290 | | | 8.820 | 39.45 | |
| 8.033 | 4.460 | | | 16.70 | 95.94 | |
| 12.00 | 4.680 | | | 34.83 | 278.4 | |
| 16.00 | 5.860 | | | 55.91 | 578.2 | |
| 24.00 | 5.950 | | | 103.1 | 1524. | |
| 36.00 | 4.540 | | | 165.7 | 3384. | |
| 48.02 | 4.320 | | | 218.9 | 5617. | |
| 60.08 | 3.120 | | | 263.4 | 8008. | |
| 72.00 | 2.140 | | | 294.4 1.004 | e+004 | |
| 95.73 * | 1.320 | 1.320 | 0.0003104 | 334.7 1.3 | 38e+004 | 1.000 |
| 120.1 * | 0.8940 | 0.8927 | 0.001303 | 361.4 1.6 | 24e+004 | 1.000 |
| 144.0 * | 0.6070 | 0.6090 | -0.002041 | 379.0 1.8 | 56e+004 | 1.000 |
| 171.8 * | 0.3910 | 0.3904 | 0.0006497 | 392.7 2.0 | 70e+004 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

#### Final Parameters

Rsq

1.0000

| Dec edicated | | 1.0000 |
|--------------------------------|------------|------------|
| Rsq_adjusted<br>Corr XY | | -1.0000 |
| - | | 4 |
| No_points_lambda_z<br>Lambda_z | 1/h | 0.0160 |
| _ | | 95.7333 |
| Lambda_z_lower | h<br>h | 171.7667 |
| Lambda_z_upper | ••• | |
| HL_Lambda_z | h | 43.2657 |
| Tlag | h | 0.8167 |
| Tmax | , h | 24.0000 |
| Cmax | ng/mL | 5.9500 |
| Cmax_D | ng/mL/mg | 0.0132 |
| Tlast | , h | 171.7667 |
| Clast | ng/mL | 0.3910 |
| AUClast | h*ng/mL | 392.6793 |
| AUCall | h*ng/mL | 392.6793 |
| AUCINF_obs | h*ng/mL | 417.0852 |
| AUCINF_D_obs | h*ng/mL/mg | 0.9269 |
| AUC_%Extrap_obs | % | 5.8515 |
| Vz_F_obs | L | 67345.1331 |
| Cl_F_obs | L/h | 1078.9162 |
| AUCINF_pred | h*ng/mL | 417.0447 |
| AUCINF_D_pred | h*ng/mL/mg | 0.9268 |
| AUC_%Extrap_pred | % | 5.8424 |
| Vz_F_pred | L | 67351.6817 |
| Cl_F_pred | L/h | 1079.0211 |
| AUMClast | h*h*ng/mL | 20701.6217 |
| AUMCINF_obs | h*h*ng/mL | 26417.1454 |
| AUMC_%Extrap_obs | % | 21.6357 |
| AUMCINF_pred | h*h*ng/mL | 26407.6485 |
| AUMC_%Extrap_pred | % | 21.6075 |
| MRTlast | h | 52.7189 |
| MRTINF_obs | h | 63.3375 |
| MRTINF_pred | h | 63.3209 |
| AUC0_24 | h*ng/mL | 103.1464 |

WinNonlin 7.0.0.2535

PARAMCD=M7A,SUBJID=p\_\_\_\_\_,APERIOD=2,TRTAN=1,TRTA=5 x 100 mg TF3

Date: PI 09:27:24 Time:


### Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 18

0.00 Dose time: Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values
Weighting for lambda\_z calculations: Uniform weighting
Lambda\_z method: Find best fit for lambda\_z, Log regression

| summary rable | | | | | | |
|---------------|--------|-------|----------|---------|--------------|--------|
| Time | Conc. | Pred. | Residual | AUC | AUMC | Weight |
| h | ng/mL | ng/mL | ng/mL | h*ng/m | nL h*h*ng/mL | |
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.000 | 0.1310 | | | 0.01638 | 0.01638 | |
| 1.500 | 0.2120 | | | 0.1021 | 0.1286 | |
| 2.000 | 0.3430 | | | 0.2409 | 0.3796 | |
| 3.000 | 1.250 | | | 1.037 | 2.598 | |

| 4.000 | 2.360 | | | 2.842 | 9.193 | |
|---------|-------|-------|----------|-------|-------|-------|
| 6.000 | 3.540 | | | 8.742 | 39.87 | |
| 8.000 | 4.870 | | | 17.15 | 100.1 | |
| 12.00 | 4.990 | | | 36.87 | 297.8 | |
| 16.00 | 5.560 | | | 57.97 | 595.4 | |
| 24.00 | 6.110 | | | 104.7 | 1538. | |
| 36.00 * | 4.470 | 4.527 | -0.05666 | 167.6 | 3407. | 1.000 |
| 48.00 * | 3.790 | 3.548 | 0.2423 | 217.1 | 5476. | 1.000 |
| 60.00 * | 2.530 | 2.780 | -0.2504 | 254.5 | 7481. | 1.000 |
| 72.00 * | 2.270 | 2.179 | 0.09094 | 283.3 | 9377. | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

| Rsq | | 0.9516 |
|--------------------|------------|------------|
| Rsq_adjusted | | 0.9274 |
| Corr_XY | | -0.9755 |
| No_points_lambda_z | | 4 |
| Lambda_z | 1/h | 0.0203 |
| Lambda_z_lower | h | 36.0000 |
| Lambda_z_upper | h | 72.0000 |
| HL_Lambda_z | h | 34.1316 |
| Tlag | h | 0.7500 |
| Tmax | h | 24.0000 |
| Cmax | ng/mL | 6.1100 |
| Cmax D | ng/mL/mg | 0.0136 |
| Tlast | h | 72.0000 |
| Clast | ng/mL | 2.2700 |
| AUClast | h*ng/mL | 283.2524 |
| AUCall | h*ng/mL | 283.2524 |
| AUCINF_obs | h*ng/mL | 395.0305 |
| AUCINF_D_obs | h*ng/mL/mg | 0.8778 |
| AUC %Extrap obs | % | 28.2961 |
| Vz_F_obs | L | 56093.4985 |
| CI_F_obs | L/h | 1139.1526 |
| AUCINF_pred | h*ng/mL | 390.5524 |
| AUCINF_D_pred | h*ng/mL/mg | 0.8679 |
| AUC_%Extrap_pred | % | 27.4739 |
| Vz_F_pred | L | 56736.6747 |
| CI_F_pred | L/h | 1152.2143 |
| AUMClast | h*h*ng/mL | 9376.8831 |
| AUMCINF_obs | h*h*ng/mL | 22929.0119 |
| AUMC_%Extrap_obs | % | 59.1047 |
| AUMCINF_pred | h*h*ng/mL | 22386.0770 |
| AUMC_%Extrap_pred | % | 58.1129 |
| MRTlast | h | 33.1043 |
| MRTINF_obs | h | 58.0437 |
| MRTINF_pred | h | 57.3190 |
| AUC0_24 | h*ng/mL | 104.6524 |
| _ | - | |

WinNonlin 7.0.0.2535

PARAMCD=M7A,SUBJID=PI \_\_\_\_\_,APERIOD=2,TRTAN=1,TRTA=5 x 100 mg TF3

Date: PI Time: 09:27:26


## Settings

-----

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00

Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

```
Π
П
Π
\, 0
                                       П
Π
П
Π
Π
```

AUC0\_24 h\*ng/mL 135.0296

WinNonlin 7.0.0.2535 PARAMCD=M7A,SUBJID=PI ,APERIOD=2,TRTAN=1,TRTA=5 x 100 mg TF3

> PI 09:27:26 Date: Time:


## Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

### Summary Table

| Time | Conc. | Pred. | Residual | AUC | AUMC | Weight |
|---------|--------|--------|----------|-----------|------------|--------|
| h | ng/mL | ng/mL | ng/mL | . h*ng/ml | . h*h*ng/n | nL |
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.500 | 0.1860 | | | 0.04650 | 0.06975 | |
| 2.000 | 0.3530 | | | 0.1813 | 0.3160 | |
| 3.000 | 0.9730 | | | 0.8443 | 2.129 | |
| 4.000 | 1.850 | | | 2.256 | 7.288 | |
| 6.000 | 3.210 | | | 7.316 | 33.95 | |
| 8.000 | 4.180 | | | 14.71 | 86.65 | |
| 12.00 | 4.810 | | | 32.69 | 269.0 | |
| 16.00 | 5.180 | | | 52.67 | 550.2 | |
| 24.00 | 6.560 | | | 99.63 | 1511. | |
| 36.00 | 4.490 | | | 165.1 | 3452. | 4 000 |
| 48.00 * | 4.820 | 4.658 | 0.1622 | 221.0 | 5810. | 1.000 |
| 60.00 * | 3.210 | 3.532 | -0.3216 | 268.5 | 8357. | 1.000 |
| 72.00 * | 2.730 | 2.678 | 0.05231 | 304.1 1.0 | | 1.000 |
| 96.00 * | 1.680 | 1.539 | 0.1406 | 356.0 1.5 | | 1.000 |
| 120.0 * | 0.8000 | 0.8850 | -0.08496 | | 04e+004 | 1.000 |
| 144.0 * | 0.5740 | 0.5088 | 0.06524 | | )19e+004 | 1.000 |
| 168.0 * | 0.2740 | 0.2925 | -0.01848 | 410.5 2.1 | 69e+004 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

### Final Parameters

| Rsq | | 0.9927 |
|--------------------|----------|----------|
| Rsq_adjusted | | 0.9912 |
| Corr_XY | | -0.9963 |
| No_points_lambda_z | | 7 |
| Lambda_z | 1/h | 0.0231 |
| Lambda_z_lower | h | 48.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 30.0508 |
| Tlag | h | 1.0000 |
| Tmax | h | 24.0000 |
| Cmax | ng/mL | 6.5600 |
| Cmax_D | ng/mL/mg | 0.0146 |

| Tlast | h | 168.0000 |
|-------------------|------------|------------|
| Clast | ng/mL | 0.2740 |
| AUClast | h*ng/mL | 410.5374 |
| AUCall | h*ng/mL | 410.5374 |
| AUCINF_obs | h*ng/mL | 422.4164 |
| AUCINF_D_obs | h*ng/mL/mg | 0.9387 |
| AUC_%Extrap_obs | % | 2.8122 |
| Vz_F_obs | L | 46185.1053 |
| CI_F_obs | L/h | 1065.2996 |
| AUCINF_pred | h*ng/mL | 423.2174 |
| AUCINF_D_pred | h*ng/mL/mg | 0.9405 |
| AUC_%Extrap_pred | % | 2.9961 |
| Vz_F_pred | L | 46097.6871 |
| Cl_F_pred | L/h | 1063.2832 |
| AUMClast | h*h*ng/mL | 21691.3891 |
| AUMCINF_obs | h*h*ng/mL | 24202.0695 |
| AUMC_%Extrap_obs | % | 10.3738 |
| AUMCINF_pred | h*h*ng/mL | 24371.3761 |
| AUMC_%Extrap_pred | % | 10.9965 |
| MRTlast | h | 52.8366 |
| MRTINF_obs | h | 57.2943 |
| MRTINF_pred | h | 57.5859 |
| AUC0_24 | h*ng/mL | 99.6258 |

WinNonlin 7.0.0.2535

PARAMCD=M7A,SUBJID=PI ,APERIOD=1,TRTAN=1,TRTA=5 x 100 mg TF3

PI 09:27:24 Date: Time:


## Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 450.00 Dose amount:

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values
Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

| Time | Conc. | Pred. | Residual | AUC | AUMC | Weight |
|---------|--------|-------|----------|-------------|-----------|--------|
| h | ng/mL | ng/mL | ng/mL | h*ng/mL | h*h*ng/mL | |
| 0.0000 | 0.0000 | | | 0.0000 | 0.000 | |
| 0.0000 | 0.0000 | | | | 0.0000 | |
| 0.2500 | 0.0000 | | | | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.050 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 2.017 | 0.0000 | | | 0.0000 | 0.0000 | |
| 3.000 | 0.2540 | | | 0.1249 | 0.3746 | |
| 4.000 | 0.4630 | | | 0.4834 | 1.682 | |
| 6.000 | 0.9970 | | | 1.943 | 9.516 | |
| 8.000 | 1.880 | | | 4.820 | 30.54 | |
| 12.00 | 3.440 | | | 15.46 | 143.2 | |
| 16.00 | 5.380 | | | 33.10 | 397.9 | |
| 24.00 | 8.540 | | | 88.78 | 1562. | |
| 36.00 | 7.510 | | | 184.9 | 4435. | |
| 48.00 | 8.340 | | | 280.0 | 8459. | |
| 60.00 | 5.230 | | | 360.0 1.274 | e+004 | |
| 72.00 * | 5.150 | 5.444 | -0.2944 | 422.3 1.68 | | 1.000 |
| 96.07 * | 3.580 | 3.484 | 0.09622 | 526.2 2.55 | | 1.000 |

| 120.0 * | 2.300 | 2.235 | 0.06526 | 595.4 3.292e+004 | 1.000 |
|---------|--------|--------|----------|------------------|-------|
| 144.1 * | 1.550 | 1.429 | 0.1214 | 641.3 3.894e+004 | 1.000 |
| 168.6 * | 0.8360 | 0.9074 | -0.07141 | 669.6 4.333e+004 | 1.000 |

#### Final Parameters

0.9911 Rsq Rsq\_adjusted 0.9881 Corr\_XÝ -0.9955 No\_points\_lambda\_z 5 Lambda\_z 1/h 0.0186 Lambda z lower h 72.0000 Lambda\_z\_upper 168.5833 h HL\_Lambda\_z h 37.3639 Tlag 2.0167 h 24.0000 Tmax h Cmax 8.5400 ng/mL Cmax\_D ng/mL/mg 0.0190 Tlast h 168.5833 0.8360 Clast ng/mL AUClast h\*ng/mL 669.5743 AUCall h\*ng/mL 669,5743 AUCINF\_obs 714.6386 h\*ng/mL AUCINF\_D\_obs h\*ng/mL/mg 1.5881 AUC\_%Extrap\_obs Vz\_F\_obs CLF\_obs AUCINF\_pred 6.3059 33943.1733 L L/h 629.6889 h\*ng/mL 718.4881 AUCINF\_D\_pred h\*ng/mL/mg 1.5966 AUC\_%Extrap\_pred % 6.8079 Vz\_F\_pred L 33761.3157 626.3152 CI\_F\_pred L/h **AUM**Clast h\*h\*ng/mL 43329.7220 AUMCINF obs 53355.9896 h\*h\*ng/mL AUMC\_%Extrap\_obs 18.7913 AUMCINF\_pred h\*h\*ng/mL 54212.4459 AUMC\_%Extrap\_pred 20.0742 MRTlast 64.7123 MRTINF\_obs 74.6615 h MRTINF\_pred h 75.4535 88.7804 AUC0\_24 h\*ng/mL

WinNonlin 7.0.0.2535

PARAMCD=M7A,SUBJID=PI ,APERIOD=1,TRTAN=1,TRTA=5 x 100 mg TF3

Date: PI Time: 09:27:25


Settings

-----

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

Summary Table

-----

| Time<br>h | Conc.<br>ng/mL | Pred.<br>ng/mL | | | AUM (<br>nL h*h*ng | |
|---|---|---|---|---|---|---|
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7667 | 0.1070 | | | 0.01427 | 0.01094 | |
| 1.000 | 0.2280 | | | 0.05335 | 0.04711 | |
| 1.500 | 0.6630 | | | 0.2761 | 0.3527 | |
| 2.000 | 1.230 | | | 0.7494 | 1.216 | |
| 3.000 | 2.320 | | | 2.524 | 5.926 | |
| 4.000 | 3.350 | | | 5.359 | 16.11 | |
| 6.000 | 4.170 | | | 12.88 | 54.53 | |
| 8.017 | 5.570 | | | 22.70 | 124.8 | |
| 12.00 | 6.490 | | | 46.72 | 368.8 | |
| 16.00 | 8.380 | | | 76.46 | 792.7 | |
| 24.02 | 12.80 | | | 161.4 | 2562. | |
| 36.00 | 8.250 | | | 285.5 | 6233. | |
| 48.00 | 8.230 | | | 384.4 1.0 | 39e+004 | |
| 60.00 | 5.030 | | | 462.4 1.4 | 56e+004 | |
| 72.00 * | 5.480 | 5.497 | -0.01679 | 525.4 1. | 874e+004 | 1.000 |
| 96.00 * | 3.840 | 3.623 | 0.2174 | 636.1 2. | 796e+004 | 1.000 |
| 120.0 * | 2.130 | 2.387 | -0.2574 | 705.7 3. | 539e+004 | 1.000 |
| 144.0 * | 1.680 | 1.573 | 0.1066 | 751.2 4. | 138e+004 | 1.000 |
| 168.0 * | 1.030 | 1.037 | -0.006921 | 783.1 4 | .632e+004 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

| Rsq | | 0.9882 |
|--------------------|------------|------------|
| Rsq_adjusted | | 0.9843 |
| Corr_XY | | -0.9941 |
| No_points_lambda_z | | 5 |
| Lambda_z | 1/h | 0.0174 |
| Lambda_z_lower | h | 72.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL Lambda z | h | 39.8956 |
| Tlag | h | 0.5000 |
| Tmax | h | 24.0167 |
| Cmax | ng/mL | 12.8000 |
| Cmax_D | ng/mL/mg | 0.0284 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 1.0300 |
| AUClast | h*ng/mL | 783.1276 |
| AUCall | h*ng/mL | 783,1276 |
| AUCINF_obs | h*ng/mL | 842.4114 |
| AUCINF_D_obs | h*ng/mL/mg | 1.8720 |
| AUC_%Extrap_obs | % | 7.0374 |
| Vz_F_obs | L | 30745.9066 |
| CI F obs | L/h | 534.1808 |
| AUCINF_pred | h*ng/mL | 842.8098 |
| AUCINF_D_pred | h*ng/mL/mg | 1.8729 |
| AUC %Extrap_pred | % | 7.0813 |
| Vz_F_pred | L | 30731.3737 |
| CI F pred | L/h | 533.9283 |
| AUMClast | h*h*ng/mL | 46323,1661 |
| AUMCINF_obs | h*h*ng/mL | 59695.0555 |
| AUMC %Extrap obs | % | 22,4003 |
| AUMCINF_pred | h*h*ng/mL | 59784.9126 |
| AUMC %Extrap pred | % | 22,5170 |
| MRTlast | h | 59,1515 |
| MRTINF_obs | h | 70.8621 |
| MRTINF_pred | h | 70.9352 |
| AUC0 24 | h*ng/mL | 161.1433 |
| | • | |

WinNonlin 7.0.0.2535
PARAMCD=M7A,SUBJID=PI ,APERIOD=1,TRTAN=1,TRTA=5 x 100 mg TF3

```
0000000000
                                                      0000000
00000000
0\,0\,0\,0\,0\,0\,0\,0\,0\,0\,0\,0\,0\,0\,0\,0
             000000
П
0000000000000
00000000000000000
П
Π
П
Π
Π
П
П
                                              0000 000 00
00000000
```

| Vz_F_obs | L | 35112.3993 |
|-------------------|------------|------------|
| CI_F_obs | L/h | 665.5952 |
| AUCINF_pred | h*ng/mL | 676.7689 |
| AUCINF_D_pred | h*ng/mL/mg | 1.5039 |
| AUC_%Extrap_pred | % | 6.7187 |
| Vz_F_pred | L | 35077.0009 |
| CI_F_pred | L/h | 664.9242 |
| AUMClast | h*h*ng/mL | 39029.9218 |
| AUMCINF_obs | h*h*ng/mL | 48916.9406 |
| AUMC_%Extrap_obs | % | 20.2119 |
| AUMCINF_pred | h*h*ng/mL | 49067.5565 |
| AUMC_%Extrap_pred | % | 20.4568 |
| MRTlast | h | 61.8248 |
| MRTINF_obs | h | 72.3531 |
| MRTINF_pred | h | 72.5027 |
| AUC0_24 | h*ng/mL | 117.9921 |
| | _ | |

WinNonlin 7.0.0.2535

PARAMCD=M7A,SUBJID=PI ,APERIOD=1,TRTAN=1,TRTA=5 x 100 mg TF3

Date: PI 09:27:25 Time:


## Settings

Model: Plasma Data, Extravascular Administration Number of nonmissing observations: 22

Dose time: 0.00 450.00 Dose amount:

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values
Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

| Time<br>h | Conc.<br>ng/mL | Pred.<br>ng/mL | Residual<br>ng/mL | AUC<br>h*ng/m | AUMC<br>L h*h*ng/n | Weight<br>nL |
|---|---|---|---|---|---|---|
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.8167 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.017 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.500 | 0.1290 | | | | 0.04676 | |
| 2.000 | 0.2920 | | | 0.1364 | 0.2411 | |
| 3.000 | 0.9400 | | | 0.7524 | 1.943 | |
| 4.000 | 1.370 | | | 1.907 | 6.093 | |
| 6.000 | 2.170 | | | 5.447 | 24.59 | |
| 8.000 | 2.860 | | | 10.48 | 60.49 | |
| 12.00 | 4.110 | | | 24.42 | 204.9 | |
| 16.00 | 5.630 | | | 43.90 | 483.7 | |
| 24.00 | 8.360 | | | 99.86 | 1647. | |
| 36.00 | 10.00 | | | 210.0 | 5010. | |
| 48.00 | 11.60 | | | 339.6 1.05 | | |
| 60.00 | 9.000 | 0.707 | 0.4167 | 462.6 1.71 | | 1.000 |
| 72.00 *<br>96.00 * | 9.380<br>7.050 | 9.797<br>6.670 | -0.4167<br>0.3804 | 572.8 2.4 | 75e+004 | 1.000 |
| 120.0 * | 4.730 | 4.541 | 0.3804 | | 71e+004 | 1.000 |
| 144.0 * | 2.870 | 3.091 | -0.2212 | 997.5 6.7 | | 1.000 |
| 168.0 * | 2.150 | 2.104 | 0.04551 | | 371e+004 | 1.000 |
| 100.0 | 2.100 | 2.104 | 0.04001 | 1007. 7.0 | ,,,,,,,,, | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

| Rsq | | 0.9915 |
|--------------------|------------|-------------|
| Rsq_adjusted | | 0.9887 |
| Corr_XY | | -0.9958 |
| No_points_lambda_z | | 5 |
| Lambda_z | 1/h | 0.0160 |
| Lambda_z_lower | h | 72.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 43.2660 |
| Tlag | h | 1.0167 |
| Tmax | h | 48.0000 |
| Cmax | ng/mL | 11.6000 |
| Cmax D | ng/mL/mg | 0.0258 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 2.1500 |
| AUClast | h*ng/mL | 1057.3563 |
| AUCall | h*ng/mL | 1057.3563 |
| AUCINF_obs | h*ng/mL | 1191.5586 |
| AUCINF_D_obs | h*ng/mL/mg | 2.6479 |
| AUC_%Extrap_obs | % | 11.2628 |
| Vz_F_obs | L | 23573.2159 |
| CI_F_obs | L/h | 377.6566 |
| AUCINF_pred | h*ng/mL | 1188.7181 |
| AUCINF_D_pred | h*ng/mL/mg | 2.6416 |
| AUC_%Extrap_pred | % | 11.0507 |
| Vz_F_pred | L | 23629.5458 |
| Cl_F_pred | L/h | 378.5591 |
| AUMClast | h*h*ng/mL | 76708.7918 |
| AUMCINF_obs | h*h*ng/mL | 107631.6638 |
| AUMC_%Extrap_obs | % | 28.7303 |
| AUMCINF_pred | h*h*ng/mL | 106977.1495 |
| AUMC_%Extrap_pred | % | 28.2942 |
| MRTlast | h | 72.5477 |
| MRTINF_obs | h | 90.3285 |
| MRTINF_pred | h | 89.9937 |
| AUC0_24 | h*ng/mL | 99.8574 |

WinNonlin 7.0.0.2535

PARAMCD=M7A,SUBJID=PI ,APERIOD=1,TRTAN=1,TRTA=5 x 100 mg TF3

PI 09:27:26 Date: Time:


### Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values, Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

| _ | Time<br>h | Conc.<br>ng/mL | Pred.<br>ng/mL | Residual<br>ng/mL | AUC<br>h*ng/mL | AUMC<br>h*h*ng/mL | Weight |
|---|---|---|---|---|---|---|---|
| _ | 0.0000<br>0.2667<br>0.5000<br>0.7500 | 0.0000<br>0.0000<br>0.0000<br>0.0000 | | | 0.0000<br>0.0000 | 0.0000<br>0.0000<br>0.0000<br>0.0000 | |

```
Π
Π
Π
Π
П
000000
Π
```

# WinNonlin Core Output - Tepotinib Metabolite MSC2571109A

WinNonlin 7.0.0.2535

PARAMCD=M9A,SUBJID=PI ,APERIOD=1,TRTAN=2,TRTA=2 x 250 mg TF3

Date: PI Time: 09:24:10


### Settings

\_\_\_\_

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

### Summary Table

| Time | Conc. | Pred. | Residual | AUC | AUMC | Weight |
|---------|--------|-------|----------|-------------|-----------|--------|
| h | ng/mL | ng/mL | ng/mL | h*ng/mL | h*h*ng/mL | |
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.000 | 1.080 | | | 0.1350 | 0.1350 | |
| 1.600 | 1.850 | | | 1.014 | 1.347 | |
| 2.217 | 4.960 | | | 3.114 | 5.650 | |
| 3.000 | 10.20 | | | 9.051 | 21.94 | |
| 4.000 | 16.60 | | | 22.45 | 70.44 | |
| 6.000 | 24.10 | | | 63.15 | 281.4 | |
| 8.000 | 34.30 | | | 121.6 | 700.4 | |
| 12.00 | 42.00 | | | 274.2 | 2257. | |
| 16.00 | 52.20 | | | 462.6 | 4936. | |
| 24.02 | 85.10 | | | 1013. 1.648 | e+004 | |
| 36.00 | 79.70 | | | 2000. 4.603 | e+004 | |
| 48.02 | 97.90 | | | 3067. 9.151 | e+004 | |
| 60.00 | 72.60 | | | 4081. 1.460 | e+005 | |
| 72.00 | 70.50 | | | 4940. 2.026 | e+005 | |
| 96.02 * | 52.40 | 52.27 | 0.1324 | 6405. 3.24 | 8e+005 | 1.000 |
| 120.0 * | 32.90 | 32.66 | 0.2448 | 7410. 4.32 | 4e+005 | 1.000 |
| 144.1 * | 19.90 | 20.36 | -0.4553 | 8033. 5.14 | 1e+005 1 | 1.000 |
| 168.0 * | 12.90 | 12.74 | 0.1618 | 8419. 5.74 | 0e+005 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

### Final Parameters

| Rsq | | 0.9993 |
|--------------------|-------|----------|
| Rsq_adjusted | | 0.9990 |
| Corr_XY | | -0.9997 |
| No_points_lambda_z | | 4 |
| Lambda z | 1/h | 0.0196 |
| Lambda z lower | h | 96.0167 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 35.3421 |
| Tlag | h | 0.7500 |
| Tmax | h | 48.0167 |
| Cmax | ng/mL | 97,9000 |

Cmax\_D ng/mL/mg 0.2176 168.0000 Tlast h Clast ng/mL 12.9000 8418.6346 AUClast h\*ng/mL **AUCall** 8418.6346 h\*ng/mL AUCINF\_obs h\*ng/mL 9076.3791 AUCINF\_Dobs
AUCINF\_D\_obs
AUC\_%Extrap\_obs
Vz\_F\_obs
CI\_F\_obs
AUCINF\_pred
AUCINF\_D\_pred
AUCINF\_D\_pred h\*ng/mL/mg 20.1697 % 7.2468 L 2527.9436 L/h 49.5792 h\*ng/mL 9068.1286 h\*ng/mL/mg 20.1514 AUC\_%Extrap\_pred 7.1624 % Vz\_F\_pred L 2530.2436 CI\_F\_pred L/h 49.6244 **AUMClast** h\*h\*ng/mL 573981.3758 AUMCINF\_obs 718019.4828 h\*h\*ng/mL AUMC\_%Extrap\_obs 20.0605 AUMCINF\_pred AUMC\_%Extrap\_pred 716212.7199 h\*h\*ng/mL 19.8588 MRTlast 68.1799 MRTINF\_obs 79.1086 h MRTINF\_pred h 78.9813 AUC0\_24 1011.4778 h\*ng/mL

WinNonlin 7.0.0.2535

PARAMCD=M9A,SUBJID=PI ,APERIOD=1,TRTAN=2,TRTA=2 x 250 mg TF3

Date: PI Time: 09:24:10


## Settings

-----

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

| Cummary racio | | | | | | |
|---------------|--------|-------|----------|-------------|-----------|--------|
| Time | Conc. | Pred. | Residual | AUC | AUMC | Weight |
| h | ng/mL | ng/mL | ng/mL | h*ng/mL | h*h*ng/mL | |
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7333 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.000 | 0.6050 | | | 0.08067 0 | .08067 | |
| 1.500 | 2.360 | | | 0.8219 | 1.117 | |
| 2.000 | 5.220 | | | 2.717 | 4.612 | |
| 3.000 | 12.80 | | | 11.73 | 29.03 | |
| 4.000 | 21.10 | | | 28.68 | 90.43 | |
| 6.000 | 26.90 | | | 76.68 | 336.2 | |
| 8.050 | 37.00 | | | 142.2 | 807.0 | |
| 12.00 | 47.70 | | | 309.5 | 2526. | |
| 16.05 | 60.30 | | | 528.2 | 5645. | |
| 24.02 | 86.20 | | | 1112, 1,775 | e+004 | |
| 36.00 | 85.00 | | | 2137, 4,851 | e+004 | |
| 48.00 | 91.00 | | | 3193, 9,308 | | |
| 60.00 | 58.80 | | | 4078. 1.405 | | |
| 72.00 * | 63.10 | 56.58 | 6.516 | 4810, 1.88 | | 1.000 |
| , 2.00 | 00.10 | 00.00 | 0.010 | 40 10. 1.00 | 00.000 | |

| 95.73 * | 26.90 | 27.77 | -0.8672 | 5817. 2.717e+005 | 1.000 |
|---------|-------|-------|---------|------------------|-------|
| 120.0 * | 12.00 | 13.41 | -1.410 | 6265. 3.193e+005 | 1.000 |
| 144.0 * | 5.800 | 6.528 | -0.7281 | 6470. 3.460e+005 | 1.000 |
| 168.0 * | 3.700 | 3.178 | 0.5220 | 6582. 3.634e+005 | 1.000 |

#### Final Parameters

| Rsq | | 0.9881 |
|--------------------|------------|-------------|
| Rsq_adjusted | | 0.9842 |
| Corr_XY | | -0.9941 |
| No_points_lambda_z | | 5 |
| Lambda_z | 1/h | 0.0300 |
| Lambda_z_lower | h | 72.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 23.1091 |
| Tlag | h | 0.7333 |
| Tmax | h | 48.0000 |
| Cmax | ng/mL | 91.0000 |
| Cmax_D | ng/mL/mg | 0.2022 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 3.7000 |
| AUClast | h*ng/mL | 6582.0447 |
| AUCall | h*ng/mL | 6582.0447 |
| AUCINF_obs | h*ng/mL | 6705.4004 |
| AUCINF_D_obs | h*ng/mL/mg | 14.9009 |
| AUC_%Extrap_obs | % | 1.8396 |
| Vz_F_obs | L | 2237.4090 |
| CI_F_obs | L/h | 67.1101 |
| AUCINF_pred | h*ng/mL | 6687.9971 |
| AUCINF_D_pred | h*ng/mL/mg | 14.8622 |
| AUC_%Extrap_pred | % | 1.5842 |
| Vz_F_pred | L | 2243.2311 |
| Cl_F_pred | L/h | 67.2847 |
| AUMClast | h*h*ng/mL | 363436.8272 |
| AUMCINF_obs | h*h*ng/mL | 388273.1926 |
| AUMC_%Extrap_obs | % | 6.3966 |
| AUMCINF_pred | h*h*ng/mL | 384769.2189 |
| AUMC_%Extrap_pred | % | 5.5442 |
| MRTlast | h | 55.2164 |
| MRTINF_obs | h | 57.9045 |
| MRTINF_pred | h | 57.5313 |
| AUC0_24 | h*ng/mL | 1110.2790 |
| | _ | |

WinNonlin 7.0.0.2535

PARAMCD=M9A,SUBJID=PI ,APERIOD=2,TRTAN=1,TRTA=5 x 100 mg TF3

PI 09:24:11 Date: Time:


## Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 450.00 Dose amount:

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values
Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

| Time<br>h | Conc.<br>ng/mL | Pred.<br>ng/mL | Residual<br>ng/mL | AUC<br>h*ng/m | AUMC<br>L h*h*ng/r | Weight<br>mL |
|---|---|---|---|---|---|---|
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.6840 | | | 0.08550 | 0.06413 | |
| 1.000 | 1.620 | | | 0.3735 | 0.3308 | |
| 1.500 | 4.940 | | | 2.014 | 2.588 | |
| 2.000 | 8.610 | | | 5.401 | 8.746 | |
| 3.000 | 16.00 | | | 17.71 | 41.36 | |
| 4.000 | 21.30 | | | 36.36 | 108.0 | |
| 6.033 | 27.10 | | | 85.56 | 360.8 | |
| 8.000 | 43.00 | | | 154.5 | 859.8 | |
| 12.00 | 52.80 | | | 346.1 | 2815. | |
| 16.03 | 73.20 | | | 600.2 | 6460. | |
| 24.00 | 106.0 | | | 1314. 2.12 | 27e+004 | |
| 36.00 | 101.0 | | | 2556. 5.84 | l6e+004 | |
| 48.00 | 132.0 | | | 3954. 1.18 | 33e+005 | |
| 60.00 | 84.00 | | | 5228. 1.86 | 55e+005 | |
| 72.00 | 92.50 | | | 6287. 2.56 | 7e+005 | |
| 96.00 | 50.30 | | | 7950. 3.94 | 14e+005 | |
| 120.0 * | 19.00 | 18.81 | 0.1944 | 8721. 4.7 | 762e+005 | 1.000 |
| 144.0 * | 9.760 | 9.963 | -0.2030 | 9054. 5.1 | 97e+005 | 1.000 |
| 168.0 * | 5.340 | 5.285 | 0.05474 | 9230. 5.4 | 469e+005 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

| Rsq | | 0.9992 |
|--------------------|------------|-------------|
| Rsq_adjusted | | 0.9984 |
| Corr_XY | | -0.9996 |
| No_points_lambda_z | | 3 |
| Lambda_z | 1/h | 0.0264 |
| Lambda_z_lower | h | 119.9833 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 26.2226 |
| Tlag | h | 0.5000 |
| Tmax | h | 48.0000 |
| Cmax | ng/mL | 132.0000 |
| Cmax_D | ng/mL/mg | 0.2933 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 5.3400 |
| AUClast | h*ng/mL | 9229.8441 |
| AUCall | h*ng/mL | 9229.8441 |
| AUCINF_obs | h*ng/mL | 9431.8627 |
| AUCINF_D_obs | h*ng/mL/mg | 20.9597 |
| AUC %Extrap obs | % | 2.1419 |
| Vz_F_obs | L | 1804.9497 |
| CI F obs | L/h | 47.7106 |
| AUCINF_pred | h*ng/mL | 9429.7918 |
| AUCINF D pred | h*ng/mL/mg | 20.9551 |
| AUC_%Extrap_pred | % | 2.1204 |
| Vz_F_pred | L | 1805.3460 |
| CI_F_pred | L/h | 47.7211 |
| AUMClast | h*h*ng/mL | 546937.6967 |
| AUMCINF_obs | h*h*ng/mL | 588519.4215 |
| AUMC_%Extrap_obs | % | 7.0655 |
| AUMCINF_pred | h*h*ng/mL | 588093.1737 |
| AUMC %Extrap pred | % | 6.9981 |
| MRTlast | h | 59.2575 |
| MRTINF_obs | h | 62.3969 |
| MRTINF_pred | h | 62.3654 |
| AUC0_24 | h*ng/mL | 1314.0077 |
| | • | |

WinNonlin 7.0.0.2535
PARAMCD=M9A,SUBJID=PI ,APERIOD=2,TRTAN=1,TRTA=5 x 100 mg TF3
```
0 \ 0 \ 0000 \ 0 \ 0 \ 0
\begin{smallmatrix}0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0
000000000000000000
0 00 0 00 0 00 0 0 0 0 00 0
\begin{smallmatrix}0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0&0
```

| % | 5.0286 |
|---|---|
| L | 2492.1375 |
| L/h | 52.8860 |
| h*ng/mL | 8521.6327 |
| h*ng/mL/mg | 18.9370 |
| % | 5.1708 |
| L | 2488.4063 |
| L/h | 52.8068 |
| h*h*ng/mL | 520000.0031 |
| h*h*ng/mL | 612060.0678 |
| % | 15.0410 |
| h*h*ng/mL | 614805.1625 |
| % | 15.4204 |
| h | 64.3485 |
| h | 71.9320 |
| h | 72.1464 |
| h*ng/mL | 1050.1452 |
| | L L/h h*ng/mL m*ng/mL/mg % L L/h h*h*ng/mL h*h*ng/mL % h*h*ng/mL h*h h h |

WinNonlin 7.0.0.2535

PARAMCD=M9A,SUBJID=PI ,APERIOD=1,TRTAN=1,TRTA=5 x 100 mg TF3

Date: PI Time: 09:24:10


#### Settings

----

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

| - | | | | | | |
|---|---|---|---|---|---|---|
| Time<br>h | Conc.<br>ng/mL | Pred.<br>ng/mL | Residual<br>ng/mL | AUC<br>h*ng/mL | AUMC<br>h*h*ng/mL | Weight |
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.033 | 0.8570 | | | 0.1214 ( | 0.1255 | |
| 1.500 | 2.350 | | | 0.8697 | 1.155 | |
| 2.017 | 4.400 | | | 2.613 | 4.357 | |
| 3.000 | 13.90 | | | 11.61 | 29.22 | |
| 4.000 | 20.70 | | | 28.91 | 91.47 | |
| 6.000 | 29.50 | | | 79.11 | 351.3 | |
| 8.000 | 39.50 | | | 148.1 | 844.3 | |
| 12.00 | 61.70 | | | 350.5 | 2957. | |
| 16.00 | 77.30 | | | 628.5 | 6911. | |
| 24.03 | 113.0 | | | 1393. 2.279 | e+004 | |
| 36.00 | 127.0 | | | 2829. 6.639 | e+004 | |
| 48.00 | 133.0 | | | 4389. 1.321 | e+005 | |
| 60.00 | 99.30 | | | 5773. 2.065 | e+005 | |
| 72.00 | 94.70 | | | 6937. 2.832 | e+005 | |
| 96.00 * | 77.00 | 73.84 | 3.155 | 8990. 4.54 | 8e+005 | 1.000 |
| 120.3 * | 39.90 | 44.30 | -4.405 1.03 | 36e+004 6.01 | 1e+005 | 1.000 |
| 144.0 * | 29.20 | 26.88 | 2.318 1.1 | 17e+004 7.08 | 31e+005 | 1.000 |
| 168.0 * | 15.90 | 16.22 | -0.3189 1.1 | 70e+004 7.89 | 94e+005 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

| Rsq | | 0.9846 |
|--------------------|------------|-------------|
| Rsq_adjusted | | 0.9769 |
| Corr_XY | | -0.9923 |
| No_points_lambda_z | | 4 |
| Lambda_z | 1/h | 0.0211 |
| Lambda_z_lower | h | 96.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 32.9246 |
| Tlag | h | 0.7500 |
| Tmax | h | 48.0000 |
| Cmax | ng/mL | 133.0000 |
| Cmax_D | ng/mL/mg | 0.2956 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 15.9000 |
| AUClast | h*ng/mL | 11697.6472 |
| AUCall | h*ng/mL | 11697.6472 |
| AUCINF_obs | h*ng/mL | 12452.9008 |
| AUCINF_D_obs | h*ng/mL/mg | 27.6731 |
| AUC_%Extrap_obs | % | 6.0649 |
| Vz_F_obs | L | 1716.4757 |
| Cl_F_obs | L/h | 36.1362 |
| AUCINF_pred | h*ng/mL | 12468.0506 |
| AUCINF_D_pred | h*ng/mL/mg | 27.7068 |
| AUC_%Extrap_pred | % | 6.1790 |
| Vz_F_pred | L | 1714.3901 |
| Cl_F_pred | L/h | 36.0923 |
| AUMClast | h*h*ng/mL | 789355.4269 |
| AUMCINF_obs | h*h*ng/mL | 952112.7497 |
| AUMC_%Extrap_obs | % | 17.0943 |
| AUMCINF_pred | h*h*ng/mL | 955377.5311 |
| AUMC_%Extrap_pred | % | 17.3776 |
| MRTlast | h | 67.4798 |
| MRTINF_obs | h | 76.4571 |
| MRTINF_pred | h | 76.6261 |
| AUC0_24 | h*ng/mL | 1389.1184 |

WinNonlin 7.0.0.2535

PARAMCD=M9A,SUBJID=PI ,APERIOD=2,TRTAN=1,TRTA=5 x 100 mg TF3

PI 09:24:13 Date: Time:


# Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 450.00 Dose amount:

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values
Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

# Summary Table

AUC AUMC Time Conc. Pred. Residual Weight h\*ng/mL h\*h\*ng/mL h ng/mL ng/mL ng/mL 0.0000 0.0000 0.0000 0.0000 0.2500 0.0000 0.0000 0.0000 0.0000 0.5000 0.0000 0.0000

| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
|---------|--------|-------|---------|----------|-----------|-------|
| 1.000 | 0.5660 | | | 0.07075 | 0.07075 | |
| 1.500 | 0.9810 | | | 0.4575 | 0.5801 | |
| 2.000 | 2.040 | | | 1.213 | 1.968 | |
| 3.000 | 4.780 | | | 4.623 | 11.18 | |
| 4.000 | 11.10 | | | 12.56 | 40.55 | |
| 6.000 | 16.50 | | | 40.16 | 183.9 | |
| 8.000 | 28.70 | | | 85.36 | 512.5 | |
| 12.00 | 53.00 | | | 248.8 | 2244. | |
| 16.00 | 78.30 | | | 511.4 | 6021. | |
| 24.00 | 119.0 | | | 1301. 2. | 246e+004 | |
| 36.00 | 93.30 | | | 2568. 6. | 018e+004 | |
| 48.00 | 110.0 | | | 3788. 1. | 120e+005 | |
| 60.00 | 75.00 | | | 4885. 1. | 708e+005 | |
| 72.00 | 69.80 | | | 5753. 2. | 281e+005 | |
| 96.00 * | 64.30 | 63.99 | 0.3098 | 7361. 3 | .629e+005 | 1.000 |
| 120.0 * | 32.70 | 35.39 | -2.692 | 8483. 4 | .825e+005 | 1.000 |
| 144.0 * | 22.60 | 19.57 | 3.025 | 9139. 5 | .686e+005 | 1.000 |
| 168.0 * | 10.10 | 10.83 | -0.7263 | 9511.6 | .262e+005 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

| Rsq | | 0.9822 |
|--------------------|------------|-------------|
| Rsq_adjusted | | 0.9733 |
| Corr XY | | -0.9911 |
| No_points_lambda_z | | 4 |
| Lambda z | 1/h | 0.0247 |
| Lambda_z_lower | h | 96.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL Lambda z | h | 28.0887 |
| Tlag | h | 0.7500 |
| Tmax | h | 24.0000 |
| Cmax | ng/mL | 119.0000 |
| Cmax_D | ng/mL/mg | 0.2644 |
| Tlast | , h | 168.0000 |
| Clast | ng/mL | 10.1000 |
| AUClast | h*ng/mL | 9511.4885 |
| AUCall | h*ng/mL | 9511.4885 |
| AUCINF_obs | h*ng/mL | 9920.7752 |
| AUCINF_D_obs | h*ng/mL/mg | 22.0462 |
| AUC_%Extrap_obs | % | 4.1256 |
| Vz_F_obs | L | 1838.1174 |
| Cl_F_obs | L/h | 45.3594 |
| AUCINF_pred | h*ng/mL | 9950.2083 |
| AUCINF_D_pred | h*ng/mL/mg | 22.1116 |
| AUC_%Extrap_pred | % | 4.4092 |
| Vz_F_pred | L | 1832.6802 |
| CI_F_pred | L/h | 45.2252 |
| AUMClast | h*h*ng/mL | 626161.4043 |
| AUMCINF_obs | h*h*ng/mL | 711507.2909 |
| AUMC_%Extrap_obs | % | 11.9951 |
| AUMCINF_pred | h*h*ng/mL | 717644.7709 |
| AUMC_%Extrap_pred | % | 12.7477 |
| MRTlast | h | 65.8321 |
| MRTINF_obs | h | 71.7189 |
| MRTINF_pred | h | 72.1236 |
| AUC0_24 | h*ng/mL | 1300.5628 |

WinNonlin 7.0.0.2535

PARAMCD=M9A,SUBJID=PI ,APERIOD=2,TRTAN=1,TRTA=5 x 100 mg TF3

Date: PI Time: 09:24:12

WINNONLIN NONCOMPARTMENTAL ANALYSIS PROGRAM 7.0.0.2535

```
0 0 0000 0 0 0
\begin{smallmatrix} 0 \end{smallmatrix} \ 0 \\ \ 0 \end{smallmatrix} \ 0 \end{smallmatrix} \ 0 \\ \ 0 \end{smallmatrix} \ 0 \\ \ 0 \end{smallmatrix} \ 0 \\ \ 0 
000000000000000
^{\circ}
```

CI\_F\_pred L/h 21.2205 **AUMClast** h\*h\*ng/mL 1462502.4585 AUMCINF\_obs h\*h\*ng/mL 2115761.4405 AUMC\_%Extrap\_obs 30.8758 AUMCINF\_pred AUMC\_%Extrap\_pred h\*h\*ng/mL 2160427.5432 32.3050 MRTlast 80.3874 MRTINF\_obs 100.6875 h MRTINF\_pred h 101.8783 AUC0\_24 h\*ng/mL 1353.5810

WinNonlin 7.0.0.2535

PARAMCD=M9A,SUBJID=PI ,APERIOD=2,TRTAN=1,TRTA=5 x 100 mg TF3

Date: PI Time: 09:24:11


### Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

# Summary Table

| Time | Conc. | Pred. | Residual | AUC | AUMC | Weight |
|---------|--------|-------|----------|-------------|-----------|--------|
| h | ng/mL | ng/mL | ng/mL | h*ng/mL | h*h*ng/mL | |
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5333 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.500 | 1.160 | | | 0.2900 | .4350 | |
| 2.000 | 1.880 | | | 1.050 | 1.810 | |
| 3.000 | 5.630 | | | 4.805 | 12.14 | |
| 4.000 | 10.60 | | | 12.92 | 41.78 | |
| 6.000 | 16.90 | | | 40.42 | 185.6 | |
| 8.000 | 27.90 | | | 85.22 | 510.2 | |
| 12.00 | 48.90 | | | 238.8 | 2130. | |
| 16.00 | 66.00 | | | 468.6 | 5416. | |
| 24.02 | 91.50 | | | 1100. 1.846 | e+004 | |
| 36.00 | 102.0 | | | 2259. 5.363 | e+004 | |
| 48.00 | 112.0 | | | 3543. 1.079 | e+005 | |
| 60.02 | 92.00 | | | 4765. 1.737 | e+005 | |
| 72.00 * | 77.40 | 77.13 | 0.2688 | 5778. 2.40 | 3e+005 | 1.000 |
| 96.00 * | 48.90 | 49.49 | -0.5938 | 7267. 3.64 | 1e+005 | 1.000 |
| 120.0 * | 32.50 | 31.76 | 0.7406 | 8231. 4.67 | 3e+005 | 1.000 |
| 144.0 * | 19.90 | 20.38 | -0.4795 | 8847. 5.48 | 1e+005 | 1.000 |
| 168.0 * | 13.20 | 13.08 | 0.1228 | 9239. 6.08 | 9e+005 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

#### Final Parameters

Rsq 0.9993 Rsq\_adjusted 0.9991 Corr\_XY -0.9997

| No_points_lambda_z | | 5 |
|--------------------|------------|-------------|
| Lambda_z | 1/h | 0.0185 |
| Lambda_z_lower | h | 72.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 37.4961 |
| Tlag | h | 1.0000 |
| Tmax | h | 48.0000 |
| Cmax | ng/mL | 112.0000 |
| Cmax_D | ng/mL/mg | 0.2489 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 13.2000 |
| AUClast | h*ng/mL | 9238.7096 |
| AUCall | h*ng/mL | 9238.7096 |
| AUCINF_obs | h*ng/mL | 9952.7703 |
| AUCINF_D_obs | h*ng/mL/mg | 22.1173 |
| AUC_%Extrap_obs | % | 7.1745 |
| Vz_F_obs | L | 2445.8495 |
| Cl_F_obs | L/h | 45.2135 |
| AUCINF_pred | h*ng/mL | 9946.1262 |
| AUCINF_D_pred | h*ng/mL/mg | 22.1025 |
| AUC_%Extrap_pred | % | 7.1125 |
| Vz_F_pred | L | 2447.4834 |
| Cl_F_pred | L/h | 45.2437 |
| AUMClast | h*h*ng/mL | 608898.1387 |
| AUMCINF_obs | h*h*ng/mL | 767487.8146 |
| AUMC_%Extrap_obs | % | 20.6635 |
| AUMCINF_pred | h*h*ng/mL | 766012.1980 |
| AUMC_%Extrap_pred | % | 20.5106 |
| MRTlast | h | 65.9073 |
| MRTINF_obs | h | 77.1130 |
| MRTINF_pred | h | 77.0161 |
| AUC0_24 | h*ng/mL | 1098.4079 |

WinNonlin 7.0.0.2535

PARAMCD=M9A,SUBJID=PI ,APERIOD=1,TRTAN=2,TRTA=2 x 250 mg TF3

PI 09:24:11 Date: Time:


# Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 450.00 Dose amount:

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values
Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

| Time<br>h | Conc.<br>ng/mL | Pred.<br>ng/mL | Residual<br>ng/mL | AUC<br>h*ng/ml | AUMC<br>L h*h*ng/mL | Weight |
|---|---|---|---|---|---|---|
| 0.0000<br>0.2500 | 0.0000<br>0.0000 | | | 0.0000<br>0.0000 | 0.0000<br>0.0000 | |
| 0.5000<br>0.7500<br>1.033 | 0.0000<br>0.0000<br>0.0000 | | | 0.0000<br>0.0000<br>0.0000 | 0.0000<br>0.0000<br>0.0000 | |
| 1.500<br>2.000 | 0.6930<br>2.370 | | | 0.1617<br>0.9275 | 0.2426<br>1.687 | |
| 3.000<br>4.000<br>6.000 | 7.170<br>13.00<br>21.90 | | | 5.697<br>15.78<br>50.68 | 14.81<br>51.57<br>235.0 | |

| 8.000 | 31.00 | | | 103.6 614.4 | |
|---------|-------|-------|---------|------------------|-------|
| 12.00 | 47.20 | | | 260.0 2243. | |
| 16.00 | 66.50 | | | 487.4 5504. | |
| 24.00 | 78.60 | | | 1068. 1.731e+004 | |
| 36.00 | 85.30 | | | 2051. 4.705e+004 | |
| 48.00 | 97.50 | | | 3148. 9.355e+004 | |
| 60.00 | 77.70 | | | 4195. 1.498e+005 | |
| 72.00 | 69.20 | | | 5075. 2.078e+005 | |
| 96.00 * | 48.90 | 48.76 | 0.1356 | 6478. 3.247e+005 | 1.000 |
| 120.0 * | 28.30 | 28.04 | 0.2587 | 7382. 4.214e+005 | 1.000 |
| 144.0 * | 15.70 | 16.12 | -0.4248 | 7895. 4.885e+005 | 1.000 |
| 168.0 * | 9.410 | 9.272 | 0.1377 | 8190. 5.342e+005 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

| Rsq | | 0.9993 |
|------------------------|------------|--------------------|
| Rsq adjusted | | 0.9990 |
| Corr XY | | -0.9997 |
| No points lambda z | | 4 |
| Lambda z | 1/h | 0.0231 |
| Lambda_z_lower | h | 96.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 30.0649 |
| Tlag | h | 1.0333 |
| Tmax | h | 48.0000 |
| Cmax | ng/mL | 97.5000 |
| Cmax_D | ng/mL/mg | 0.2167 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 9.4100 |
| AUClast | h*ng/mL | 8190.3625 |
| AUCall | h*ng/mL | 8190.3625 |
| AUCINF_obs | h*ng/mL | 8598.5159 |
| AUCINF_D_obs | h*ng/mL/mg | 19.1078 |
| AUC_%Extrap_obs | % | 4.7468 |
| Vz_F_obs | L | 2269.9838 |
| Cl_F_obs | L/h | 52.3346 |
| AUCINF_pred | h*ng/mL | 8592.5451 |
| AUCINF_D_pred | h*ng/mL/mg | 19.0945 |
| AUC_%Extrap_pred | . % | 4.6806 |
| Vz_F_pred | L | 2271.5612 |
| Cl_F_pred | L/h | 52.3710 |
| AUMClast | h*h*ng/mL | 534231.3564 |
| AUMCINF_obs | h*h*ng/mL | 620504.5365 |
| AUMC_%Extrap_obs | % | 13.9037 |
| AUMCINF_pred | h*h*ng/mL | 619242.4596 |
| AUMC_%Extrap_pred | % | 13.7282 |
| MRTlast | h | 65.2268 |
| MRTINF_obs | h<br>h | 72.1641<br>72.0674 |
| MRTINF_pred<br>AUC0 24 | | 1067.7825 |
| AUCU_24 | h*ng/mL | 1007.7625 |

WinNonlin 7.0.0.2535

PARAMCD=M9A,SUBJID=pj ,APERIOD=1,TRTAN=2,TRTA=2 x 250 mg TF3

Date: PI Time: 09:24:12


# Settings

-----

Model: Plasma Data, Extravascular Administration Number of nonmissing observations: 22

Dose time: 0.00

```
\begin{smallmatrix} 0 \end{smallmatrix} \ 0 \\ \ 0 \end{smallmatrix} \ 0 \end{smallmatrix} \ 0 \end{smallmatrix} \ 0 \\ \ 0 \end{smallmatrix} \ 0 \\ \ 0 \end{smallmatrix} \ 0 \\ \ 0 \end{smallmatrix} \ 0 \\ \ 0 
0 00 0 00 0 00 0 0 0 0 0
^{\circ}
^{\circ}
```

MRTINF\_obs MRTINF\_pred AUC0\_24 h 100.1916 100.0458 h 1197.8551 h\*ng/mL

WinNonlin 7.0.0.2535

PARAMCD=M9A,SUBJID=PI ,APERIOD=1,TRTAN=2,TRTA=2 x 250 mg TF3

> Date: PI 09:24:12 Time:


#### Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 450.00 Dose amount:

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

#### Summary Table

| Time<br>h | Conc.<br>ng/mL | Pred.<br>ng/mL | Residual<br>ng/mL | AUC<br>h*ng/mL | AUMC<br>h*h*ng/mL | Weight |
|---|---|---|---|---|---|---|
| 0.0000<br>0.2500<br>0.5000<br>0.7500<br>1.000<br>1.500<br>2.000<br>3.000<br>4.000<br>6.000<br>8.000 | 0.0000<br>0.0000<br>0.0000<br>0.0000<br>0.0000<br>0.0000<br>1.650<br>4.080<br>8.480<br>14.20<br>24.20 | | | 0.0000<br>0.0000<br>0.0000<br>0.0000<br>0.0000<br>0.0000<br>0.4125<br>3.278<br>9.558<br>32.24<br>70.64 | 0.0000<br>0.0000<br>0.0000<br>0.0000<br>0.0000<br>0.0000<br>0.8250<br>8.595<br>31.68<br>150.8<br>429.6 | |
| 12.00<br>16.00<br>24.00<br>36.00<br>48.00<br>60.00<br>72.00<br>96.00 *<br>120.0 *<br>144.0 * | 47.00<br>61.40<br>129.0<br>131.0<br>156.0<br>110.0<br>116.0<br>90.90<br>58.80<br>37.10<br>20.90 | 93.68<br>57.56<br>35.37<br>21.73 | 1.733 1.2 | | 2e+004<br>le+005<br>2e+005<br>3e+005<br>3e+005<br>17e+005<br>00e+005 | 1.000<br>1.000<br>1.000<br>1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

# Final Parameters

| Rsq | | 0.9957 |
|--------------------|-----|----------|
| Rsq_adjusted | | 0.9935 |
| Corr_XY | | -0.9978 |
| No_points_lambda_z | | 4 |
| Lambda_z | 1/h | 0.0203 |
| Lambda_z_lower | h | 96.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 34.1553 |
| Tlag | h | 1.5000 |
| Tmax | h | 48.0000 |

156.0000 Cmax ng/mL ng/mL/mg Cmax D 0.3467 168.0000 Tlast h ng/mL 20.9000 Clast **AUClast** h\*ng/mL 13456.8835 13456.8835 AUCall h\*ng/mL AUCINF\_obs 14486.7451 h\*ng/mL AUCINF\_D\_obs h\*ng/mL/mg 32.1928 AUC\_%Extrap\_obs Vz\_F\_obs 7.1090 1530,6443 CI\_F\_obs L/h 31.0629 AUCINF\_pred AUCINF\_D\_pred h\*ng/mL 14527.6863 h\*ng/mL/mg 32.2837 AUC\_%Extrap\_pred 7.3708 Vz\_F\_pred 1526.3307 L CI\_F\_pred L/h 30.9753 **AUMClast** h\*h\*ng/mL 964871.5723 AUMCINF\_obs h\*h\*ng/mL 1188635.4435 AUMC\_%Extrap\_obs 18.8253 AUMCINF\_pred h\*h\*ng/mL 1197530.9708 AUMC\_%Extrap\_pred 19.4283 MRTlast 71.7010 h MRTINF\_obs h 82.0499 MRTINF\_pred 82.4309 h AUC0\_24 h\*ng/mL 1191.4375

WinNonlin 7.0.0.2535

PARAMCD=M9A,SUBJID=pj ,APERIOD=2,TRTAN=2,TRTA=2 x 250 mg TF3

Date: pj Time: 09:24:10


# Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

### Summary Table

Pred. AUC AUMC Weight Time Conc. Residual h\*ng/mL h\*h\*ng/mL h ng/mL ng/mL ng/mL 0.0000 0.0000 0.0000 0.0000 0.2667 0.0000 0.0000 0.0000 0.5000 0.0000 0.0000 0.0000 0.7500 0.0000 0.0000 0.0000 1.017 0.0000 0.0000 0.0000 1.500 1.700 0.4108 0.6162 2.000 4.060 1.851 3.284 3.000 24.89 11.70 9.731 4.000 22.70 26.93 87.84 76.33 6.000 26.70 338.8 8.000 44.10 147.1 851.8 12.00 63.60 362.5 3084. 16.00 81.20 652.1 7209. 24.00 122.0 1465. 2.412e+004 36.00 108.0 2843. 6.530e+004 48.00 126.0 4247. 1.249e+005 5591. 1.972e+005 60.00 99.10

| 72.73 | 89.60 | | 6792. 2.767e+005 | |
|---------|-------|-------|------------------------------|-------|
| 96.03 | 74.40 | | 8697. 4.368e+005 | |
| 120.0 * | 52.40 | 50.19 | 2.210 1.020e+004 5.982e+005 | 1.000 |
| 144.0 * | 23.80 | 25.94 | -2.143 1.107e+004 7.116e+005 | 1.000 |
| 168.0 * | 14.00 | 13.41 | 0.5906 1.151e+004 7.803e+005 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

| Rsq | | 0.9874 |
|--------------------|------------|-------------|
| Rsq_adjusted | | 0.9747 |
| Corr_XY | | -0.9937 |
| No_points_lambda_z | | 3 |
| Lambda z | 1/h | 0.0275 |
| Lambda z lower | h | 120.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL Lambda z | h | 25.2082 |
| Tlag | h | 1.0167 |
| Tmax | h | 48.0000 |
| Cmax | ng/mL | 126.0000 |
| Cmax D | ng/mL/mg | 0.2800 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 14.0000 |
| AUClast | h*ng/mL | 11513.9438 |
| AUCall | h*ng/mL | 11513.9438 |
| AUCINF obs | h*ng/mL | 12023.0928 |
| AUCINF_D_obs | h*ng/mL/mg | 26.7180 |
| AUC_%Extrap_obs | % | 4.2348 |
| Vz_F_obs | L | 1361.1727 |
| Cl_F_obs | L/h | 37.4280 |
| AUCINF_pred | h*ng/mL | 12001.6152 |
| AUCINF_D_pred | h*ng/mL/mg | 26.6703 |
| AUC_%Extrap_pred | % | 4.0634 |
| Vz_F_pred | L | 1363.6086 |
| Cl_F_pred | L/h | 37.4950 |
| AUMClast | h*h*ng/mL | 780326.2198 |
| AUMCINF_obs | h*h*ng/mL | 884379.8860 |
| AUMC_%Extrap_obs | % | 11.7657 |
| AUMCINF_pred | h*h*ng/mL | 879990.5652 |
| AUMC_%Extrap_pred | % | 11.3256 |
| MRTlast | h | 67.7723 |
| MRTINF_obs | h | 73.5568 |
| MRTINF_pred | h | 73.3227 |
| AUC0_24 | h*ng/mL | 1464.9308 |

WinNonlin 7.0.0.2535

PARAMCD=M9A,SUBJID=pj ,APERIOD=1,TRTAN=1,TRTA=5 x 100 mg TF3

Date: PI 09:24:10 Time:


# Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 450.00 Dose amount:

Calculation method: Linear Trapezoidal Rule for for Increasing Values, Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

```
0 0 0 0 0 0 0 0 0 0 0 0 0
000000000000000000
0 \ 00 \ 0 \ 000 \ 0 \ 000 \ 0 \ 000 \ 0
000000000000000000
^{\circ}
^\circ
```

0 00 0 0 0 000 00 00 00 00 0 0 0 0

Date: PI 09:24:11 Time:


### Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values, Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

### Summary Table

| Time | Conc. | Pred. | Residual | AUC | AUMO | Weight |
|---------|--------|-------|-------------|-------------|----------|--------|
| h | ng/mL | ng/mL | ng/mL | | | |
| | | | | | g | |
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7667 | 0.5190 | | | 0.06920 | 0.05305 | |
| 1.000 | 1.020 | | | 0.2488 | 0.2185 | |
| 1.500 | 4.760 | | | 1.694 | 2.258 | |
| 2.000 | 7.340 | | | 4.719 | 7.713 | |
| 3.000 | 16.70 | | | 16.74 | 40.10 | |
| 4.000 | 24.60 | | | 37.39 | 114.4 | |
| 6.000 | 28.40 | | | 90.39 | 383.2 | |
| 8.017 | 42.00 | | | 161.4 | 894.5 | |
| 12.00 | 52.60 | | | 349.8 | 2822. | |
| 16.00 | 78.60 | | | 612.2 | 6600. | |
| 24.02 | 139.0 | | | 1484. 2.50 | 02e+004 | |
| 36.00 | 89.00 | | | 2828. 6.47 | 75e+004 | |
| 48.00 | 122.0 | | | 4094, 1,19 | 91e+005 | |
| 60.00 | 76.70 | | | 5266. 1.81 | 18e+005 | |
| 72.00 | 86.40 | | | 6244. 2.46 | 8e+005 | |
| 96.00 * | 62.30 | 62.69 | -0.3926 | 8013. 3.9 | 42e+005 | 1.000 |
| 120.0 * | 34.80 | 34.98 | -0.1822 | 9146. 5.1 | 53e+005 | 1.000 |
| 144.0 * | 20.10 | 19.52 | 0.5801 | 9789. 5.9 | 994e+005 | 1.000 |
| 168.0 * | 10.70 | 10.89 | -0.1920 1.0 | 015e+004 6. | 548e+005 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

#### Final Parameters

| Rsq | | 0.9993 |
|--------------------|----------|------------|
| Rsq_adjusted | | 0.9989 |
| Corr_XY | | -0.9996 |
| No_points_lambda_z | | 4 |
| Lambda_z | 1/h | 0.0243 |
| Lambda_z_lower | h | 96.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 28.5145 |
| Tlag | h | 0.5000 |
| Tmax | h | 24.0167 |
| Cmax | ng/mL | 139.0000 |
| Cmax_D | ng/mL/mg | 0.3089 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 10.7000 |
| AUClast | h*ng/mL | 10146.7471 |
| AUCall | h*ng/mL | 10146.7471 |
| AUCINF_obs | h*ng/mL | 10586.9216 |

AUCINF\_D\_obs h\*ng/mL/mg 23.5265 AUC\_%Extrap\_obs Vz\_F\_obs Cl\_F\_obs 4.1577 1748.5734 42.5053 L/h AUCINF\_pred AUCINF\_D\_pred h\*ng/mL 10594.8198 23.5440 h\*ng/mL/mg AUC\_%Extrap\_pred 4.2292 Vz\_F\_pred Cl\_F\_pred AUMClast 1747.2699 L L/h 42.4736 h\*h\*ng/mL 654771.4914 AUMCINF\_obs 746828.6060 h\*h\*ng/mL AUMC\_%Extrap\_obs AUMCINF\_pred 12.3264 748480.4180 h\*h\*ng/mL AUMC\_%Extrap\_pred 12.5199 MRTlast 64.5302 h MRTINF obs h 70.5426 MRTINF\_pred AUC0\_24 70.6459 h h\*ng/mL 1482.0848

WinNonlin 7.0.0.2535

PARAMCD=M9A,SUBJID=PI ,APERIOD=1,TRTAN=1,TRTA=5 x 100 mg TF3

Date: pj Time: 09:24:10


# Settings

-----

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

| Time | Conc. | Pred. | Residual | AUC | AUMC | Weight |
|---------|--------|-------|------------|--------------|-----------|--------|
| h | ng/mL | ng/mL | ng/mL | h*ng/mL | h*h*ng/mL | |
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.050 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 2.017 | 0.9720 | | | 0.2511 | 0.5064 | |
| 3.000 | 2.510 | | | 1.963 | 5.172 | |
| 4.000 | 4.580 | | | 5.508 | 18.10 | |
| 6.000 | 10.60 | | | 20.69 | 100.0 | |
| 8.000 | 20.50 | | | 51.79 | 327.6 | |
| 12.00 | 40.10 | | | 173.0 | 1618. | |
| 16.00 | 61.70 | | | 376.6 | 4555. | |
| 24.00 | 108.0 | | | 1055. 1.887 | /e+004 | |
| 36.00 | 124.0 | | | 2447. 6.121 | le+004 | |
| 48.00 | 150.0 | | | 4091. 1.312 | 2e+005 | |
| 60.00 | 108.0 | | | 5626. 2.135 | e+005 | |
| 72.00 * | 100.0 | 106.1 | -6.101 | 6873. 2.95 | 8e+005 | 1.000 |
| 96.07 * | 69.70 | 67.16 | 2.538 | 8893. 4.64 | 1e+005 | 1.000 |
| 120.0 * | 43.20 | 42.62 | 0.5787 1.0 | 22e+004 6.0 | 60e+005 | 1.000 |
| 144.1 * | 29.70 | 26.95 | 2.746 1.1 | 09e+004 7.2 | 01e+005 | 1.000 |
| 168.6 * | 15.50 | 16.93 | -1.433 1.1 | 62e+004 8.03 | 30e+005 | 1.000 |

### \*) Starred values were included in the estimation of Lambda\_z.

# Final Parameters

| Rsq | | 0.9895 |
|--------------------|------------|--------------|
| Rsq_adjusted | | 0.9860 |
| Corr_XY | | -0.9947 |
| No_points_lambda_z | | 5 |
| Lambda_z | 1/h | 0.0190 |
| Lambda_z_lower | h | 72.0000 |
| Lambda_z_upper | h | 168.5833 |
| HL_Lambda_z | h | 36.4801 |
| Tlag | h | 1.5000 |
| Tmax | h | 48.0000 |
| Cmax | ng/mL | 150.0000 |
| Cmax_D | ng/mL/mg | 0.3333 |
| Tlast | h | 168.5833 |
| Clast | ng/mL | 15.5000 |
| AUClast | h*ng/mL | 11622.1791 |
| AUCall | h*ng/mL | 11622.1791 |
| AUCINF_obs | h*ng/mL | 12437.9382 |
| AUCINF_D_obs | h*ng/mL/mg | 27.6399 |
| AUC_%Extrap_obs | % | 6.5586 |
| Vz_F_obs | L | 1904.1201 |
| CI_F_obs | L/h | 36.1796 |
| AUCINF_pred | h*ng/mL | 12513.3305 |
| AUCINF_D_pred | h*ng/mL/mg | 27.8074 |
| AUC_%Extrap_pred | % | 7.1216 |
| Vz_F_pred | L | 1892.6479 |
| CI_F_pred | L/h | 35.9616 |
| AUMClast | h*h*ng/mL | 802966.8658 |
| AUMCINF_obs | h*h*ng/mL | 983423.3415 |
| AUMC_%Extrap_obs | % | 18.3498 |
| AUMCINF_pred | h*h*ng/mL | 1000101.1085 |
| AUMC_%Extrap_pred | % | 19.7114 |
| MRTlast | h | 69.0892 |
| MRTINF_obs | h | 79.0664 |
| MRTINF_pred | h | 79.9229 |
| AUC0_24 | h*ng/mL | 1055.3881 |

WinNonlin 7.0.0.2535

PARAMCD=M9A,SUBJID=PI ,APERIOD=1,TRTAN=1,TRTA=5 x 100 mg TF3

Date: PI 09:24:12 Time:


### Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 450.00 Dose amount:

Calculation method: Linear Trapezoidal Rule for for Increasing Values, Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

| Time | Conc. | Pred. | Residual | AUC | AUMC | Weight |
|---|---|---|---|---|---|---|
| h | ng/mL | ng/mL | ng/mL | h*ng/mL | h*h*ng/mL | |
| 0.0000<br>0.2667 | 0.0000<br>0.0000 | | | | .0000 | |

| 0 | ).5000 | 0.0000 | | | 0.0000 | 0.0000 | |
|---|---------|--------|-------|-----------|----------|------------|-------|
| ( | ).7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| | 1.000 | 0.9330 | | | 0.1166 | 0.1166 | |
| | 1.500 | 2.800 | | | 1.050 | 1.400 | |
| | 2.000 | 5.830 | | | 3.207 | 5.365 | |
| | 3.000 | 12.10 | | | 12.17 | 29.34 | |
| | 4.000 | 19.80 | | | 28.12 | 87.09 | |
| | 6.000 | 28.20 | | | 76.12 | 335.5 | |
| | 8.000 | 43.60 | | | 147.9 | 853.5 | |
| | 12.00 | 50.00 | | | 335.1 | 2751. | |
| | 16.00 | 66.50 | | | 568.1 | 6079. | |
| | 24.00 | 84.70 | | | 1173. 1. | 847e+004 | |
| | 36.00 | 71.60 | | | 2109. 4. | 638e+004 | |
| | 48.00 | 82.90 | | | 3036. 8. | 572e+004 | |
| | 60.00 | 47.60 | | | 3799. 1. | 265e+005 | |
| | 72.00 | 52.30 | | | 4398. 1. | 663e+005 | |
| | 96.00 * | 24.50 | 25.16 | -0.6629 | 5278. 2 | .388e+005 | 1.000 |
| | 120.2 * | 16.20 | 15.36 | 0.8446 | 5763. 2 | 2.908e+005 | 1.000 |
| | 144.0 * | 9.180 | 9.428 | -0.2481 | 6058. 3 | 3.294e+005 | 1.000 |
| | 168.0 * | 5.770 | 5.771 | -0.001056 | 6234. | 3.567e+005 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

| Rsq | | 0.9964 |
|--------------------|------------|-------------|
| Rsq_adjusted | | 0.9947 |
| Corr XY | | -0.9982 |
| No points lambda z | | 4 |
| Lambda z | 1/h | 0.0205 |
| Lambda_z_lower | h | 96.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL Lambda z | h | 33.8921 |
| Tlag | h | 0.7500 |
| Tmax | h | 24.0000 |
| Cmax | ng/mL | 84.7000 |
| Cmax_D | ng/mL/mg | 0.1882 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 5.7700 |
| AUClast | h*ng/mL | 6233.8544 |
| AUCall | h*ng/mL | 6233.8544 |
| AUCINF_obs | h*ng/mL | 6515.9838 |
| AUCINF_D_obs | h*ng/mL/mg | 14.4800 |
| AUC_%Extrap_obs | % | 4.3298 |
| Vz_F_obs | L | 3376.7981 |
| CI_F_obs | L/h | 69.0609 |
| AUCINF_pred | h*ng/mL | 6516.0354 |
| AUCINF_D_pred | h*ng/mL/mg | 14.4801 |
| AUC_%Extrap_pred | % | 4.3306 |
| Vz_F_pred | L | 3376.7713 |
| Cl_F_pred | L/h | 69.0604 |
| AUMClast | h*h*ng/mL | 356739.5529 |
| AUMCINF_obs | h*h*ng/mL | 417932.2728 |
| AUMC_%Extrap_obs | % | 14.6418 |
| AUMCINF_pred | h*h*ng/mL | 417943.4680 |
| AUMC_%Extrap_pred | % | 14.6441 |
| MRTlast | h | 57.2262 |
| MRTINF_obs | h | 64.1396 |
| MRTINF_pred | h | 64.1408 |
| AUC0_24 | h*ng/mL | 1172.9224 |

WinNonlin 7.0.0.2535 PARAMCD=M9A,SUBJID=PI ,APERIOD=1,TRTAN=1,TRTA=5 x 100 mg TF3

PI 09:24:11 Date: Time:

```
0\ 0
0\ 00\ 0\ 000\ 0\ 00\ 0\ 0\ 0
0 \  \, 
^{\circ}
```

Vz\_F\_pred Cl\_F\_pred AUMClast L 1738.6070 L/h 28.7614 h\*h\*ng/mL 1037749.8400 1431322.9332 AUMCINF\_obs h\*h\*ng/mL AUMC\_%Extrap\_obs AUMCINF\_pred 27.4972 h\*h\*ng/mL 1435098.3570 AUMC\_%Extrap\_pred 27.6879 74.6227 MRTlast h MRTINF\_obs h 91.5787 MRTINF\_pred AUC0\_24 91.7233 h 1147.1918 h\*ng/mL

WinNonlin 7.0.0.2535

PARAMCD=M9A,SUBJID=pj ,APERIOD=2,TRTAN=1,TRTA=5 x 100 mg TF3

Date: **PI** Time: 09:24:10


### Settings

-----

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 18

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting

Lambda\_z method: Find best fit for lambda\_z, Log regression

# Summary Table

| Time | Conc. | Pred. | Residual | AUC | AUMC | Weight |
|---------|--------|-------|----------|------------|-----------|--------|
| h | ng/mL | ng/mL | ng/mL | . h*ng/m | L h*h*ng/ | mL |
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.000 | 0.7480 | | | 0.09350 | 0.09350 | |
| 1.500 | 1.590 | | | 0.6780 | 0.8768 | |
| 2.000 | 3.230 | | | 1.883 | 3.088 | |
| 3.000 | 8.730 | | | 7.863 | 19.41 | |
| 4.000 | 16.40 | | | 20.43 | 65.31 | |
| 6.000 | 25.90 | | | 62.73 | 286.3 | |
| 8.000 | 41.20 | | | 129.8 | 771.3 | |
| 12.00 | 48.60 | | | 309.4 | 2597. | |
| 16.00 | 68.10 | | | 542.8 | 5943. | |
| 24.00 | 76.80 | | | 1122. 1.76 | 67e+004 | |
| 36.00 * | 61.70 | 62.22 | -0.5229 | 1950. 4.2 | 32e+004 | 1.000 |
| 48.00 * | 56.30 | 52.89 | 3.408 | 2658. 7.1 | 97e+004 | 1.000 |
| 60.00 * | 40.70 | 44.96 | -4.261 | 3235. 1.0 | 29e+005 | 1.000 |
| 72.00 * | 40.00 | 38.22 | 1.782 | 3719. 1.3 | 49e+005 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

# Final Parameters

Rsq 0.8921
Rsq\_adjusted 0.8382
Corr\_XY -0.9445
No\_points\_lambda\_z 4
Lambda\_z 1/h 0.0135
Lambda\_z\_lower h 36.0000

| Lambda_z_upper | h | 72.0000 |
|-------------------|------------|-------------|
| HL_Lambda_z | h | 51.1963 |
| Tlag | h | 0.7500 |
| Tmax | h | 24.0000 |
| Cmax | ng/mL | 76.8000 |
| Cmax_D | ng/mL/mg | 0.1707 |
| Tlast | h | 72.0000 |
| Clast | ng/mL | 40.0000 |
| AUClast | h*ng/mL | 3718.7655 |
| AUCall | h*ng/mL | 3718.7655 |
| AUCINF_obs | h*ng/mL | 6673.1936 |
| AUCINF_D_obs | h*ng/mL/mg | 14.8293 |
| AUC_%Extrap_obs | % | 44.2731 |
| Vz_F_obs | L | 4980.7212 |
| Cl_F_obs | L/h | 67.4340 |
| AUCINF_pred | h*ng/mL | 6541.6103 |
| AUCINF_D_pred | h*ng/mL/mg | 14.5369 |
| AUC_%Extrap_pred | % | 43.1521 |
| Vz_F_pred | L | 5080.9075 |
| CI_F_pred | L/h | 68.7904 |
| AUMClast | h*h*ng/mL | 134890.2742 |
| AUMCINF_obs | h*h*ng/mL | 565825.2498 |
| AUMC_%Extrap_obs | % | 76.1604 |
| AUMCINF_pred | h*h*ng/mL | 546632.4136 |
| AUMC_%Extrap_pred | % | 75.3234 |
| MRTlast | h | 36.2729 |
| MRTINF_obs | h | 84.7908 |
| MRTINF_pred | h | 83.5624 |
| AUC0_24 | h*ng/mL | 1122.4280 |

WinNonlin 7.0.0.2535 PARAMCD=M9A,SUBJID=PI ,APERIOD=2,TRTAN=1,TRTA=5 x 100 mg TF3

> PI 09:24:12 Date: Time:


### Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount:

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

| Time | Conc. | Pred. | Residual | AUC | AUM | C Weight |
|--------|--------|-------|----------|---------|----------|----------|
| h | ng/mL | ng/mL | ng/mL | h*ng/n | nL h*h*n | g/mL |
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.000 | 0.5330 | | | 0.06663 | 0.06663 | |
| 1.500 | 1.650 | | | 0.6124 | 0.8186 | |
| 2.000 | 3.140 | | | 1.810 | 3.007 | |
| 3.000 | 8.460 | | | 7.610 | 18.84 | |
| 4.000 | 15.50 | | | 19.59 | 62.53 | |
| 6.000 | 24.80 | | | 59.89 | 273.3 | |
| 8.000 | 37.00 | | | 121.7 | 718.1 | |
| 12.00 | 49.90 | | | 295.5 | 2508. | |
| 16.00 | 60.70 | | | 516.7 | 5648. | |

| 24.00 | 93.90 | | | 1135. 1.855e+004 | |
|---------|-------|-------|---------|------------------|-------|
| 36.00 | 79.60 | | | 2174. 4.953e+004 | |
| 48.00 | 82.00 | | | 3143. 9.034e+004 | |
| 60.00 | 59.50 | | | 3985. 1.355e+005 | |
| 72.00 | 46.60 | | | 4619. 1.772e+005 | |
| 96.00 * | 34.80 | 33.44 | 1.360 | 5588. 2.581e+005 | 1.000 |
| 120.0 * | 14.10 | 15.87 | -1.772 | 6138. 3.165e+005 | 1.000 |
| 144.0 * | 8.470 | 7.533 | 0.9366 | 6404. 3.512e+005 | 1.000 |
| 168.0 * | 3.440 | 3.576 | -0.1356 | 6537. 3.719e+005 | 1.000 |

\*) Starred values were included in the estimation of Lambda\_z.

# Final Parameters

| Rsq | | 0.9890 |
|--------------------|------------|-------------|
| Rsq_adjusted | | 0.9835 |
| Corr_XY | | -0.9945 |
| No_points_lambda_z | | 4 |
| Lambda_z | 1/h | 0.0311 |
| Lambda_z_lower | h | 96.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 22.3233 |
| Tlag | h | 0.7500 |
| Tmax | h | 24.0000 |
| Cmax | ng/mL | 93.9000 |
| Cmax_D | ng/mL/mg | 0.2087 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 3.4400 |
| AUClast | h*ng/mL | 6537.4920 |
| AUCall | h*ng/mL | 6537.4920 |
| AUCINF_obs | h*ng/mL | 6648.2798 |
| AUCINF_D_obs | h*ng/mL/mg | 14.7740 |
| AUC_%Extrap_obs | % | 1.6664 |
| Vz_F_obs | L | 2179.9013 |
| CI_F_obs | L/h | 67.6867 |
| AUCINF_pred | h*ng/mL | 6652.6473 |
| AUCINF_D_pred | h*ng/mL/mg | 14.7837 |
| AUC_%Extrap_pred | % | 1.7310 |
| Vz_F_pred | L | 2178.4702 |
| Cl_F_pred | L/h | 67.6422 |
| AUMClast | h*h*ng/mL | 371890.3110 |
| AUMCINF_obs | h*h*ng/mL | 394070.6732 |
| AUMC_%Extrap_obs | % | 5.6285 |
| AUMCINF_pred | h*h*ng/mL | 394945.0669 |
| AUMC_%Extrap_pred | % | 5.8375 |
| MRTlast | h | 56.8858 |
| MRTINF_obs | h | 59.2741 |
| MRTINF_pred | h | 59.3666 |
| AUC0_24 | h*ng/mL | 1135.0899 |
| | - | |

WinNonlin 7.0.0.2535

PARAMCD=M9A,SUBJID=PI ,APERIOD=2,TRTAN=1,TRTA=5 x 100 mg TF3

Date: PI 09:24:11 Time:


# Settings

Model: Plasma Data, Extravascular Administration Number of nonmissing observations: 22

Dose time:

450.00 Dose amount:

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

```
0\;0\;0\;0\;0\;0\;0\;0\;0\;0\;0
000000000000000000
0\ 00\ 0\ 000\ 0\ 00\ 0\ 0\ 00\ 0
0 \  \, \varpi \  \, 0 \  \, \varpi \  \, 0 \  \, \varpi \  \, 0 \  \, 
0 \  \, 
0 \  \,
```

PARAMCD=M9A,SUBJID=PI ,APERIOD=1,TRTAN=2,TRTA=2 x 250 mg TF3

Date: 09:24:12 Time:


Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 450.00 Dose amount:

Calculation method: Linear Trapezoidal Rule for for Increasing Values, Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

# Summary Table

| Time<br>h | Conc.<br>ng/mL | Pred.<br>ng/mL | Residual<br>ng/mL | AUC<br>h*ng/mL | AUMC<br>h*h*ng/mL | Weight |
|---|---|---|---|---|---|---|
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 2.000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 3.000 | 1.690 | | | 0.8450 | 2.535 | |
| 4.000 | 4.270 | | | 3.825 | 13.61 | |
| 6.000 | 13.90 | | | 22.00 | 114.1 | |
| 8.000 | 19.40 | | | 55.30 | 352.7 | |
| 12.00 | 29.20 | | | 152.5 | 1364. | |
| 16.00 | 36.00 | | | 282.9 | 3217. | |
| 24.00 | 60.70 | | | 669.7 1.135 | | |
| 36.00 | 65.90 | | | 1429. 3.432 | | |
| 48.00 | 64.80 | | | 2213. 6.725 | | |
| 60.00 | 51.30 | | | 2907. 1.045 | 5e+005 | |
| 72.00 * | 45.80 | 46.81 | -1.009 | 3489. 1.42 | 9e+005 | 1.000 |
| 96.00 * | 27.80 | 26.11 | 1.694 | 4354. 2.14 | | 1.000 |
| 120.0 * | 14.80 | 14.56 | 0.2405 | 4849. 2.67 | | 1.000 |
| 144.0 * | 7.100 | 8.120 | -1.020 | 5101. 3.00 | | 1.000 |
| 168.0 * | 4.890 | 4.529 | 0.3614 | 5243. 3.22 | 25e+005 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

### Final Parameters

| Rsq | | 0.9917 |
|--------------------|----------|----------|
| Rsq_adjusted | | 0.9889 |
| Corr_XY | | -0.9958 |
| No_points_lambda_z | | 5 |
| Lambda_z | 1/h | 0.0243 |
| Lambda_z_lower | h | 72.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 28.4898 |
| Tlag | h | 2.0000 |
| Tmax | h | 36.0000 |
| Cmax | ng/mL | 65.9000 |
| Cmax_D | ng/mL/mg | 0.1464 |
| Tlast | h | 168.0000 |

Clast ng/mL 4.8900 **AUClast** h\*ng/mL 5242.9444 **AUCall** h\*ng/mL 5242.9444 AUCINF\_obs 5443.9334 h\*ng/mL AUCINF\_D\_obs AUC\_%Extrap\_obs h\*ng/mL/mg 12.0976 3.6920 Vz\_F\_obs Cl\_F\_obs L 3397.5292 82.6608 L/h AUCINF\_pred AUCINF\_D\_pred h\*ng/mL 5429.0808 h\*ng/mL/mg 12.0646 AUC\_%Extrap\_pred % 3.4285 Vz\_F\_pred Cl\_F\_pred L 3406.8240 L/h 82.8870 **AUMClast** h\*h\*ng/mL 322456.6593 AUMCINF\_obs h\*h\*ng/mL 364483.8764 AUMC %Extrap obs 11.5306 AUMCINF\_pred h\*h\*ng/mL 361378.1689 AUMC\_%Extrap\_pred 10.7703 61.5030 MRTlast h MRTINF\_obs 66.9523 h MRTINF\_pred 66.5634 h 669.6950 AUC0\_24 h\*ng/mL

WinNonlin 7.0.0.2535

PARAMCD=M9A,SUBJID=PI ,APERIOD=1,TRTAN=2,TRTA=2 x 250 mg TF3

Date: PI Time: 09:24:11


# Settings

-----

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00

Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

| Time | Conc. | Pred. | Residual | AUC | AUMC | Weight |
|---------|--------|-------|----------|-----------|-------------|--------|
| h | ng/mL | ng/mL | ng/mL | h*ng/n | nL h*h*ng/r | |
| | | | | | • | |
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.000 | 0.5060 | | | 0.06325 | 0.06325 | |
| 1.500 | 1.780 | | | 0.6348 | 0.8573 | |
| 2.000 | 4.280 | | | 2.150 | 3.665 | |
| 3.000 | 8.890 | | | 8.735 | 21.28 | |
| 4.000 | 16.60 | | | 21.48 | 67.81 | |
| 6.000 | 26.40 | | | 64.48 | 292.6 | |
| 8.017 | 37.60 | | | 129.0 | 756.3 | |
| 12.00 | 48.50 | | | 300.5 | 2516. | |
| 16.00 | 62.10 | | | 521.7 | 5667. | |
| 24.00 | 94.40 | | | 1148. 1.8 | 70e+004 | |
| 36.00 | 82.00 | | | 2204.5.0 | 25e+004 | |
| 48.00 | 117.0 | | | 3398. 1.0 | 17e+005 | |
| 60.03 | 110.0 | | | 4764. 1.7 | 53e+005 | |
| 72.00 * | 109.0 | 109.7 | -0.7457 | 6074. 2. | 618e+005 | 1.000 |
| 96.03 * | 69.80 | 69.67 | 0.1272 | 8188. 4. | 375e+005 | 1.000 |
| 120.0 * | 44.10 | 44.29 | -0.1880 | 9529. 5. | 812e+005 | 1.000 |

144.0 \* 29.00 28.13 0.8657 1.039e+004 6.946e+005 1.000 168.0 \* 17.50 17.87 -0.3725 1.094e+004 7.793e+005 1.000

\*) Starred values were included in the estimation of Lambda\_z.

#### Final Parameters

Rsq 0.9993 Rsq\_adjusted 0.9991Corr\_XY -0.9997 No\_points\_lambda\_z 5 Lambda z 0.0189 1/h Lambda\_z\_lower 72.0000 h Lambda\_z\_upper h 168.0000 HL\_Lambda\_z 36.6643 h Tlag h 0.7500 Tmax h 48.0000 ng/mL 117.0000 Cmax 0.2600 Cmax\_D ng/mL/mg 168.0000 Tlast h Clast ng/mL 17.5000 **AUClast** h\*ng/mL 10940.1694 AUCall h\*ng/mL 10940.1694 AUCINF\_obs AUCINF\_D\_obs h\*ng/mL 11865.8382 h\*ng/mL/mg 26.3685 AUC\_%Extrap\_obs 7.8011 2006.0035 Vz\_F\_obs L CI F obs L/h 37.9240 AUCINF\_pred 11885.5403 h\*ng/mL AUCINF\_D\_pred h\*ng/mL/mg 26.4123 AUC\_%Extrap\_pred Vz\_F\_pred 7.9540 2002.6782 L CI\_F\_pred AUMClast L/h 37.8611 h\*h\*ng/mL 779292.5903 AUMCINF\_obs h\*h\*ng/mL 983768.5418 AUMC\_%Extrap\_obs 20.7850 AUMCINF\_pred h\*h\*ng/mL 988120.6513 AUMC\_%Extrap\_pred 21.1339 MRTlast 71.2322 MRTINF obs 82.9076 h MRTINF\_pred 83.1364 h AUC0 24 h\*ng/mL 1147.6956

WinNonlin 7.0.0.2535

PARAMCD=M9A,SUBJID=PI ,APERIOD=1,TRTAN=2,TRTA=2 x 250 mg TF3

Date: pj Time: 09:24:12


Settings

-----

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00

Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

Summary Table

\_\_\_\_\_

Time Conc. Pred. Residual AUC AUMC Weight

| h | ng/mL | ng/mL | ng/mL | . h*ng/ml | . h*h*ng | /mL |
|---------|--------|-------|--------|------------|----------|-------|
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.8167 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.017 | 0.5110 | | | | 0.05195 | |
| 1.500 | 1.450 | | | 0.5250 | 0.7031 | |
| 2.000 | 3.040 | | | 1.648 | 2.767 | |
| 3.000 | 9.990 | | | 8.163 | 20.79 | |
| 4.000 | 18.00 | | | 22.16 | 71.78 | |
| 6.000 | 25.10 | | | 65.26 | 294.4 | |
| 8.033 | 39.90 | | | 131.3 | 773.4 | |
| 12.00 | 49.70 | | | 309.0 | 2592. | |
| 16.00 | 72.10 | | | 552.6 | 6092. | |
| 24.00 | 81.40 | | | 1167. 1.85 | 2e+004 | |
| 36.00 * | 71.30 | 76.84 | -5.544 | 2082. 4.58 | 35e+004 | 1.000 |
| 48.02 * | 70.40 | 61.56 | 8.840 | 2933. 8.16 | 60e+004 | 1.000 |
| 60.08 * | 49.60 | 49.27 | 0.3295 | 3650, 1,2 | 01e+005 | 1.000 |
| 72.00 * | 42.30 | 39.54 | 2.756 | 4196. 1.56 | 31e+005 | 1.000 |
| 95.73 * | 23.70 | 25.52 | -1.819 | 4958, 2,19 | 91e+005 | 1.000 |
| 120.1 * | 13.30 | 16.27 | -2.967 | 5397, 2,66 | 60e+005 | 1.000 |
| 144.0 * | 11.30 | 10.47 | 0.8282 | 5690, 3,0 | | 1.000 |
| 171.8 * | 6.700 | 6.273 | 0.4269 | 5935. 3.4 | | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

| Rsq | | 0.9851 |
|--------------------|------------|-------------|
| Rsq_adjusted | | 0.9826 |
| Corr_XY | | -0.9925 |
| No_points_lambda_z | | 8 |
| Lambda_z | 1/h | 0.0185 |
| Lambda_z_lower | h | 36.0000 |
| Lambda_z_upper | h | 171.7667 |
| HL_Lambda_z | h | 37.5598 |
| Tlag | h | 0.8167 |
| Tmax | h | 24.0000 |
| Cmax | ng/mL | 81.4000 |
| Cmax_D | ng/mL/mg | 0.1809 |
| Tlast | h | 171.7667 |
| Clast | ng/mL | 6.7000 |
| AUClast | h*ng/mL | 5934.5185 |
| AUCall | h*ng/mL | 5934.5185 |
| AUCINF_obs | h*ng/mL | 6297.5733 |
| AUCINF_D_obs | h*ng/mL/mg | 13.9946 |
| AUC_%Extrap_obs | % | 5.7650 |
| Vz_F_obs | L | 3872.0115 |
| Cl_F_obs | L/h | 71.4561 |
| AUCINF_pred | h*ng/mL | 6274.4383 |
| AUCINF_D_pred | h*ng/mL/mg | 13.9432 |
| AUC_%Extrap_pred | % | 5.4175 |
| Vz_F_pred | L | 3886.2883 |
| Cl_F_pred | L/h | 71.7196 |
| AUMClast | h*h*ng/mL | 342895.3193 |
| AUMCINF_obs | h*h*ng/mL | 424928.9793 |
| AUMC_%Extrap_obs | % | 19.3053 |
| AUMCINF_pred | h*h*ng/mL | 419701.5427 |
| AUMC_%Extrap_pred | % | 18.3002 |
| MRTlast | h | 57.7798 |
| MRTINF_obs | h | 67.4750 |
| MRTINF_pred | h | 66.8907 |
| AUC0_24 | h*ng/mL | 1166.6475 |
| _ | • | |

WinNonlin 7.0.0.2535 PARAMCD=M9A,SUBJID=PI ,APERIOD=2,TRTAN=2,TRTA=2 x 250 mg TF3

Date: PI

```
0 0 0000 0 0 0
000000000
000000000000000000
```

CI\_F\_obs L/h 25.7033 AUCINF\_pred AUCINF\_D\_pred h\*ng/mL 17459.5559 h\*ng/mL/mg 38.7990 AUC\_%Extrap\_pred % 10.2442 Vz\_F\_pred Cl\_F\_pred 1447.5440 L L/h 25.7739 AUMClast h\*h\*ng/mL 1177233.9428 AUMCINF obs 1588918.6096 h\*h\*ng/mL AUMC\_%Extrap\_obs 25.9097 AUMCINF\_pred h\*h\*ng/mL 1578171.0701 AUMC\_%Extrap\_pred 25.4052 MRTlast 75.1220 h MRTINF\_obs 90.7564 h MRTINF\_pred 90.3901 h AUC0\_24 h\*ng/mL 1471.3888

WinNonlin 7.0.0.2535

PARAMCD=M9A,SUBJID=p\_\_\_\_\_,APERIOD=2,TRTAN=2,TRTA=2 x 250 mg TF3

Date: PI Time: 09:24:12


# Settings

\_\_\_\_

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

| - | | | | | | | |
|---|---|---|---|---|---|---|---|
| | Time<br>h | Conc.<br>ng/mL | Pred.<br>ng/mL | Residual<br>ng/mL | AUC<br>h*ng/mL | AUMC<br>h*h*ng/mL | Weight |
| - | 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| | 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| | 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| | 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| | 1.000 | 0.0000 | | | 0.0000 | 0.0000 | |
| | 1.500 | 0.5120 | | | 0.1280 | .1920 | |
| | 2.000 | 1.060 | | | 0.5210 0 | .9140 | |
| | 3.000 | 3.050 | | | 2.576 | 6.549 | |
| | 4.000 | 8.270 | | | 8.236 | 27.66 | |
| | 6.000 | 19.40 | | | 35.91 | 177.1 | |
| | 8.000 | 32.40 | | | 87.71 | 552.7 | |
| | 12.03 | 53.60 | | | 261.1 | 2376. | |
| | 16.00 | 72.50 | | | 511.2 | 5956. | |
| | 24.00 | 107.0 | | | 1229. 2.087 | e+004 | |
| | 36.00 | 102.0 | | | 2483. 5.842 | e+004 | |
| | 48.00 | 123.0 | | | 3833. 1.159 | e+005 | |
| | 60.00 | 76.90 | | | 5011. 1.789 | e+005 | |
| | 72.00 * | 73.50 | 72.12 | 1.377 | 5913. 2.384 | te+005 | 1.000 |
| | 96.07 * | 44.20 | 41.73 | 2.473 | 7300. 3.53 | 5e+005 | 1.000 |
| | 120.1 * | 23.10 | 24.19 | -1.087 | 8080. 4.368 | e+005 | 1.000 |
| | 144.0 * | 12.00 | 14.03 | -2.031 | 8485. 4.899 | e+005 | 1.000 |
| | 168.0 * | 9.220 | 8.130 | 1.090 | 8739. 5.292 | 2e+005 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

| Rsq | | 0.9848 |
|----------------------|------------|-------------|
| Rsq_adjusted | | 0.9797 |
| Corr XY | | -0.9924 |
| No_points_lambda_z | | 5 |
| Lambda_z | 1/h | 0.0227 |
| Lambda z lower | h | 72.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 30.4843 |
| Tlag | h | 1.0000 |
| Tmax | h | 48.0000 |
| Cmax | ng/mL | 123.0000 |
| Cmax_D | ng/mL/mg | 0.2733 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 9.2200 |
| AUClast | h*ng/mL | 8738.5962 |
| AUCall | h*ng/mL | 8738.5962 |
| AUCINF_obs | h*ng/mL | 9144.0870 |
| AUCINF_D_obs | h*ng/mL/mg | 20.3202 |
| AUC_%Extrap_obs | % | 4.4345 |
| Vz F obs | L | 2164.3238 |
| Vz_F_obs<br>Cl_F_obs | L/h | 49.2121 |
| AUCINF_pred | h*ng/mL | 9096.1409 |
| AUCINF_D_pred | h*ng/mL/mg | 20.2136 |
| AUC_%Extrap_pred | % | 3.9307 |
| Vz_F_pred | L | 2175.7321 |
| Cl_F_pred | L/h | 49.4715 |
| AUMClast | h*h*ng/mL | 529238.5537 |
| AUMCINF_obs | h*h*ng/mL | 615194.2807 |
| AUMC_%Extrap_obs | % | 13.9721 |
| AUMCINF_pred | h*h*ng/mL | 605030.6982 |
| AUMC_%Extrap_pred | % | 12.5270 |
| MRTlast | h | 60.5633 |
| MRTINF_obs | h | 67.2778 |
| MRTINF_pred | h | 66.5151 |
| AUC0_24 | h*ng/mL | 1229.2377 |
| | - | |

WinNonlin 7.0.0.2535

PARAMCD=M9A,SUBJID=PI ,APERIOD=2,TRTAN=2,TRTA=2 x 250 mg TF3

Date: PI Time: 09:24:11


# Settings

\_\_\_\_

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

### Summary Table

Pred. AUC AUMC Time Conc. Residual Weight h\*ng/mL h\*h\*ng/mL ng/mL ng/mL ng/mL 0.0000 0.0000 0.5200 0.0000 0.2667 0.0000 0.06933 0.0000 0.5000 0.0000 0.06933 0.0000 0.7500 0.0000 0.06933 0.0000 1.000 0.9000 0.1818 0.1125

| 1.500 | 2.810 | | 1.109 1.391 | |
|---------|-------|-------|------------------------------|-------|
| 2.000 | 6.160 | | 3.352 5.525 | |
| 3.000 | 13.50 | | 13.18 31.94 | |
| 4.000 | 23.00 | | 31.43 98.19 | |
| 6.000 | 29.90 | | 84.33 369.6 | |
| 8.000 | 60.40 | | 174.6 1032. | |
| 12.00 | 75.30 | | 446.0 3806. | |
| 16.00 | 98.10 | | 792.8 8752. | |
| 24.00 | 197.0 | | 1973. 3.394e+004 | |
| 36.00 | 147.0 | | 4023. 9.482e+004 | |
| 48.00 | 193.0 | | 6063. 1.822e+005 | |
| 60.00 | 113.0 | | 7856. 2.780e+005 | |
| 72.00 * | 139.0 | 133.8 | 5.249 9368. 3.788e+005 | 1.000 |
| 96.00 * | 76.20 | 81.55 | -5.347 1.188e+004 5.864e+005 | 1.000 |
| 120.0 * | 53.80 | 49.72 | 4.082 1.342e+004 7.521e+005 | 1.000 |
| 144.0 * | 27.20 | 30.31 | -3.113 1.436e+004 8.744e+005 | 1.000 |
| 168.0 * | 19.60 | 18.48 | 1.119 1.491e+004 9.609e+005 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

| Rsq | | 0.9889 |
|--------------------|------------|--------------|
| Rsq_adjusted | | 0.9852 |
| Corr_XÝ | | -0.9944 |
| No_points_lambda_z | | 5 |
| Lambda z | 1/h | 0.0206 |
| Lambda z lower | h | 72.0000 |
| Lambda z upper | h | 168.0000 |
| HL Lambda z | h | 33.6205 |
| Tlag | h | 0.0000 |
| Tmax | h | 24.0000 |
| Cmax | ng/mL | 197.0000 |
| Cmax D | ng/mL/mg | 0.4378 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 19.6000 |
| AUClast | h*ng/mL | 14912.4021 |
| AUCall | h*ng/mL | 14912.4021 |
| AUCINF obs | h*ng/mL | 15863.0829 |
| AUCINF_D_obs | h*ng/mL/mg | 35.2513 |
| AUC_%Extrap_obs | % | 5.9930 |
| Vz_F_obs | L | 1375.9529 |
| CI_F_obs | L/h | 28.3678 |
| AUCINF_pred | h*ng/mL | 15808.8258 |
| AUCINF_D_pred | h*ng/mL/mg | 35.1307 |
| AUC_%Extrap_pred | % | 5.6704 |
| Vz_F_pred | L | 1380.6752 |
| CI_F_pred | L/h | 28.4651 |
| AUMClast | h*h*ng/mL | 960877.0560 |
| AUMCINF_obs | h*h*ng/mL | 1166703.3585 |
| AUMC_%Extrap_obs | % | 17.6417 |
| AUMCINF_pred | h*h*ng/mL | 1154956.4826 |
| AUMC_%Extrap_pred | % | 16.8040 |
| MRTlast | h | 64.4348 |
| MRTINF_obs | h | 73.5483 |
| MRTINF_pred | h | 73.0577 |
| AUC0_24 | h*ng/mL | 1973.2318 |
| | _ | |

WinNonlin 7.0.0.2535 PARAMCD=M9A,SUBJID=PI ,APERIOD=2,TRTAN=2,TRTA=2 x 250 mg TF3

> PI 09:24:10 Date: Time:

WINNONLIN NONCOMPARTMENTAL ANALYSIS PROGRAM 7.0.0.2535 Core Version 04Jun2007

```
\Pi \Pi \Pi \Pi \Pi \Pi \Pi
0\ 0
\begin{smallmatrix}0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0&0&0&0&0\\0&0&0&0
0 \  \, \varpi \  \, 0 \  \, \varpi \  \, 0 \  \, \varpi \  \, 0 \  \,
```

AUMCINF\_obs h\*h\*ng/mL 796632.2851 AUMC\_%Extrap\_obs 17.1957 AUMCINF\_pred 820586.4230 h\*h\*ng/mL AUMC\_%Extrap\_pred 19.6129 MRTlast 68.3280 h MRTINF\_obs 77.5158 h MRTINF\_pred 79.0092 h AUC0\_24 1163.1212 h\*ng/mL

WinNonlin 7.0.0.2535

PARAMCD=M9A,SUBJID=PI ,APERIOD=2,TRTAN=2,TRTA=2 x 250 mg TF3

Date: PI Time: 09:24:11


## Settings

----

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

#### Summary Table

| Time | Conc. | Pred. | Residual | AUC | AUMC | Weight |
|---------|--------|-------|----------|-------------|-----------|--------|
| h | ng/mL | ng/mL | ng/mL | h*ng/mL | h*h*ng/mL | |
| | | | | | • | |
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.000 | 0.8690 | | | 0.1086 | .1086 | |
| 1.500 | 1.890 | | | 0.7984 | 1.035 | |
| 2.000 | 3.160 | | | 2.061 | 3.323 | |
| 3.000 | 8.650 | | | 7.966 | 19.46 | |
| 4.000 | 18.50 | | | 21.54 | 69.43 | |
| 6.000 | 27.80 | | | 67.84 | 310.2 | |
| 8.000 | 38.90 | | | 134.5 | 788.2 | |
| 12.00 | 50.90 | | | 314.1 | 2632. | |
| 16.00 | 62.20 | | | 540.3 | 5844. | |
| 24.02 | 80.70 | | | 1113. 1.760 | e+004 | |
| 36.00 | 78.30 | | | 2066. 4.616 | e+004 | |
| 48.00 | 102.0 | | | 3148. 9.245 | e+004 | |
| 60.00 | 67.00 | | | 4147. 1.460 | e+005 | |
| 72.00 | 66.00 | | | 4945. 1.986 | e+005 | |
| 96.00 * | 58.00 | 57.98 | 0.01543 | 6431. 3.23 | 1e+005 | 1.000 |
| 120.0 * | 40.10 | 38.06 | 2.040 | 7596. 4.480 | De+005 | 1.000 |
| 144.0 * | 22.50 | 25.00 | -2.496 | 8326. 5.436 | e+005 | 1.000 |
| 168.0 * | 17.30 | 16.41 | 0.8884 | 8801. 6.17 | 5e+005 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

### Final Parameters

| Rsq | | 0.9816 |
|--------------------|-----|---------|
| Rsq_adjusted | | 0.9724 |
| Corr_XY | | -0.9908 |
| No_points_lambda_z | | 4 |
| Lambda z | 1/h | 0.0175 |

| Lambda_z_lower | h | 96.0000 |
|-------------------|------------|-------------|
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 39.5398 |
| Tlag | h | 0.7500 |
| Tmax | h | 48.0000 |
| Cmax | ng/mL | 102.0000 |
| Cmax_D | ng/mL/mg | 0.2267 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 17.3000 |
| AUClast | h*ng/mL | 8800.9454 |
| AUCall | h*ng/mL | 8800.9454 |
| AUCINF_obs | h*ng/mL | 9787.8039 |
| AUCINF_D_obs | h*ng/mL/mg | 21.7507 |
| AUC_%Extrap_obs | % | 10.0825 |
| Vz_F_obs | L | 2622.6240 |
| Cl_F_obs | L/h | 45.9756 |
| AUCINF_pred | h*ng/mL | 9737.1274 |
| AUCINF_D_pred | h*ng/mL/mg | 21.6381 |
| AUC_%Extrap_pred | % | 9.6146 |
| Vz_F_pred | L | 2636.2733 |
| Cl_F_pred | L/h | 46.2149 |
| AUMClast | h*h*ng/mL | 617454.0793 |
| AUMCINF_obs | h*h*ng/mL | 839540.5034 |
| AUMC_%Extrap_obs | % | 26.4533 |
| AUMCINF_pred | h*h*ng/mL | 828136.0830 |
| AUMC_%Extrap_pred | % | 25.4405 |
| MRTlast | h | 70.1577 |
| MRTINF_obs | h | 85.7741 |
| MRTINF_pred | h | 85.0493 |
| AUC0_24 | h*ng/mL | 1111.7870 |

WinNonlin 7.0.0.2535

PARAMCD=M9A,SUBJID=PI ,APERIOD=1,TRTAN=2,TRTA=2 x 250 mg TF3

Date: PI 09:24:13 Time:


# Settings

Model: Plasma Data, Extravascular Administration Number of nonmissing observations: 22

Dose time: 0.00 450.00 Dose amount:

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values
Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

| Time | Conc. | Pred. | Residual | AUC | AUMC | Weight |
|--------|--------|-------|----------|---------|-----------|--------|
| h | ng/mL | ng/mL | ng/mL | h*ng/mL | h*h*ng/mL | |
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.050 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.500 | 1.350 | | | 0.3038 | 0.4556 | |
| 2.000 | 3.350 | | | 1.479 | 2.637 | |
| 3.000 | 6.890 | | | 6.599 | 16.32 | |
| 4.000 | 14.40 | | | 17.24 | 55.46 | |
| 6.000 | 18.60 | | | 50.24 | 224.7 | |
| 8.017 | 31.70 | | | 101.0 | 593.4 | |
| 12.00 | 55.70 | | | 275.0 | 2431. | |

| 16.03 | 72.10 | | | 532.8 6110. | |
|---------|-------|-------|------------|---------------------|-------|
| 24.00 | 154.0 | | | 1433. 2.544e+004 | |
| 36.07 | 115.0 | | | 3045. 7.336e+004 | |
| 48.00 | 148.0 | | | 4614. 1.405e+005 | |
| 60.00 | 87.60 | | | 5996. 2.144e+005 | |
| 72.00 * | 112.0 | 111.5 | 0.4918 | 7194. 2.943e+005 | 1.000 |
| 96.00 * | 64.50 | 63.59 | 0.9050 | 9260. 4.656e+005 | 1.000 |
| 120.0 * | 35.10 | 36.27 | -1.169 1.0 | 042e+004 5.894e+005 | 1.000 |
| 144.0 * | 20.80 | 20.68 | 0.1150 1. | 108e+004 6.753e+005 | 1.000 |
| 168.0 * | 11.90 | 11.80 | 0.1030 1. | 146e+004 7.346e+005 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

| Rsq | | 0.9996 |
|--------------------|------------|-------------|
| Rsq_adjusted | | 0.9994 |
| Corr_XY | | -0.9998 |
| No_points_lambda_z | | 5 |
| Lambda_z | 1/h | 0.0234 |
| Lambda_z_lower | h | 72.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 29.6236 |
| Tlag | h | 1.0500 |
| Tmax | h | 24.0000 |
| Cmax | ng/mL | 154.0000 |
| Cmax D | ng/mL/mg | 0.3422 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 11.9000 |
| AUClast | h*ng/mL | 11457.7246 |
| AUCall | h*ng/mL | 11457.7246 |
| AUCINF_obs | h*ng/mL | 11966.3048 |
| AUCINF D obs | h*ng/mL/mg | 26.5918 |
| AUC_%Extrap_obs | % | 4.2501 |
| Vz_F_obs | L | 1607.1816 |
| Cl_F_obs | L/h | 37.6056 |
| AUCINF_pred | h*ng/mL | 11961.9025 |
| AUCINF_D_pred | h*ng/mL/mg | 26.5820 |
| AUC_%Extrap_pred | % | 4.2149 |
| Vz_F_pred | L | 1607.7731 |
| Cl_F_pred | L/h | 37.6194 |
| AUMClast | h*h*ng/mL | 734572.8306 |
| AUMCINF_obs | h*h*ng/mL | 841749.9263 |
| AUMC_%Extrap_obs | % | 12.7327 |
| AUMCINF_pred | h*h*ng/mL | 840822.1979 |
| AUMC_%Extrap_pred | % | 12.6364 |
| MRTlast | h | 64.1116 |
| MRTINF_obs | h | 70.3433 |
| MRTINF_pred | h | 70.2917 |
| AUC0_24 | h*ng/mL | 1433.3963 |
| | - | |

WinNonlin 7.0.0.2535

PARAMCD=M9A,SUBJID=PI ,APERIOD=2,TRTAN=2,TRTA=2 x 250 mg TF3

Date: PI Time: 09:24:10


# Settings

-----

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00

Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

```
000000000000000000
0 00 0 00 0 0 00 0 0 0 0 0
0 \  \, \varpi \  \, 0 \  \, \varpi \  \, 0 \  \, 
0 \  \,
```

AUC0\_24 h\*ng/mL 1381.0613

WinNonlin 7.0.0.2535 PARAMCD=M9A,SUBJID=PI ,APERIOD=2,TRTAN=2,TRTA=2 x 250 mg TF3

> Date: PI 09:24:11 Time:


# Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

### Summary Table

| Time | Conc.<br>ng/mL | Pred.<br>ng/mL | Residual<br>ng/mL | AUC<br>h*ng/m | AUMC<br>nL h*h*ng/ | |
|---|---|---|---|---|---|---|
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.000 | 0.6120 | | | 0.07650 | 0.07650 | |
| 1.500 | 1.530 | | | 0.6120 | 0.8033 | |
| 2.000 | 4.120 | | | 2.025 | 3.437 | |
| 3.000 | 8.820 | | | 8.495 | 20.79 | |
| 4.000 | 17.20 | | | 21.50 | 68.42 | |
| 6.000 | 22.90 | | | 61.60 | 274.6 | |
| 8.000 | 34.00 | | | 118.5 | 684.0 | |
| 12.00 | 59.60 | | | 305.7 | 2658. | |
| 16.00 | 79.70 | | | 584.3 | 6639. | |
| 24.00 | 117.0 | | | 1371. 2.2 | 97e+004 | |
| 36.03 | 118.0 | | | 2785. 6.5 | 45e+004 | |
| 48.00 | 118.0 | | | 4197, 1.2 | 48e+005 | |
| 60.00 | 80.80 | | | 5376. 1.8 | 80e+005 | |
| 72.00 * | 79.00 | 83.55 | -4.553 | 6335. 2.5 | 12e+005 | 1.000 |
| 96.00 * | 51.00 | 44.13 | 6.870 | 7870. 3.7 | 789e+005 | 1.000 |
| 120.0 * | 22.10 | 23.31 | -1.208 | 8700. 4.6 | 71e+005 | 1.000 |
| 144.0 * | 11.10 | 12.31 | -1.211 | 9083. 5.1 | 72e+005 | 1.000 |
| 168.0 * | 6.960 | 6.502 | 0.4580 | 9296. 5. | 502e+005 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

### Final Parameters

| Rsq | | 0.9897 |
|--------------------|----------|----------|
| Rsq_adjusted | | 0.9863 |
| Corr_XY | | -0.9949 |
| No_points_lambda_z | | 5 |
| Lambda_z | 1/h | 0.0266 |
| Lambda_z_lower | h | 72.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 26.0605 |
| Tlag | h | 0.7500 |
| Tmax | h | 36.0333 |
| Cmax | ng/mL | 118.0000 |
| Cmax_D | ng/mL/mg | 0.2622 |
| Tlast | h | 168.0000 |
|-------------------|------------|-------------|
| Clast | ng/mL | 6.9600 |
| AUClast | h*ng/mL | 9295.8206 |
| AUCall | h*ng/mL | 9295.8206 |
| AUCINF_obs | h*ng/mL | 9557.4986 |
| AUCINF_D_obs | h*ng/mL/mg | 21.2389 |
| AUC_%Extrap_obs | % | 2.7379 |
| Vz_F_obs | L | 1770.2161 |
| Cl_F_obs | L/h | 47.0834 |
| AUCINF_pred | h*ng/mL | 9540.2794 |
| AUCINF_D_pred | h*ng/mL/mg | 21.2006 |
| AUC_%Extrap_pred | % | 2.5624 |
| Vz_F_pred | L | 1773.4111 |
| Cl_F_pred | L/h | 47.1684 |
| AUMClast | h*h*ng/mL | 550187.6112 |
| AUMCINF_obs | h*h*ng/mL | 603987.9364 |
| AUMC_%Extrap_obs | % | 8.9075 |
| AUMCINF_pred | h*h*ng/mL | 600447.7210 |
| AUMC_%Extrap_pred | % | 8.3704 |
| MRTlast | h | 59.1866 |
| MRTINF_obs | h | 63.1952 |
| MRTINF_pred | h | 62.9382 |
| AUC0_24 | h*ng/mL | 1371.1045 |

WinNonlin 7.0.0.2535

PARAMCD=M9A,SUBJID=PI ,APERIOD=2,TRTAN=2,TRTA=2 x 250 mg TF3

PI 09:24:12 Date: Time:

## WINNONLIN NONCOMPARTMENTAL ANALYSIS PROGRAM 7.0.0.2535 Core Version 04Jun2007

# Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 450.00 Dose amount:

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values
Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

## Summary Table

| Time | Conc. | Pred. | Residual | AUC | AUMC | Weight |
|--------|--------|-------|----------|-------------|-----------|--------|
| h | ng/mL | ng/mL | ng/mL | h*ng/mL | h*h*ng/mL | |
| 0.0000 | 0.5070 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.5350 | | | 0.1303 0 | .01672 | |
| 0.5000 | 0.5140 | | | 0.2614 0 | .06577 | |
| 0.7500 | 0.6730 | | | 0.4097 | 0.1610 | |
| 1.000 | 1,110 | | | 0.6326 | 0.3628 | |
| 1.500 | 2.000 | | | 1.410 | 1.390 | |
| 2.000 | 3.470 | | | 2.778 | 3.875 | |
| 3.000 | 7.310 | | | 8.168 | 18.31 | |
| 4.000 | 11.00 | | | 17.32 | 51.28 | |
| 6.000 | 20.60 | | | 48.92 | 218.9 | |
| 8.000 | 31.10 | | | 100.6 | 591.3 | |
| 12.00 | 48.90 | | | 260.6 | 2262. | |
| 16.00 | 71.90 | | | 502.2 | 5737. | |
| 24.02 | 104.0 | | | 1207, 2,036 | e+004 | |
| 36.00 | 96.60 | | | 2409, 5,632 | | |
| 48.00 | 124.0 | | | 3732, 1,129 | | |
| 60.00 | 112.0 | | | 5147, 1,892 | | |
| 72.00 | 122.0 | | | 6551, 2,822 | | |
| 96.00 | 90.60 | | | 9084, 4,934 | | |
| 30.00 | 55.00 | | | 000 1. 4.00 | 0.000 | |

| 120.0 * | 57.60 | 57.14 | 0.4626 1.083e+004 6.807e+005 | 1.000 |
|---------|-------|-------|-------------------------------|-------|
| 144.0 * | 46.50 | 47.26 | -0.7560 1.208e+004 8.444e+005 | 1.000 |
| 168.0 * | 39.40 | 39.08 | 0.3164 1.311e+004 1.005e+006 | 1.000 |

\*) Starred values were included in the estimation of Lambda\_z.

#### Final Parameters

0.9946 Rsq Rsq\_adjusted 0.9892 Corr\_XY -0.9973No\_points\_lambda\_z 3 Lambda\_z 1/h 0.0079 Lambda z lower h 120.0000 Lambda\_z\_upper 168.0000 h HL\_Lambda\_z h 87.6115 Tlag 0.0000 h 48.0000 Tmax h Cmax 124.0000 ng/mL Cmax\_D ng/mL/mg 0.2756 Tlast h 168.0000 39,4000 Clast ng/mL AUClast h\*ng/mL 13105.0983 AUCall h\*ng/mL 13105.0983 AUCINF\_obs 18085.1283 h\*ng/mL AUCINF\_D\_obs h\*ng/mL/mg 40.1892 AUC\_%Extrap\_obs Vz\_F\_obs CI\_F\_obs AUCINF\_pred 27.5366 L 3145.0435 L/h 24.8823 h\*ng/mL 18045.1310 AUCINF\_D\_pred h\*ng/mL/mg 40.1003 AUC\_%Extrap\_pred % 27.3760 Vz\_F\_pred L 3152.0145 CI\_F\_pred L/h 24.9375 **AUM**Clast h\*h\*ng/mL 1004510.3979 AUMCINF obs h\*h\*ng/mL 2470614.7820 AUMC\_%Extrap\_obs 59.3417 AUMCINF\_pred h\*h\*ng/mL 2458839.7159 AUMC\_%Extrap\_pred 59.1470 MRTlast 76.6504 MRTINF\_obs 136.6103 h MRTINF\_pred h 136.2606 1205.5557 AUC0\_24 h\*ng/mL

WinNonlin 7.0.0.2535

PARAMCD=M9A,SUBJID=PI ,APERIOD=1,TRTAN=1,TRTA=5 x 100 mg TF3

Date: PI Time: 09:24:11


Settings

----

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 Dose amount: 450.00

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

Summary Table

-----

| Time<br>h | Conc.<br>ng/mL | Pred.<br>ng/mL | Residual<br>ng/mL | AUC<br>h*ng/mL | AUMC<br>h*h*ng/mL | Weight |
|---|---|---|---|---|---|---|
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7833 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.500 | 0.7050 | | | 0.1763 | 0.2644 | |
| 2.000 | 1.770 | | | 0.7950 | 1.414 | |
| 3.000 | 6.240 | | | 4.800 | 12.54 | |
| 4.000 | 12.40 | | | 14.12 | 46.70 | |
| 6.000 | 25.20 | | | 51.72 | 247.5 | |
| 8.000 | 35.40 | | | 112.3 | 681.9 | |
| 12.00 | 53.00 | | | 289.1 | 2520. | |
| 16.00 | 63.90 | | | 522.9 | 5837. | |
| 24.00 | 100.0 | | | 1179, 1,953 | e+004 | |
| 36.00 | 91.60 | | | 2327. 5.389 | e+004 | |
| 48.00 | 112.0 | | | 3549. 1.059 | e+005 | |
| 60.00 | 100.0 | | | 4820. 1.744 | e+005 | |
| 72.00 * | 109.0 | 114.6 | -5.600 | 6074, 2,575 | 5e+005 | 1.000 |
| 96.00 * | 84.20 | 79.75 | 4.450 | 8379. 4.50 | 0e+005 | 1.000 |
| 120.0 * | 52.10 | 55.50 | -3.398 | 9984. 6.218 | 3e+005 | 1.000 |
| 144.0 * | 45.50 | 38.62 | 6.879 1.1 | 15e+004 7.75 | 58e+005 | 1.000 |
| 168.0 * | 24.20 | 26.88 | | 96e+004 9.01 | | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

## Final Parameters

| Rsq | | 0.9652 |
|--------------------|------------|--------------|
| Rsq_adjusted | | 0.9537 |
| Corr XY | | -0.9825 |
| No_points_lambda_z | | 5 |
| Lambda_z | 1/h | 0.0151 |
| Lambda_z_lower | h | 72,0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 45.8851 |
| Tlag | h | 1.0000 |
| Tmax | h | 48.0000 |
| Cmax | ng/mL | 112.0000 |
| Cmax D | ng/mL/mg | 0.2489 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 24.2000 |
| AUClast | h*ng/mL | 11963.2267 |
| AUCall | h*ng/mL | 11963.2267 |
| AUCINF_obs | h*ng/mL | 13565.2245 |
| AUCINF_D_obs | h*ng/mL/mg | 30.1449 |
| AUC_%Extrap_obs | % | 11.8096 |
| Vz_F_obs | L | 2195.9987 |
| Cl_F_obs | L/h | 33.1731 |
| AUCINF_pred | h*ng/mL | 13742.4177 |
| AUCINF_D_pred | h*ng/mL/mg | 30.5387 |
| AUC_%Extrap_pred | % | 12.9467 |
| Vz_F_pred | L | 2167.6838 |
| Cl_F_pred | L/h | 32.7453 |
| AUMClast | h*h*ng/mL | 901108.7591 |
| AUMCINF_obs | h*h*ng/mL | 1276293.8569 |
| AUMC_%Extrap_obs | % | 29.3965 |
| AUMCINF_pred | h*h*ng/mL | 1317792.1958 |
| AUMC_%Extrap_pred | % | 31.6198 |
| MRTlast | h | 75.3232 |
| MRTINF_obs | h | 94.0857 |
| MRTINF_pred | h | 95.8923 |
| AUC0_24 | h*ng/mL | 1178.5200 |

WinNonlin 7.0.0.2535 PARAMCD=M9A,SUBJID=PI ,APERIOD=1,TRTAN=1,TRTA=5 x 100 mg TF3

```
00000000
0 \ 0 \ 0 \ 0 \ 0 \ 00 \ 00 \ 0 \ 00 \ 0
0000000000000000
0\ 00\ 0\ 000\ 0\ 00\ 0\ 0\ 00\ 0
00000000000000000
```

| Vz_F_obs | L | 1753.2571 |
|-------------------|------------|-------------|
| CI_F_obs | L/h | 42.1696 |
| AUCINF_pred | h*ng/mL | 10676.2794 |
| AUCINF_D_pred | h*ng/mL/mg | 23.7251 |
| AUC_%Extrap_pred | % | 7.1353 |
| Vz_F_pred | L | 1752.4203 |
| Cl_F_pred | L/h | 42.1495 |
| AUMClast | h*h*ng/mL | 712752.7128 |
| AUMCINF_obs | h*h*ng/mL | 871424.9340 |
| AUMC_%Extrap_obs | % | 18.2084 |
| AUMCINF_pred | h*h*ng/mL | 872493.5266 |
| AUMC_%Extrap_pred | % | 18.3085 |
| MRTlast | h | 71.8900 |
| MRTINF_obs | h | 81.6615 |
| MRTINF_pred | h | 81.7226 |
| AUC0_24 | h*ng/mL | 1516.6890 |

WinNonlin 7.0.0.2535

PARAMCD=M9A,SUBJID=PI ,APERIOD=1,TRTAN=1,TRTA=5 x 100 mg TF3

Date: PI 09:24:11 Time:

## WINNONLIN NONCOMPARTMENTAL ANALYSIS PROGRAM 7.0.0.2535 Core Version 04Jun2007

## Settings

Model: Plasma Data, Extravascular Administration Number of nonmissing observations: 22

Dose time: 0.00 450.00 Dose amount:

Calculation method: Linear Trapezoidal Rule for for Increasing Values,

Log Trapezoidal Rule for Decreasing Values
Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

# Summary Table

| Time<br>h | Conc.<br>ng/mL | Pred.<br>ng/mL | Residual<br>ng/mL | AUC<br>h*ng/mL | AUMC<br>h*h*ng/mL | Weight |
|---|---|---|---|---|---|---|
| 0.0000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.2500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.5000 | 0.0000 | | | 0.0000 | 0.0000 | |
| 0.7500 | 0.0000 | | | 0.0000 | 0.0000 | |
| 1.000 | 0.0000 | | | 0.0000 0 | .0000 | |
| 1.500 | 1.520 | | | 0.3800 0 | .5700 | |
| 2.000 | 2.410 | | | 1.363 | 2.345 | |
| 3.000 | 6.010 | | | 5.573 | 13.77 | |
| 4.000 | 8.680 | | | 12.92 | 10.15 | |
| 6.000 | 13.50 | | | 35.10 | 155.9 | |
| 8.000 | 18.50 | | | | 384.9 | |
| 12.00 | 34.20 | | | | 1502. | |
| 16.00 | 44.70 | | | | 3753. | |
| 24.00 | 69.50 | | | 787.1 1.329 | | |
| 36.00 | 93.60 | | | 1766. 4.351 | | |
| 48.00 | 107.0 | | | 2969. 9.454 | | |
| 60.03 | 65.40 | | | 3986. 1.490 | | |
| 72.00 * | 56.90 | 56.02 | 0.8754 | 4717. 1.97 <sup>-</sup> | | 1.000 |
| 96.00 * | 29.60 | 31.70 | -2.096 | 5719. 2.800 | | 1.000 |
| 120.0 * | 18.50 | 17.93 | 0.5678 | 6286. 3.40 | | 1.000 |
| 144.0 * | 11.00 | 10.15 | 0.8548 | 6632. 3.86 | | 1.000 |
| 168.0 * | 5.410 | 5.740 | -0.3297 | 6821. 4.153 | 3e+005 | 1.000 |

<sup>\*)</sup> Starred values were included in the estimation of Lambda\_z.

#### Final Parameters

| Rsq | | 0.9951 |
|--------------------|------------|-------------|
| Rsq_adjusted | | 0.9935 |
| Corr_XY | | -0.9976 |
| No_points_lambda_z | | 5 |
| Lambda_z | 1/h | 0.0237 |
| Lambda_z_lower | h | 72.0000 |
| Lambda_z_upper | h | 168.0000 |
| HL_Lambda_z | h | 29.2058 |
| Tlag | h | 1.0000 |
| Tmax | h | 48.0000 |
| Cmax | ng/mL | 107.0000 |
| Cmax_D | ng/mL/mg | 0.2378 |
| Tlast | h | 168.0000 |
| Clast | ng/mL | 5.4100 |
| AUClast | h*ng/mL | 6821.3604 |
| AUCall | h*ng/mL | 6821.3604 |
| AUCINF_obs | h*ng/mL | 7049.3110 |
| AUCINF_D_obs | h*ng/mL/mg | 15.6651 |
| AUC_%Extrap_obs | % | 3.2337 |
| Vz_F_obs | L | 2689.7336 |
| Cl_F_obs | L/h | 63.8360 |
| AUCINF_pred | h*ng/mL | 7063.2019 |
| AUCINF_D_pred | h*ng/mL/mg | 15.6960 |
| AUC_%Extrap_pred | % | 3.4240 |
| Vz_F_pred | L | 2684.4438 |
| Cl_F_pred | L/h | 63.7105 |
| AUMClast | h*h*ng/mL | 415268.7757 |
| AUMCINF_obs | h*h*ng/mL | 463169.1793 |
| AUMC_%Extrap_obs | % | 10.3419 |
| AUMCINF_pred | h*h*ng/mL | 466088.1406 |
| AUMC_%Extrap_pred | % | 10.9034 |
| MRTlast | h | 60.8777 |
| MRTINF_obs | h | 65.7042 |
| MRTINF_pred | h | 65.9882 |
| AUC0_24 | h*ng/mL | 787.0975 |
| | _ | |

WinNonlin 7.0.0.2535

PARAMCD=M9A,SUBJID=PI ,APERIOD=2,TRTAN=1,TRTA=5 x 100 mg TF3

> Date: PI 09:24:10 Time:


# Settings

Model: Plasma Data, Extravascular Administration

Number of nonmissing observations: 22

Dose time: 0.00 450.00 Dose amount:

Calculation method: Linear Trapezoidal Rule for for Increasing Values, Log Trapezoidal Rule for Decreasing Values

Weighting for lambda\_z calculations: Uniform weighting Lambda\_z method: Find best fit for lambda\_z, Log regression

## Summary Table

| Time | Conc. | Pred. | Residual | AUC | AUMC | Weight |
|---|---|---|---|---|---|---|
| h | ng/mL | ng/mL | ng/mL | h*ng/ml | L h*h*ng/mL | |
| 0.0000<br>0.2500<br>0.5167<br>0.7500 | 0.0000<br>0.0000<br>0.0000<br>0.5200 | | | 0.0000<br>0.0000<br>0.0000<br>0.06067 | 0.0000<br>0.0000<br>0.0000<br>0.04550 | |

```
0 \  \, 
0 \  \,
```

# WinNonlin Plots - Tepotinib








































































## WinNonlin Plots - Tepotinib Metabolite MSC2571107A








































































## WinNonlin Plots - Tepotinib Metabolite MSC2571109A







































































